Prediction of Findings from the Ongoing COBRRA Trial Using Healthcare Database Analyses

DUPLICATE – COBRRA VTE

March 11<sup>th</sup>, 2022

#### 1. RCT Details

This section provides a high-level overview of an **ongoing** RCT that the described real-world evidence study is trying to replicate as closely as possible given the remaining limitations inherent in the healthcare databases.

#### 1.1 Title

Comparison of Bleeding Risk Between Rivaroxaban and Apixaban for the Treatment of Acute Venous Thromboembolism (COBRRA)

#### 1.2 <u>Intended aim(s)</u>

To compare the incidence of major and clinically relevant non-major bleeding events among subjects recently hospitalized with VTE initiating apixaban or rivaroxaban.

#### 1.3 Primary endpoint for replication

Time from randomization to the first confirmed, adjudicated occurrence of a major bleeding or clinically relevant non-major bleeding event through 90 days of anticoagulation treatment.

# 1.4 Required power for primary endpoint and noninferiority margin (if applicable)

The hazard ratio for the clinical trial is unknown because the trial is still ongoing. Based upon a recent meta-analysis comparing the safety of apixaban and rivaroxaban in a real-world evidence context, power was calculated using an array of effect sizes (Aryal et al. 2019).

#### 1.5 Secondary endpoint for replication (assay sensitivity) and RCT finding

- Adjudicated major bleeding events
- o Adjudicated clinically relevant non-major bleeding events
- Recurrent VTE
- All-cause mortality

# 1.6 Trial estimate

The trial is ongoing and scheduled to complete in June of 2023.

#### 2. Person responsible for implementation of replication in Aetion

Luke Zabotka, BA and Mufaddal Mahesri, MD, MPH, implemented the study design in the Aetion Evidence Platform. They are not responsible for the validity of the design and analytic choices. All implementation steps are recorded, and the implementation history is archived in the platform.

### 3. Data Source(s)

Optum CDM, IBM® MarketScan®, CMS NOAC

### 4. Study Design Diagram

The study design diagram visualizes key aspects of the longitudinal study design for expedited review.

Figure 1.



#### 5. Cohort Identification

#### 5.1 Cohort Summary

An active-comparator, new-user design, propensity score matched, retrospective cohort study will be applied to compare patients that received apixaban or rivaroxaban. Subjects will be selected on the basis of having one or more diagnoses codes indicating hospitalization for PE or DVT and being of age 18 or older. Subjects will be excluded if they were not treatment-naïve with respect to the use of another DOAC or warfarin in the prior 180 days or have had any indication of stage IV or V CKD, ESRD, an active bleeding episode, cancer, obesity, liver disease, or another indication for long-term anticoagulation, such as atrial fibrillation (AF), in the prior 180 days. Patients were also excluded if they have used any contraindicated medications in the prior 180 days. All patients were required to have continuous enrollment for 180 days prior to cohort entry to ensure incident use of the study drugs.

#### 5.2 Important steps for cohort formation

New use of the exposure (apixaban or rivaroxaban) is defined as no use of either drug in 180 days prior to meeting all eligibility criteria and initiation of exposure.

#### 5.2.1 Eligible cohort entry dates

The apixaban indication for treatment of DVT and PE was approved by the FDA on Aug 21, 2014. Rivaroxaban was initially approved for the same indication on Nov. 2, 2012.

- IBM® MarketScan®: Aug 21, 2014 December 31, 2019 (end of available data)
- Optum CDM: Aug 21, 2014 June 30, 2020 (end of available data)
- CMS NOAC: Aug 21, 2014 Dec 31, 2017 (end of available data)
- 5.2.2 Specify <u>inclusion/exclusion</u> criteria for cohort entry and define the index date Inclusion and exclusion criteria were adapted from the trial as closely as possible. Definitions for all inclusion/exclusion are provided in the **Appendix** and are summarized in the flowcharts below.

# 5.3 Flowchart of the study cohort assembly

For Apixaban vs. Rivaroxaban

| | Optun | n CDM | IBM® Ma | arketScan® | CMS - | CMS - NOAC |
|---|---|---|---|---|---|---|
| | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients | Less<br>Excluded<br>Patients | Remaining<br>Patients |
| All patients in our database | | 81,796,156 | | 205,537,714 | | 6,886,908 |
| Patients with Apixaban/Rivaroxaban [measured between Aug 21, 2014 and June 30, 2020.] | | 815,310 | | 592,812 | | 1,877,831 |
| Excluded due to insufficient enrollment [- 180, 0] | -114,272<br>(14%) | 701,038 | -44,015 (7%) | 548,797 | -211,569<br>(11%) | 1,666,262 |
| After wash-out for prior use of reference (Rivaroxaban) [-180, -1] | -216,874<br>(31%) | 484,164 | -203,091<br>(37%) | 345,706 | -622,705<br>(37%) | 1,043,557 |
| After wash-out for prior use of exposure (Apixaban) [-180, -1] | -333,847<br>(69%) | 150,317 | -205,703<br>(60%) | 140,003 | -682,837<br>(65%) | 360,720 |
| Excluded because patient qualified in >1 exposure category | -14 (<1%) | 150,303 | -23 (<1%) | 139,980 | -48 (<1%) | 360,672 |
| Exclusion of Missing Age [-180, 0] | -5 (<1%) | 150,298 | -0 (<1%) | 139,980 | -120 (<1%) | 360,552 |
| Exclusion of Gender (Exclude Missing Values) [start of all available data, 0] | -15 (<1%) | 150,283 | -0 (<1%) | 139,980 | - | - |
| Inclusion of Age >= 18 [0,0] | -141 (<1%) | 150,142 | -332 (<1%) | 139,648 | - | - |
| Inclusion of Proximal DVT or PE<br>Hospitalization [Day -14, Day 0] | -135,497<br>(90%) | 14,645 | -124,142<br>(89%) | 15,506 | -323,753<br>(90%) | 36,798 |
| Exclusion of Anticoagulant Use [-180, 0] | -311 (2%) | 14,334 | -308 (2%) | 15,198 | -1,602 (4%) | 35,196 |
| Exclusion of CKD Stage 4/5 or ESRD [-180, Day 0] | -345 (2%) | 13,989 | -171 (1%) | 15,027 | -1,265 (4%) | 33,931 |
| Exclusion of Dialysis or Renal Transplant) [ - 180, 0] | -30 (<1%) | 13,959 | -43 (<1%) | 14,984 | -141 (<1%) | 33,790 |
| Exclusion of Bleeding [-180, 0] | -805 (6%) | 13,154 | -1,750 (12%) | 13,234 | -5,812 (17%) | 27,978 |
| Exclusion of Cancer [-180, 0] | -1,592 (12%) | 11,562 | -796 (6%) | 12,438 | -2,795 (10%) | 25,183 |
| <b>Exclusion of Weight &gt; 120 kg</b> [-180, 0] | -868 (8%) | 10,694 | -549 (4%) | 11,889 | - | - |

| Exclusion of Significant Liver Disease [-180, | -356 (3%) | 10,338 | -199 (2%) | 11,690 | - | - |
|---|---|---|---|---|---|---|
| 0] | | | | | | |
| Exclusion of Use of Contraindicated | -80 (<1%) | 10,258 | -85 (<1%) | 11,605 | -281 (1%) | 22,790 |
| Medications [-180, 0] | | | | | | |
| <b>Exclusion of Prosthetic Heart Valve</b> [-180, 0] | -24 (<1%) | 10,234 | -8 (<1%) | 11,597 | - | - |
| Exclusion of Pregnancy [-180, 0] | -8 (<1%) | 10,226 | -17 (<1%) | 11,580 | - | - |
| Exclusion of Dual Antiplatelet Therapy [- | -176 (2%) | 10,050 | -164 (1%) | 11,416 | -624 (3%) | 22,115 |
| 180, Day 0 | | | | | | |
| Exclusion of Coagulopathy [-180, Day 0] | -196 (2%) | 9,854 | -132 (1%) | 11,284 | -338 (2%) | 21,777 |
| Exclusion of Atrial Fibrillation [-180, Day 0] | -261 (3%) | 9,593 | -142 (1%) | 11,142 | -637 (3%) | 21,140 |
| Final cohort | | 9,593 | | 11,142 | | 21,140 |

<sup>\*</sup>Data may be omitted to comply with the CMS cell suppression policy

#### 6. Variables

#### 6.1 Exposure-related variables:

#### Study drug:

The study exposure of interest is defined by a prescription drug claim indicating apixaban dispensation. New initiation will be defined by no such records of apixaban in the prior 180 days before treatment initiation (washout period) and fulfillment of study eligibility criteria.

### Comparator agent:

The comparator is defined by a prescription drug claim indicating rivaroxaban dispensation. New initiation will be defined by no such records of rivaroxaban in the prior 180 days before treatment initiation (washout period) and fulfillment of study eligibility criteria.

# 6.2 <u>Preliminary Covariates:</u>

- Age
- Gender
- CCI score

The covariate listed above represents only a small subset of the covariate vector that will ultimately be controlled for in the design and analysis. We use the covariates above only for initial feasibility analyses to judge whether there is likely to be sufficient overlap between treatment groups to proceed with the study. Remaining covariates are defined only after the study has passed the initial feasibility analysis and the initial power assessment and are listed in Table 1 (Appendix B).

#### 6.3 Outcome variables and study follow-up:

#### 6.3.1 Outcome variables

Effectiveness outcome variables of interest (definitions provided in **Appendix**):

- **Primary outcome:** Major bleeding and clinically relevant non-major bleeding through 3 months of treatment with apixaban or rivaroxaban.
- Secondary outcomes:
  - To assess the frequency of major bleeding events and clinically relevant non-major bleeding individually
  - o To assess extracranial and intracranial major bleeding events separately
  - To assess recurrent VTE
  - All-cause mortality

### 6.3.2 Study follow-up

Both as-treated (AT) and intention-to-treat (ITT) analyses will be conducted with treatment defined as the index drug on day of cohort entry. The **as-treated** will be the primary analysis. An allowable gap of 10 days between records indicating each treatment will qualify as "continuous therapy" with respect to follow-up in the as-treated analysis.

The follow-up will start the day after drug initiation (i.e., cohort entry date), and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest
- The date of end of continuous registration in the database
- End of the study period at 90 days

- Measured death event occurs
- Switch
- Discontinuation (10-day allowable grace period and risk window)
- Nursing home admission
- Initiation of another DOAC (dabigatran or edoxaban) or warfarin

In the secondary ITT analysis, we will not censor for discontinuation or switching among study drugs

### 7. Initial Feasibility Analysis

#### Aetion report name:

For apixaban vs. rivaroxaban

Optum CDM - <a href="https://bwh-dope.aetion.com/projects/details/1775/rwrs/78117">https://bwh-dope.aetion.com/projects/details/1775/rwrs/78117</a>
IBM® MarketScan® - <a href="https://bwh-dope.aetion.com/projects/details/1776/rwrs/78118">https://bwh-dope.aetion.com/projects/details/1776/rwrs/78118</a>
CMS NOAC - <a href="https://bwh-dope.aetion.com/projects/details/1777/rwrs/78119">https://bwh-dope.aetion.com/projects/details/1777/rwrs/78119</a>

Date conducted: Updated 01/13/2022

Complete Aetion feasibility analysis using age, gender, and CCI as the only covariates and the primary endpoint (Section 6.3.1) as the outcome. No measures of association will be computed, nor will incidence rates be stratified by treatment group.

- Report patient characteristics by treatment group
  - Apixaban vs Rivaroxaban

| | Optum CDM | | | IBM® MarketScan® | | | CMS - NOAC | | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Rivaroxaban -<br>Comparator | Apixaban<br>- Exposure | Difference | Rivaroxaban -<br>Comparator | Apixaban - Exposure | Difference | Rivaroxaban -<br>Comparator | Apixaban - Exposure | Difference |
| Number of patients | 4,502 | 5,091 | | 6,339 | 4,781 | | 12,786 | 8,329 | |

| Age | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| mean (sd) | 61.82 (16.97) | 69.00<br>(15.57) | -7.18 (-<br>7.83, -6.52) | 53.93 (15.65) | 57.11<br>(15.97) | -3.18 (-<br>3.78, -2.59) | 70.91 (13.02) | 74.18<br>(12.37) | -3.28 (-<br>3.63, -2.93) |
| median<br>[IQR] | 64.00 [51.00,<br>75.00] | 72.00<br>[60.00,<br>81.00] | | 55.00 [44.00,<br>63.00] | 57.00<br>[47.00,<br>66.00] | | 72.00 [66.00,<br>80.00] | 75.00<br>[68.00,<br>83.00] | |
| Gender | | | | | | | | | |
| М | 2,248 (49.9%) | 2,172<br>(42.7%) | 7.3% (5.3%,<br>9.3%) | 3,418 (53.9%) | 2,483<br>(51.9%) | 2.0% (0.1%,<br>3.9%) | 5,549 (43.4%) | 3,206<br>(38.5%) | 4.9% (3.5%,<br>6.3%) |
| F | 2,254 (50.1%) | 2,919<br>(57.3%) | -7.3% (-<br>9.3%, -<br>5.3%) | 2,921 (46.1%) | 2,298<br>(48.1%) | -2.0% (-<br>3.9%, -<br>0.1%) | 7,237 (56.6%) | 5,123<br>(61.5%) | -4.9% (-<br>6.3%, -<br>3.5%) |
| U | | | | | | | | | |
| CCI (180<br>Days | | | | | | | | | |
| mean (sd) | 2.62 (2.35) | 3.65 (2.64) | -1.04 (-<br>1.14, -0.94) | 1.61 (1.72) | 2.19 (1.89) | -0.58 (-<br>0.65, -0.51) | 2.17 (2.08) | 2.74 (2.27) | -0.58 (-<br>0.64, -0.52) |
| median<br>[IQR] | 2.00 [1.00,<br>4.00] | 3.00 [2.00,<br>5.00] | | 1.00 [0.00,<br>3.00] | 2.00 [1.00,<br>3.00] | | 2.00 [1.00,<br>3.00] | 2.00 [1.00,<br>4.00] | |

# • Report summary parameters of study population **FEASIBILITY- FOR STUDY OUTCOME**

# • For Apixaban vs Rivaroxaban

| FEASIBILITY FOR STUDY OUTCOME | | | |
|---|---|---|---|
| | Optum CDM IBM® MarketScan® CMS - NOAC | | |
| Number of patients in full cohort | 9,593 | 11,142 | 21,140 |

| Number of patients dropped as incomplete cases | 0 | 0 | 0 |
|---|---|---|---|
| Number of patients that did not begin follow-up | 7 | 22 | 25 |
| Number of patients in analytic cohort | 9,586 | 11,120 | 21,115 |
| Number of events | 172 | 213 | 1,049 |
| Number of person-years | 1,433.02 | 1,933.00 | 3,484.88 |
| Number of patients in group: Rivaroxaban - Comparator | 4,499 | 6,339 | 12,786 |
| Number of patients in group: Apixaban - Exposure | 5,087 | 4,781 | 8,329 |
| Risk per 1,000 patients | 17.94 | 19.15 | 49.68 |
| Rate per 1,000 person-years | 120.03 | 110.19 | 301.01 |

- Report median follow-up time by treatment group
  - For Apixaban vs Rivaroxaban

| FOLLOW-UP TIME FOR STUDY OUTCOME<br>Median Follow-Up Time (Days) [IQR] – At 10 days gap | | | |
|---|---|---|---|
| Patient Group Optum CDM IBM® MarketScan® CMS - NOAC | | | |
| Overall Patient Population | 57 [27, 90] | 79 [38, 90] | 67 [38, 90] |
| Referent - Rivaroxaban | 54 [29, 90] | 68 [38, 90] | 62 [38, 90] |
| Exposure - Apixaban | 61 [18, 90] | 90 [38, 90] | 75 [38, 90] |

- Report reasons for censoring in the overall study population
  - For Apixaban vs Rivaroxaban

| CENSORING REASONS FOR STUDY OUTCOME | | | |
|---|---|---|---|
| Reasons | Optum CDM IBM® MarketScan® CMS | | |
| Outcome | 123 (0.8%) | 187 (0.8%) | 601 (1.4%) |
| Death | 79 (0.5%) | 1 (0.0%) | 459 (1.1%) |

| Start of an additional exposure | 219 (1.5%) | 369 (1.5%) | 682 (1.6%) |
|---|---|---|---|
| End of index exposure | 5,485 (36.6%) | 10,122 (40.6%) | 16,677 (38.5%) |
| Maximum follow-up time reached | 6,595 (44.0%) | 10,590 (42.5%) | 18,372 (42.4%) |
| End of patient data | 0 (0.0%) | 1,218 (4.9%) | 2,779 (6.4%) |
| End of patient enrollment | 427 (2.8%) | 1,455 (5.8%) | 402 (0.9%) |
| DOAC or Warfarin Initiation + Nursing Home Admission | 2,073 (13.8%) | 961 (3.9%) | 3,393 (7.8%) |

• Report overall risk of the primary outcome.

| | Optum CDM | IBM® MarketScan® | CMS - NOAC | Pooled |
|---|---|---|---|---|
| Risk per 1,000 patients | 17.92974044 | 19.11685514 | 49.62157048 | 34.24477612 |

#### 8. Initial Power Assessment

### Aetion report name:

- For Apixaban vs Rivaroxaban
  - Optum CDM <a href="https://bwh-dope.aetion.com/projects/details/1775/rwrs/78120">https://bwh-dope.aetion.com/projects/details/1775/rwrs/78120</a>
  - IBM® MarketScan®- <a href="https://bwh-dope.aetion.com/projects/details/1776/rwrs/78121">https://bwh-dope.aetion.com/projects/details/1776/rwrs/78121</a>
  - CMS NOAC <a href="https://bwh-dope.aetion.com/projects/details/1777/rwrs/78122">https://bwh-dope.aetion.com/projects/details/1777/rwrs/78122</a>

# Date conducted: Updated 01/13/2022

In order to complete the initial power analysis, a dummy outcome indicating a 90-day gap in database enrollment will be used. This outcome is used to ensure that no information on the comparative risks of the outcomes of interest are available at this stage. A 1:1 PS-matched comparative analysis was performed, including age, gender, and CCI score as the only covariates. Power calculations are based on the formulas from Chow et al. (2008).

This emulation is of a trial that is not yet completed. The trial investigators have not published their power calculations. Therefore, we present a range of power calculations for different effect sizes given the feasibility counts and alpha of 0.05. The range in

potential hazard rations come from prior studies in Aryal et al. (2019) comparing bleeding outcomes for apixaban versus rivaroxaban. The target enrollment for the trial is 2,760 patients. We anticipate having around 41,875 patients in our cohort.

### 1. Pooled

| Superiority Analysis - Pooled | | | | | |
|---|---|---|---|---|---|
| Number of patients matched | 32,390 | 32,390 | 32,390 | 32,390 | 32,390 |
| Reference | 16,195 | 16,195 | 16,195 | 16,195 | 16,195 |
| Exposure | 16,195 | 16,195 | 16,195 | 16,195 | 16,195 |
| Risk per 1,000 patients | 34.24477612 | 34.24477612 | 34.24477612 | 34.24477612 | 34.24477612 |
| Alpha (2-sided | 0.05 | 0.05 | 0.05 | 0.05 | 0.05 |
| Desired HR from RCT | 0.8 | 0.7 | 0.6 | 0.5 | 0.4 |
| Number of events expected | 1109.188299 | 1109.188299 | 1109.188299 | 1109.188299 | 1109.188299 |
| Power | 0.960445201 | 0.999965466 | 1 | 1 | 1 |

# 2. Optum CDM

| Superiority Analysis - Optum | | | | | |
|---|---|---|---|---|---|
| Number of patients matched | 12,138 | 12,138 | 12,138 | 12,138 | 12,138 |
| Reference | 6,069 | 6,069 | 6,069 | 6,069 | 6,069 |
| Exposure | 6,069 | 6,069 | 6,069 | 6,069 | 6,069 |
| Risk per 1,000 patients | 8.19945337 | 8.19945337 | 8.19945337 | 8.19945337 | 8.19945337 |
| Alpha (2-sided | 0.05 | 0.05 | 0.05 | 0.05 | 0.05 |
| Desired HR from RCT | 0.8 | 0.7 | 0.6 | 0.5 | 0.4 |
| Number of events expected | 99.524965 | 99.524965 | 99.524965 | 99.524965 | 99.524965 |
| Power | 0.19958509 | 0.4283428 | 0.72176747 | 0.93287238 | 0.99548076 |

# 3. IBM® MarketScan®

| Superiority Analysis - MarketScan | | | | | |
|---|---|---|---|---|---|
| Number of patients matched | 9,016 | 9,016 | 9,016 | 9,016 | 9,016 |
| Reference | 4,508 | 4,508 | 4,508 | 4,508 | 4,508 |
| Exposure | 4,508 | 4,508 | 4,508 | 4,508 | 4,508 |
| Risk per 1,000 patients | 19.11685514 | 19.11685514 | 19.11685514 | 19.11685514 | 19.11685514 |
| Alpha (2-sided | 0.05 | 0.05 | 0.05 | 0.05 | 0.05 |
| Desired HR from RCT | 0.8 | 0.7 | 0.6 | 0.5 | 0.4 |
| Number of events expected | 172.357566 | 172.357566 | 172.357566 | 172.357566 | 172.357566 |
| Power | 0.310539399 | 0.648532959 | 0.918223967 | 0.995201595 | 0.999974911 |

# 4. <u>CMS – NOAC</u>

| Superiority Analysis – CMS NOAC | | | | | |
|---|---|---|---|---|---|
| Number of patients matched | 16,030 | 16,030 | 16,030 | 16,030 | 16,030 |
| Reference | 8,015 | 8,015 | 8,015 | 8,015 | 8,015 |
| Exposure | 8,015 | 8,015 | 8,015 | 8,015 | 8,015 |
| Risk per 1,000 patients | 49.62157048 | 49.62157048 | 49.62157048 | 49.62157048 | 49.62157048 |
| Alpha (2-sided | 0.05 | 0.05 | 0.05 | 0.05 | 0.05 |
| Desired HR from RCT | 0.8 | 0.7 | 0.6 | 0.5 | 0.4 |
| Number of events expected | 795.4337748 | 795.4337748 | 795.4337748 | 795.4337748 | 795.4337748 |
| Power | 0.882335738 | 0.998928865 | 0.999999921 | 1 | 1 |

• Stop analyses until feasibility and power are reviewed by primary investigators and FDA. Reviewers evaluate the results of the analyses described above in Sections 7 and 8, including numbers of patients, patient characteristics, follow-up time, and reasons for censoring by treatment group, as well as overall rates of outcomes and study power. These parameters are re-evaluated and reported in the subsequent sections, after incorporating feedback and refining the protocol.

| Reviewed by PI: | Shirley Wang | Initial Date reviewed: | 08/03/2021 |
|-------------------------|--------------|------------------------|------------|
| Reviewed by FDA: | Ken Quinto | Initial Date reviewed: | 08/18/2021 |
| Reasons for stopping | | | |
| analysis (if required): | | | |

#### 9. Balance Assessment

#### Aetion report name:

- For Apixaban vs Rivaroxaban
  - Optum CDM <a href="https://bwh-dope.aetion.com/projects/details/1775/rwrs/79764">https://bwh-dope.aetion.com/projects/details/1775/rwrs/79764</a>
  - IBM® MarketScan®- <a href="https://bwh-dope.aetion.com/projects/details/1776/rwrs/79768">https://bwh-dope.aetion.com/projects/details/1776/rwrs/79768</a>
  - CMS NOAC https://bwh-dope.aetion.com/projects/details/1777/rwrs/80116

<u>Date conducted:</u> 02/25/2022 and 03/08/2022

After review of initial feasibility and power analyses, complete creation of the remaining covariates from Section 6.2. Again, using the dummy outcome of a 90-day gap in database enrollment, complete a 1:1 PS-matched analysis. The PS should include the complete list of covariates.

- 1. Provide plot of PS distributions stratified by treatment group.
  - a. See Appendix B
- 2. Report covariate balance after matching.
  - a. See Appendix B

\*Data may be omitted to comply with the CMS cell suppression policy

3. Report reasons for censoring by treatment group.

| Censoring Reasons for Study Outcome | | | |
|---|---|---|---|
| Reasons | Overall | Referent | Exposure |
| Death | 439 (1.0%) | 197 (0.8%) | 242 (1.3%) |
| Start of an additional exposure | 609 (1.5%) | 354 (1.5%) | 255 (1.4%) |
| End of index exposure | 15,737 (37.6%) | 9,948 (42.1%) | 5,789 (31.8%) |
| Maximum follow-up time | 18,479 (44.2%) | 9,898 (41.9%) | 8,581 (47.2%) |
| End of patient data | 1,676 (4.0%) | 761 (3.2%) | 915 (5.0%) |
| End of patient enrollment | 1,169 (2.8%) | 660 (2.8%) | 509 (2.8%) |
| DOAC or warfarin initiation + nursing home admission | 3,712 (8.9%) | 1,806 (7.6%) | 1,906 (10.5%) |

4. Report follow-up time by treatment group.

| FOLLOW-UP TIME FOR STUDY OUTCOME<br>Median Follow-Up Time (Days) [IQR] – At 10 days gap | | | |
|---|---|---|---|
| Patient Group Optum CDM IBM® MarketScan® CMS - NOAC | | | |
| Overall Patient Population | 65 [31, 90] | 74 [38, 90] | 67 [38, 90] |
| Referent - Rivaroxaban | 61 [35, 90] | 67 [38, 90] | 62 [34, 90] |
| Exposure - Apixaban | 68 [28, 90] | 88 [38, 90] | 76 [38, 90] |

### 10. Final Power Assessment

Date conducted: 03/08/2022

Re-calculate power in the appropriate excel table, using the revised number of matched patients from the PS-match in Section 9. All other parameters in the table should be the same as in Section 8.

#### 1. Pooled

| Superiority Analysis - Pooled | | | | | |
|---|---|---|---|---|---|
| Number of patients matched | 28,404 | 28,404 | 28,404 | 28,404 | 28,404 |
| Reference | 14,202 | 14,202 | 14,202 | 14,202 | 14,202 |
| Exposure | 14,202 | 14,202 | 14,202 | 14,202 | 14,202 |
| Risk per 1,000 patients | 17.898823 | 17.898823 | 17.898823 | 17.898823 | 17.898823 |
| Alpha (2-sided | 0.05 | 0.05 | 0.05 | 0.05 | 0.05 |
| Desired HR from RCT | 0.8 | 0.7 | 0.6 | 0.5 | 0.4 |
| Number of events expected | 508.398168 | 508.398168 | 508.398168 | 508.398168 | 508.398168 |
| Power | 0.71080316 | 0.98035484 | 0.99992736 | 1 | 1 |

# 2. Optum CDM

| Superiority Analysis - Optum | | | | | |
|---|---|---|---|---|---|
| Number of patients matched | 6,064 | 6,064 | 6,064 | 6,064 | 6,064 |
| Reference | 3,032 | 3,032 | 3,032 | 3,032 | 3,032 |
| Exposure | 3,032 | 3,032 | 3,032 | 3,032 | 3,032 |
| Risk per 1,000 patients | 11.5111765 | 11.5111765 | 11.5111765 | 11.5111765 | 11.5111765 |
| Alpha (2-sided | 0.05 | 0.05 | 0.05 | 0.05 | 0.05 |
| Desired HR from RCT | 0.8 | 0.7 | 0.6 | 0.5 | 0.4 |
| Number of events expected | 69.8037746 | 69.8037746 | 69.8037746 | 69.8037746 | 69.8037746 |
| Power | 0.1539359 | 0.31946556 | 0.56907891 | 0.82526402 | 0.96910355 |

# 3. IBM® MarketScan®

| Superiority Analysis - MarketScan | | | | | |
|-----------------------------------|-------|-------|-------|-------|-------|
| Number of patients matched | 7,388 | 7,388 | 7,388 | 7,388 | 7,388 |
| Reference | 3,694 | 3,694 | 3,694 | 3,694 | 3,694 |
| Exposure | 3,694 | 3,694 | 3,694 | 3,694 | 3,694 |

| Risk per 1,000 patients | 8.02773904 | 8.02773904 | 8.02773904 | 8.02773904 | 8.02773904 |
|---|---|---|---|---|---|
| Alpha (2-sided | 0.05 | 0.05 | 0.05 | 0.05 | 0.05 |
| Desired HR from RCT | 0.8 | 0.7 | 0.6 | 0.5 | 0.4 |
| Desired HR from RCT Number of events expected | <b>0.8</b> 59.308936 | <b>0.7</b> 59.308936 | <b>0.6</b> 59.308936 | <b>0.5</b> 59.308936 | <b>0.4</b> 59.308936 |

# 4. <u>CMS – NOAC</u>

| Superiority Analysis – CMS NOAC | | | | | |
|---|---|---|---|---|---|
| Number of patients matched | 14,952 | 14,952 | 14,952 | 14,952 | 14,952 |
| Reference | 7,476 | 7,476 | 7,476 | 7,476 | 7,476 |
| Exposure | 7,476 | 7,476 | 7,476 | 7,476 | 7,476 |
| Risk per 1,000 patients | 27.146628 | 27.146628 | 27.146628 | 27.146628 | 27.146628 |
| Alpha (2-sided | 0.05 | 0.05 | 0.05 | 0.05 | 0.05 |
| Desired HR from RCT | 0.8 | 0.7 | 0.6 | 0.5 | 0.4 |
| Number of events expected | 405.896382 | 405.896382 | 405.896382 | 405.896382 | 405.896382 |
| Power | 0.61328522 | 0.94876319 | 0.99927824 | 0.99999974 | 1 |

• Stop analyses until balance and final power assessment are reviewed by primary investigators, FDA, and assigned members of advisory board.

| Reviewed by PI: | Date reviewed: |
|-------------------------|----------------|
| Reviewed by FDA: | Date reviewed: |
| Reasons for stopping | |
| analysis (if required): | |

# **11. Study Confidence and Concerns**

# <u>Deadline for voting on study confidence and listing concerns:</u> Date votes and concerns are summarized:

- If final feasibility and power analyses are reviewed and approved, proceed to the remaining protocol steps.
- All study team and advisory board members that review this protocol should at this stage provide their level of confidence for the
  success of the RWD study in the Google Form. This form also provides space for reviewers to list any concerns that they feel may
  contribute to a failure to replicate the findings of the RCT, including differences in study populations, poor measurement of study
  variables, or residual confounding. All responses will be kept confidential and individual-level results will only be shared with the
  individual respondent.
- After the deadline for voting has passed, provide the distribution of responses and summarize all concerns here.

### 12. Register study protocol on clinicalTrials.gov

#### Date conducted:

Register the study on clinicalTrials.gov and upload this document.

### 13. Comparative Analyses

Aetion report name:

Date conducted:

- 13.1 For primary analysis:
- 13.2 For sensitivity analyses:

### 14. Requested Results

14.1 Table 1: Baseline characteristics before and after adjustment

| Variable | Before adjustment | | | After adjustment | | |
|---|---|---|---|---|---|---|
| | Referent | Exposure | Std. diff. | Referent | Exposure | Std. diff. |
| Number of patients | | | - | | | - |
| Age categories | | | | | | |

# 14.2 <u>Table 2: Follow-up time</u>

| Patient Group | Median Follow-Up Time (Days) [IQR] |
|----------------------------|------------------------------------|
| Overall Patient Population | |
| Referent | |
| Exposure | |

# 14.3 <u>Table 3: Censoring events</u>

| | Overall | Referent | Exposure |
|---------------------------------|---------|----------|----------|
| Outcome | | | |
| Death | | | |
| Start of an additional exposure | | | |
| End of index exposure | | | |
| Specified date reached | | | |
| End of patient data | | | |
| End of patient enrollment | | | |

# 14.4 <u>Table 4: Results from primary analyses;</u>

| Analysis | No. exposed events | No. referent events | Exposed rate | Referent rate | HR (95% CI) |
|---|---|---|---|---|---|
| Crude | | | | | |

| Analysis 1 |
|------------|
| Analysis 2 |

HR, Hazard Ratio; CI, Confidence Interval.

# 14.5 Table 5: Results from secondary analyses;

### 15. References

Chow S, Shao J, Wang H. 2008. Sample Size Calculations in Clinical Research. 2nd Ed. Chapman & Hall/CRC Biostatistics Series. page 177

Madan Raj Aryal, Rohit Gosain, Anthony Donato, Han Yu, Anjan Katel, Yashoda Bhandari, Rashmi Dhital, Peter A. Kouides; Systematic review and meta-analysis of the efficacy and safety of apixaban compared to rivaroxaban in acute VTE in the real world. *Blood Adv* 2019; 3 (15) 2381 – 2387, doi: https://doi.org/10.1182/bloodadvances.2019000572.

| | 000004 VMT - 1 1 1 6 VV | to other control or to another con- | noferon (not) and | |
|---|---|---|---|---|
| | COBRRA - VTE trial definitions | Implementation in routine care Hease see the following Google Drive for Earther details or any missing information: https://drive.google.com/drive/folders/1VDG18-wyw/f6xt/ft/tost-VCnb68-gt/hap-sharing | References/Rationale | Color coding |
| | | ICD-10 codes are not listed in this decement because of exect cell size limitations and excessive number of ICD-10 codes. Full ICD-10 code first will be available in the above Google Drive Folder (link above). ICD-9 to ICD-10 code conversions were completed using a SAS macros that implements forward/backward mapping based on the CMS ICD-9 to ICD-10 mapping | | |
| | | TRIAL DETAILS EXPOSURE vs. COMPARISON | | Can be replicated in claims |
| | Apixaban 10 mg PO BID for 1 week, then 5 mg PO BID for 3 months of treatment vs. Novacreaban 15 mg PO BID for 3 weeks, then 20 mg PO OD for 3 months of treatment | Aginahan Al generic Vs. Warroundur Al generic | | Using dummy definitions for<br>measuring in claims |
| | Rivaroxaban 15 mg POBID for 3 weeks, then 20 mg PO OD for 3 months of treatment | PRIMARY OUTCOME | | Can't be measured in claims |
| | The rate of adjudicated clinically relevant bleeding (CRB) events (Time Frame: For the duration of the study: 3 months) - CRB events are | Major Meeding:<br>See "Major Weeding" Sheet | Graham DJ, Reichman ME, Wennecke M, et al. Stroke,<br>Bleeding, and Mortality Risks in Elderly Medicare<br>Beneficiaries Treated With Dabigatran or<br>Rivaroxaban for Nonvalvular Afrial Fibrillation. JAMA | Can't be measured in claims<br>but not important for the<br>analysis |
| | The rate of adjudicated clinically relevant blending (CRB) events [Time Frame: For the duration of the study: 3 months] - CRB events are defined as the composite of major blending (MB) events and clinically relevant non-major blending (CRRMS) events. | Measured (0,90) in an inpatient setting in any diagnoses position (transfusion codes NOT included for non-critical sites) | | but not important for the<br>analysis |
| | | Clinically Balesont Mon Major Meeding Frents:<br>See there "CANA filends" | doi:10.1001/jamainternmed.2016.5954 | |
| ı | | INCLUSION CRITERIA | | |
| | | Measured [-14, 0] in any diagnosis position in an inputient setting: Pulmonary Embolism: | | |
| | | Pulmonary Inholium:<br>CDB Pulmonic 415.1,415.10,415.11,415.12,415.13,415.5,415.16,415.17,415.19,415.199<br>CDB Diagnosis 15.6,16.63,176.02,16.69,16.69,16.69,16.690 | | |
| 1 | Confirmed newly diagnosed symptomatic acute VTE (proximal power extremity DVT or segmental or greater PE) | <u>Proximal DVT</u><br>ICD-0 diagnosis: 451.1x, 451.2x, 451.81, 451.9x, 453.1x, 453.2x, 453.8x, 453.9x, 453.40, 453.41, 453.42, 453.0 | | |
| | | 100-10-diagnosis: 80.1°, 180.2, 180.3, 180.9, 182.0, 182.1, 182.2° (EXCEPT 182.2.1), 182.4°, 182.80, 182.90, 182.81°, 18 | | |
| 2 | Age >= 18 years | Age>=18 | | |
| | Informed consent obtained | N/A EXCLUSION CRITERIA | | |
| | Have received >72 hours of thereapeutic anticoagulation | EXCLUSION CRITERIA Measured (-180, 0) in prexription claims | | |
| 1 | nave receives >/ 2 nours or tree-expectic annicologisation | Prior vas of a DOAC or Warfarin:<br>Apixaban, Rivaroxaban, Dabigatran, Edoxaban, or Warfarin | | |
| | | Measured [-180, 0 ] in any diagnosis position and inpatient or outpatient care setting | | |
| 2 | Creatine clearance < 30 ml/min calculated with the Cockcroft-Gault formula | COL ADM CONTROL SECTION COLD COLUMN SECTION SECTION SECTION COLD COLUMN SECTION SECTION SECTION COLD COLUMN SECTION SECTION COLUMN SECTION SECTION SECTION COLUMN SECTION COLUMN SECTION SECTION COLUMN SECTION C | | |
| | | Dishipsi/Namai Transplant San Shote "Dulysis and Renal Transplant" | | |
| | | Seed Sneed. Unaryous area wereas in remoperabils." | | |
| 3 | Any contradiction for anticoagulation with apixaban or rivaroxaban as determined by the treating physician such as, but not limited to<br>one of the following: | | | |
| | ······································ | Messared [-180, 0] in an inpatient, any diagnosis position (transfusion codes required for non-critical sites) | | |
| | | Major Beeding: Sheet | Graham DJ, Reichman ME, Wernecke M, et al. Stroke, | |
| | 1) Active Bleeding | Sao "Major Monding" Sheet Measured (-180, 0) in an inpatient, any diagnosis position (transfusion codes NOT required for non-critical sites) | Bleeding, and Mortality Risks in Elderly Medicare<br>Beneficiaries Treated With Dabigatran or | |
| • | a practite intending | measureq (-160, u) in an inparient, any originate position granisassion codes incu required for non-critical steely Clinically Relevant Non-Major Bleading Events: | Rivaroxaban for Nonvalvular Atrial Fibrillation. JAMA<br>Intern Med. 2016;176(11):1662–1671.<br>doi:10.1001/jamainternmed.2016.5954 | |
| | | See "CRNM Bleeds Sheet" | 60.10.1001/janamammad.1010.3934 | |
| | | Measured [-180, 0] in any diagnosis position in an inpatient or outpatient setting | | |
| 5 | 2) Active maligrancy, defined as all diagnosed with cancer within the past 6 months; or b) recurrent, regionally advanced or metabatic<br>disease, or c) currently receiving treatment or have received any treatment for cancer during the 6 months prior to randomization; or d)<br>a hernatologic malignancy not in complete remission | Cancer. (20 Juny 1997) 140 - 290 x (perspt 209 4x, 209 5x, 209 6x) (20 Juny 1997) 140 - 290 x (perspt 209 4x, 209 5x, 209 6x) (20 Juny 1997) 140 - 290 x (perspt 209 4x, 209 5x, 209 6x) (20 Juny 1997) 140 - 290 x (perspt 209 4x, 209 5x, 209 6x) | | |
| | a hematologic malignancy not in complete remission | For fall list, see "Cancer Sheet" | | |
| 6 | 3) Westgefer > 2-20 kg | THE STATE OF THE S | | |
| 7 | O Liver Classes (Child-Pugh Class Ser C) | Memoral (1,80) in ordinary supportant to interpolate to educate the education testing<br>September 11, 11 | | |
| | | Measured (-190,0) in prescription claims | | |
| | | Stong CPD44 hishibror/Inducacy hishibror/ Kindoccy hishibror/ Kindoccy hishibror/ Kindoccy hishibror/ Kindoccy hishibror/ | | |
| 8 | 5) Use of contraindicated medications | P-sp inhibitors/Indusers: | https://depts.wishington.edu/anticoleg/home/cont<br>ent/apixaban | |
| | | cobicistat, conivaptan, tipranavir | CYP3A's Copied from PLATO: https://bwh-<br>dope.aetion.com/measures/details/211908/948/0/t | |
| | | Measurerd [-180, 0] in any diagnosis position in an inpatient or cupatient setting | emplates/simpleEventSet?&tab=0 | |
| | | mediate last plans, year or anguno promo un meruparan menung<br>darian Herialdusi.<br>(202 Diagnoni, 427.3, 427.3), 427.32 | | |
| 9 | 6) Another indication for long-term anticoagulation (eg. atrial fibrillation) | Co. 10 (Co. 10 | | |
| | | (Ch.10 Dispensio: 255.2 Measured (-150.0) in perdiamosis position and insatient and outstailent care setting | | |
| 10 | | Premincy | | |
| | 7) Pregnancy | See Througharty Shoet Measured [-180, 0] in prescription claims | | |
| 11 | 8) Dual Antiplatelet Use | De el Antiplatet: Ney of the following colonizazol, dipyridamole, ticlopidine MC, apprin, clopidignel bisulfate, prassigni MC, ticlopidin, apprin, dipyridamole, exetimibe | | |
| | | Measured (180.0) in any diamous position and inpatient and outsident are setting | | |
| | | мешитео (-100, у) in any ожуговы розвого апо этрыхняті ато октрывать сага затоля<br><u>Совриборатіну:</u> | | |
| | 9) Coagul opathy | CO-9 Chipmonic 286, 286.1, 286.4, 286.5, 286.5, 286.53, 286.53, 286.59, 287.5, 286.0, 286.2, 286.5, 286.6, 286.7, 286.9, 287.2, 287.3, 287.4<br>CO-10 Chipmonic D67, D68, D68.1, D68.2, D68.3, D68.31, D68.311, D68.312, D68. | | |
| | | CLC-12 UIRROWN: UR1, UR6.1, UR6.1, UR6.1, UR6.1, UR6.1, UR6.11, UR6.11, UR6.11, UR6.11, UR6.2, UR6.01, | | |
| 12 | | | | |



**Information from Trial** 

<u>Trial Name:</u> COBBRA clinicaltrials.gov/ct2/show/NCT0462430

**NCT**: NCT04642430

Therapeutic Area: Cardiology

RCT Category: Equivalence/Superiority

Brand Name: Eliquis and Xarelto

Generic Name: Apixaban and Rivaroxaban

Sponsor: Ottwa Hospital Research Institute

Year: 2020 - Present

Measurable Endpoint: Major Bleeding

Exposure: Apixaban

Comparator: Rivaroxaban

**Populuation:** Men and women ages 18 and older presenting with acute VTE

No. of Patients: 3,018

Power: TBD

#### ICD-9 Dx 336.1 VASCULAR MYELOPATHIES 363.61 CHOROIDAL HEMORRHAGE UNSPECIFIED 363.62 EXPULSIVE CHOROIDAL HEMORRHAGE 376 32 ORBITAL HEMORRHAGE 377.42 HEMORRHAGE IN OPTIC NERVE SHEATHS 379 23 VITREOUS HEMORRHAGE 431 INTRACEREBRAL HEMORRHAGE 432 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE 432 NONTRAUMATIC EXTRADURAL HEMORRHAGE 432. SUBDURAL HEMORRHAGE 432.9 UNSPECIFIED INTRACRANIAL HEMORRHAGE 719. **HEMARTHROSIS** 719.1 HERARTHROSIS INVOLVING SHOULDER REGION 719.12 HEMARTHORSIS INVOLVING UPPER ARM 719.14 HEMARTHROSIS INVOLVING HAND 719.15 HEMARTHROSIS INVOLVING PELVIC REGION AND THIGH 719.17 HEMARTHROSIS INVOLVING ANKLE AND FOOT 719.19 HEMARTHROSIS INVOLVING MULTIPLE SITES 729.92 NONTRAUMATIC HEMATOMA OF SOFT TISSUE 852 SUBARACHNOID SUBDURAL AND EXTRADURAL HEMORRHAGE FOLLOWING INJURY 852 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH STATE OF CONSCIOUSNESS UNSPECIFIED 852.01 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH NO LOSS OF CONSCIOUSNESS 852 03 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH MODERATE (1 - 24 HOURS) LOSS OF CONSCIOUSNESS) 852.05 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS WITHOUT RETURN TO PRE-EXISTING CONSCIOUS LEVEL 852.06 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH LOSS OF CONSCIOUSNESS OF UNSPECIFIED DURATION 852.09 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH CONCUSSION UNSPECIFIED 852.1 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH STATE OF CONSCIOUSNESS UNSPECIFIED 852.11 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH NO LOSS OF CONSCIOUSNESS 852.12 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH BRIEF (LESS THAN ONE HOUR) LOSS OF CONSCIOUSNESS 852.15 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS WITHOUT RETURN TO PRE-EXISTING CONSCIOUS LEVEL 852.19 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH CONCUSSION UNSPECIFIED 852.2 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH STATE OF CONSCIOUSNESS UNSPECIFIED 852.22 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH BRIEF (LESS THAN ONE HOUR) LOSS OF CONSCIOUSNESS SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS WITHOUT RETURN TO PRE-EXISTING CONSCIOUS LEVEL 852.25 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND 852.3 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH STATE OF CONSCIOUSNESS UNSPECIFIED 852.3 852.31 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH NO LOSS OF CONSCIOUSNESS 852.32 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH BRIEF (LESS THAN ONE HOUR) LOSS OF CONSCIOUSNESS SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH MODERATE (1-24 HOURS) LOSS OF CONSCIOUSNESS 852.33 852.34 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS AND RETURN TO PRE-EXISTING CONSCIOUS LEVEL 852.35 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS WITHOUT RETURN TO PRE-EXISTING CONSCIOUS LEVEL 852.42 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH BRIEF (LESS THAN 1 HOUR) LOSS OF CONSCIOUSNESS 852.43 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH MODERATE 852.45 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS WITHOUT RETURN TO PRE-24 HOURS) LOSS OF CONSCIOUSNESS-EXISTING CONSCIOUS LEVEL 852.49 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH CONCUSSION UNSPECIFIED 852.54 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS AND RETURN TO PRE-EXISTING CONSCIOUS LEVEL OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH STATE OF CONSCIOUSNESS UNSPECIFIED 853 01 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH NO LOSS OF CONSCIOUSNESS OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH MODERATE (1-24 HOURS) LOSS OF CONSCIOUSNESS 853 04 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS AND RETURN TO PRE-EXISTING CONSCIOUS LEVEL 853.05 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS WITHOUT RETURN TO PRE-EXISTING CONSCIOUS LEVEL 853 1 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND 853.11 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH NO LOSS OF CONSCIOUSNESS 853 12 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH BRIEF (LESS THAN ONE HOUR) LOSS OF CONSCIOUSNESS 853.13 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH MODERATE (1-24 HOURS) LOSS OF CONSCIOUSNESS 853.14 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS AND RETURN TO PRE-EXISTING CONSCIOUS LEVEL 853.15 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS WITHOUT RETURN TO PRE-EXISTING CONSCIOUS LEVEL 866.02 LACERATION OF KIDNEY WITHOUT OPEN WOUND INTO CAVITY

363.72 HEMORRHAGIC CHOROIDAL DETACH HEMOPERICARDIUM SUBARACHNOID HEMORRHAGE 568.81 HEMOPERITONEUM (NONTRAUMATIC) 719.1 HEMARTHROSIS SITE UNSPECIFIED 719.13 HEMARTHROSIS INVOLVING FOREARM HEMARTHROSIS INVOLVING LOWER LEG 719.16 719.18 HEMARTHROSIS INVOLVING OTHER SPECIFIED SITES 852 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT MENTION OF OPEN INTRACRANIAL WOUND 852.02 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH BRIEF (LESS THAN ONE HOUR) LOSS OF CONSCIOUSNESS SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS AND RETURN TO PRE-EXISTING CONSCIOUS LEVEL 852.04 852. SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND 852.13 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH MODERATE (1-24 HOURS) LOSS OF CONSCIOUSNESS 852.14 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS AND RETURN TO PRE-EXISTING CONSCIOUS LEVEL 852.16 SUBARACHNOID HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH LOSS OF CONSCIOUSNESS OF UNSPECIFIED DURATION 852. SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT MENTION OF OPEN INTRACRANIAL WOUND 852.21 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH NO LOSS OF CONSCIOUSNESS 852.23 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH MODERATE (1-24 HOURS) LOSS OF CONSCIOUSNESS 852.24 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS AND RETURN TO PRE-EXISTING CONSCIOUS LEVEL 852.26 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH LOSS OF CONSCIOUSNESS OF UNSPECIFIED DURATION SUBDURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH CONCUSSION UNSPECIFIED 852.29 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH LOSS OF CONSCIOUSNESS OF UNSPECIFIED DURATION 852.36 SUBDURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH CONCUSSION UNSPECIFIED 852.39 852.4 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT MENTION OF OPEN INTRACRANIAL WOUND 852.4 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH STATE OF CONSCIOUSNESS UNSPECIFIED 852.41 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH NO LOSS OF CONSCIOUSNESS EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS AND RETURN TO PRE-EXISTING CONSCIOUS LEVEL 852.44 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH LOSS OF CONSCIOUSNESS OF UNSPECIFIED DURATION 852.46 852.5 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND 852.5 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH STATE OF CONSCIOUSNESS UNSPECIFIED EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH NO LOSS OF CONSCIOUSNESS 852.51 852.52 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH BRIEF (LESS THAN ONE HOUR) LOSS OF CONSCIOUSNESS 852.53 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH MODERATE (1-24 HOURS) LOSS OF CONSCIOUSNESS EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH PROLONGED (MORE THAN 24 HOURS) LOSS OF CONSCIOUSNESS WITHOUT RETURN TO PRE-EXISTING CONSCIOUS LEVEL EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH LOSS OF CONSCIOUSNESS OF UNSPECIFIED DURATION 852 59 EXTRADURAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH CONCUSSION UNSPECIFIED OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT MENTION OF OPEN INTRACRANIAL WOUND 853.02 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH BRIEF (LESS THAN ONE HOUR) LOSS OF CONSCIOUSNESS 853.06 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH LOSS OF CONSCIOUSNESS OF UNSPECIFIED 853.09 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITHOUT OPEN INTRACRANIAL WOUND WITH CONCUSSION UNSPECIFIED 853 1 OTHER AND LINSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INLIRY WITH OPEN INTRACRANIAL WOLIND WITH STATE OF CONSCIOUSNESS LINSPECIFIED 853 16 OTHER AND LINSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INILIRY WITH OPEN INTRACRANIAL WOLLD WITH LOSS OF CONSCIOUSNESS OF LINSPECIFIED DURATION 853 19 OTHER AND UNSPECIFIED INTRACRANIAL HEMORRHAGE FOLLOWING INJURY WITH OPEN INTRACRANIAL WOUND WITH CONCUSSION UNSPECIFIED 866.01 HEMATOMA OF KIDNEY WITHOUT RUPTURE OF CAPSULE WITHOUT OPEN WOUND INTO CAVITY 866.11 HEMATOMA OF KIDNEY WITHOUT RUPTURE OF CAPSULE WITH OPEN WOUND INTO CAVITY 866.12 LACERATION OF KIDNEY WITH OPEN WOUND INTO CAVIT The occurrence of Inpatient Confinement with the following attributes: **Procedure** Confinement Position) s any of: { "99.05", "99.03", "99.04", "99.06" }

Code (Any

99.05 TRANSFUSION OF PLATELETS

99.03 OTHER TRANSFUSION OF WHOLE BLOOD

99.04 TRANSFUSION OF PACKED CELLS

TRANSFUSION OF COAGULATION FACTORS

AND ICD-9 Dx

| 455.1 INTERNAL THROMOSCED HEMORRHOIDS 455.8 UNSPECIFIED THROMOSCED HEMORRHOIDS 455.8 UNSPECIFIED THROMOSCED HEMORRHOIDS 455.9 RESULULA HEMORRHOIDS WITH OTHER COMPLICATION 459. PRESULULA HEMORRHOIDS WITH OTHER COMPLICATION 459. PRESULULA HEMORRHOIDS WITH OTHER COMPLICATION 450.1 ESOPHAGITIS 530.1 ESOPHAGITIS 530.1 ESOPHAGITIS 530.1 SON THE RESOPHAGITIS 530.13 FOR THE SOPHAGITIS 530.3 FOR THE SOPHAGITIS 530.3 FOR THE SOPHAGITIS 530.13 FOR THE SOPHAGITIS 530.13 FOR THE SOPHAGITIS 530.13 FOR THE SOPHAGITIS 530.14 ESOPHAGITIS WITH HEMORRHAGE SYNDROME 530.20 ESOPHAGIA LEUGER WITH HEMORRHAGE SYNDROME 530.20 ESOPHAGIA LEUGER WITH HEMORRHAGE WITH OBSTRUCTION 531.2 ACLITE CASTRIC LUCER WITH HEMORRHAGE WITH OBSTRUCTION 531.2 ACLITE CASTRIC LUCER WITH HEMORRHAGE WITH OBSTRUCTION 531.2 ACLITE CASTRIC LUCER WITH HEMORRHAGE WITH OBSTRUCTION 531.3 ACLITE GASTRIC LUCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.4 CHORNOC ON LUSSPECIFIC OBSTRUCLUCE WITH HEMORRHAGE OF PERFORATION 531.6 CHORNOC ON LUSSPECIFIC OBSTRUCLUCE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.6 CHORNOC ON LUSSPECIFIC OBSTRUCLUCE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.6 CHORNOC ON LUSSPECIFIC OBSTRUCLUCE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.6 CHORNOC ON LUSSPECIFIC OBSTRUCLUCE WITH HEMORRHAGE OF PERFORATION WITHOUT OBSTRUCTION 531.6 CHORNOC ON LUSSPECIFIC OBSTRUCLUCE WITH HEMORRHAGE OF PERFORATION 531.6 CHORNOC ON LUSSPECIFIC OBSTRUCLUCE WITH HEMORRHAGE OF PERFORATION 531.6 CHORNOC ON LUSSPECIFIC OBSTRUCLUCE WITH HEMORRHAGE OF PERFORATION 532.1 ACUTE DUDOPHAU LUCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 532.1 ACUTE DUDOPHAU LUCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.2 ACUTE DUDOPHAU LUCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.2 ACUTE DUDOPHAU LUCER WITH HEMORRHAGE WITH OBSTRUCTION 533.2 CHORNOC OR SURSPECIFIED DES COUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 533.2 ACUTE DUDOPHAU LUCER WITH HEMORRHAGE WITH DESPORATION 533.2 ACUTE DUDOPHAU LUCER WITH HEMORRHAGE WITH DESPORATION 533.3 | | |
|---|---|---|
| MSSPECIFIED HEMORRHOODS WITH OTHER COMPLICATION | | |
| ## ASSOCIATION NOT CONTRICT OF THE PROPORTION OF THE MORRHAGE UNSPECIFIED AS ACUTE OR CHRONOL WITH DESTRUCTION ## STATE OF THE PROPORTION OF THE PROPORTION OF THE MORRHAGE OR PERFORATION ## STATE OF THE PROPORTION OF THE PROPORTION OF THE MORRHAGE AND PERFORATION OF THE PROPORTION OF THE PR | | |
| ## HEMORRHAGE UNSPECIFIED \$30.11 EOPHAGITIS \$0.2011 BORNHAGE UNSPECIFIED \$0.31.12 EOSHOPHAGITIS \$0.31.21 EOSHOPHAGITIS \$0.31.31 EOSHOPHAGITIS \$0.31.31 EOSHOPHAGITIS \$0.31.32 EOSHOPHAGITIS \$0.31.32 EOSHOPHAGITIS \$0.32.21 EOSHOPHAGITIS \$0.32.22 EOSHOPHAGITIS \$0.33.21 GASTROESOPHAGEAL LACERATION-HEMORRHAGE SYNDROME \$0.32.22 EOSHOPHAGEAL HEMORRHAGE \$0.31.22 ACUTE GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION \$0.31.21 ACUTE GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION \$0.31.21 ACUTE GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION \$0.31.21 ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION \$0.31.21 ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION \$0.31.21 ACUTE GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION \$0.31.22 ACUTE GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION \$0.31.24 CHORNIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION \$0.31.25 CHORNIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION \$0.31.26 CHORNIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE OR PERFORATION WITH OBSTRUCTION \$0.31.26 CHORNIC OR UNSPECIFIED AS ACUTE OR CRONIC WITHOUT WENTON OF HEMORRHAGE OR PERFORATION \$0.31.26 CHORNIC OR UNSPECIFIED AS ACUTE OR CRONIC WITHOUT WENTON OF HEMORRHAGE OR PERFORATION \$0.31.26 CHORNIC OR UNSPECIFIED AS ACUTE OR CRONIC WITHOUT WENTON OF HEMORRHAGE OR PERFORATION \$0.31.26 CHORNIC OR UNSPECIFIED AS ACUTE OR CRONIC WITHOUT WENTON OF HEMORRHAGE OR PERFORATION \$0.32.26 CHORNIC OR UNSPECIFIED AS ACUTE OR CRONIC WITHOUT WENTON OF HEMORRHAGE OR PERFORATION \$0.32.26 CHORNIC OR UNSPECIFIED STEW WITH HEMORRHAGE WITH OBSTRUCTION \$0.32.26 CHORNIC OR | | |
| SODIAGITS SOLIDATION OTHER ESOPHAGITS ACUTE GASTRIC ULCER WITH HEMORRHAGE SOLIDATE ACUTE GASTRIC ULCER WITH HEMORRHAGE SOLIDATE ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION ACUTE ON UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION ACUTE ON UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION ACUTE OUDDROAD ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION WITHOUT OBSTRUCTION ACUTE OUDDROAD ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION WITHOUT OBSTRUCTION ACUTE OUDDROAD ULCER WITH HEMORRHAGE ACUTE OUT ON A WITHOUT OBSTRUC | | |
| SOOPHAGTIS UNSPECIFIED SOOTHER ESOPHAGTIS SOOTHING SOOTHER ESOPHAGTIS SOOTHING SO | | |
| 530.15 530.17 530.27 530.28 530.39 530.30 53 | | |
| 30.17 SASTROSOPHAGEAL LACERATION-HEMORRHAGE SYNDROME 30.28 ESOPHAGEAL HEMORRHAGE 30.10 ACUTE GASTRIC LICER WITH HEMORRHAGE WITH OBSTRUCTION 30.11 ACUTE GASTRIC LICER WITH HEMORRHAGE WITH OBSTRUCTION 30.12 ACUTE GASTRIC LICER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 30.13 ACUTE GASTRIC LICER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 30.14 CAUTE GASTRIC LICER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 30.15 ACUTE GASTRIC LICER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 30.16 CHRONIC OR UNSPECIFIED GASTRIC LICER WITH HEMORRHAGE WITHOUT OBSTRUCTION 30.17 CHRONIC OR UNSPECIFIED GASTRIC LICER WITH HEMORRHAGE WITHOUT OBSTRUCTION 30.18 CHRONIC OR UNSPECIFIED GASTRIC LICER WITH HEMORRHAGE WITHOUT OBSTRUCTION 30.19 CHRONIC OR UNSPECIFIED GASTRIC LICER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 30.10 CHRONIC OR UNSPECIFIED GASTRIC LICER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 30.10 CHRONIC CONTROL WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 30.11 CHRONIC OR UNSPECIFIED AS ACUTE OF CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 30.12 CHRONIC OR UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 30.13 CAUTE DUDOPNAL LICER WITH HEMORRHAGE WITH DUSTRUCTION 30.14 CAUTE DUDOPNAL LICER WITH HEMORRHAGE WITH DUSTRUCTION 30.15 CHRONIC OR UNSPECIFIED DUDOPNAL LICER WITH HEMORRHAGE WITH OBSTRUCTION 30.16 CHRONIC OR UNSPECIFIED DUDOPNAL LICER WITH HEMORRHAGE WITH OBSTRUCTION 30.17 CHRONIC OR UNSPECIFIED DUDOPNAL LICER WITH HEMORRHAGE WITH OBSTRUCTION 30.18 CHRONIC OR UNSPECIFIED DUDOPNAL LICER WITH HEMORRHAGE WITH OBSTRUCTION 30.19 CHRONIC OR UNSPECIFIED SET WITH HEMORRHAGE WITH OBSTRUCTION 30.10 CHRONIC OR UNSPECIFIED SET WITH HEMORRHAGE WITH OBSTRUCTION 30.10 CHRONIC OR UNSPECIFIED SET WITH HEMORRHAGE WITH DEMORRHAGE WITHOUT OBSTRUCTION 30.10 CHRONIC OR UNSPECIFIED SET WITH HEMORRHAGE WITHOUT OBSTRUCTION 30.10 CHRONIC OR UNSPECIFIED SET WITH HEMORRHAGE WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 30.10 CHRONIC OR UNSPECIFIED SET WITH HEMORRHAGE WITHOUT ME | | |
| Sa30.82 ESOPHAGEAL HEMORRHAGE SONAGE ESOPHAGEAL HEMORRHAGE SONAGE ACUTE GASTRIC ULCER WITH HEMORRHAGE SYNDROME S13.10.1 ACUTE GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION S13.12.1 ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION S13.12.1 ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT SISTRUCTION S13.12.1 ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION CHRONIC OR ULSPECHIED GASTRIC ULCER WITH HEMORRHAGE OR PERFORATION CHRONIC OR ULSPECHIED GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION S13.15.1 CHRONIC OR ULSPECHIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION S13.10.1 CHRONIC OR ULSPECHIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION S13.10.1 CHRONIC OR ULSPECHIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION S13.10.1 CHRONIC GASTRIC ULCER WITHOUT OF HEMORRHAGE OR PERFORATION WITHOUT OBSTRUCTION S13.10.2 CHRONIC GASTRIC ULCER WITHOUT OF HEMORRHAGE OR PERFORATION ACUTE DUDOBNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION S13.1 ACUTE DUDOBNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION CHRONIC OR ULSPECHIED SUBJECT WITH HEMORRHAGE OR PERFORATION CHRONIC OR ULSPECHIED SUBJECT WITH HEMORRHAGE OR PERFORATION CHRONIC OR ULSPECHIED DUDOBNAL ULCER WITH PERFORATION CHRONIC OR ULSPECHIED SUBJECT WITH HEMORRHAGE OR PERFORATION CHRONIC OR ULSPECHIED SUBJECT WITH HEMORRHAGE OR PERFORATION CHRONIC OR ULSPECHIED SUBJECT WITH HEMORRHAGE AND PERFORATION CHRONIC OR ULSPECHIED GASTRUCIUM ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION CHRONIC OR ULSPECHIED GASTRUCIUM ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION CHRONIC OR ULSPECHIED GAST | | |
| SOPHAGEAL HEMORRHAGE 531 ACUTE GASTRIC LUCER WITH HEMORRHAGE WITH OBSTRUCTION 531.2 ACUTE GASTRIC LUCER WITH HEMORRHAGE WITH OBSTRUCTION 531.2 ACUTE GASTRIC LUCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.3 ACUTE GASTRIC LUCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.4 CARRIEG GASTRIC LUCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.5 CHORNIC OR UNSPECIFIED GASTRIC LUCER WITH HEMORRHAGE OR PERFORATION 531.6 CHORNIC OR UNSPECIFIED GASTRIC LUCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 531.6 CHORNIC OR UNSPECIFIED GASTRIC LUCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.7 CHORNIC OR UNSPECIFIED GASTRIC LUCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.8 CHORNIC OR UNSPECIFIED GASTRIC WICER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 532.1 CHORNIC CORRESPONDED ASSEMBLY OF A CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 532.2 CHORNIC CASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 532.3 CHORNIC DUDOENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 532.4 CHORNIC OR UNSPECIFIED SA CAUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 532.5 CHORNIC OR UNSPECIFIED DUDOENAL ULCER WITH HEMORRHAGE OR PERFORATION 532.6 CHORNIC OR UNSPECIFIED DUDOENAL ULCER WITH HEMORRHAGE OR PERFORATION 533.1 CHORNIC OR UNSPECIFIED DUDOENAL ULCER WITH HEMORRHAGE OR PERFORATION 533.2 CHORNIC OR UNSPECIFIED SET WITH PERFORATION 533.3 CHORNIC OR UNSPECIFIED SET WITH PERFORATION 533.4 CUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.5 CHORNIC OR UNSPECIFIED SET WITH PERFORATION 534.6 CHORNIC OR UNSPECIFIED SET WITH PERFORATION 535.5 CHORNIC OR UNSPECIFIED SET WITH HEMORRHAGE AND PERFORATION 536.6 CHORNIC OR UNSPECIFIED SET WITH HEMORRHAGE AND PERFORATION 537.6 CHORNIC OR UNSPECIFIED SET WITH HEMORRHAGE AND PERFORATION 538.6 CHORNIC OR UNSPECIFIED SET WITH HEMORRHAGE AND PERFORATION 539.7 CHORNIC OR UNSPECIFIED SET WITH HEMORRHAGE WITHOUT OBSTRUCTION 539.7 CHORNIC OR UNSPECIFIED SET WITH HEMORRHAGE WI | | |
| ACUTE GASTRIC LUCER WITH HEMORRHAGE ACUTE GASTRIC LUCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 33.1.2 ACUTE GASTRIC LUCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 33.1.3 ACUTE GASTRIC LUCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 33.1.3 ACUTE GASTRIC LUCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 33.1.5 CHONIC OR UNSPECIFIED GASTRIC LUCER WITH HEMORRHAGE OR PERFORATION 33.1.6 CHONIC OR UNSPECIFIED GASTRIC LUCER WITH PERFORATION 33.1.7 CHONIC OR UNSPECIFIED GASTRIC LUCER WITH PERFORATION 33.1.7 CHONIC OR UNSPECIFIED GASTRIC LUCER WITH PERFORATION 33.1.7 CHONIC OR UNSPECIFIED GASTRIC LUCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 33.1.7 CHONIC GASTRIC LUCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 33.1.7 CHONIC GASTRIC LUCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 34.2 CHONIC GASTRIC LUCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 35.2 CHONIC GASTRIC LUCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 35.2 CHONIC DUDOPANA LUCER WITH HEMORRHAGE WITH OBSTRUCTION 36.2 CHONIC DUDOPANA LUCER WITH HEMORRHAGE WITH OBSTRUCTION 37.2 CHONIC DUDOPANA LUCER WITH PERFORATION 37.2 CHONIC DUDOPANA LUCER WITH PERFORATION 37.2 CHONIC OR UNSPECIFIED DUDOPANA LUCER WITH HEMORRHAGE WITH OBSTRUCTION 37.2 CHONIC OR UNSPECIFIED DUDOPANA LUCER WITH PERFORATION 37.3 CHONIC OR UNSPECIFIED DUDOPANA LUCER WITH PERFORATION 37.3 CHONIC OR UNSPECIFIED DUDOPANA LUCER WITH PERFORATION 37.3 CHONIC OR UNSPECIFIED DUDOPANA LUCER WITH PERFORATION 37.3 CHONIC OR UNSPECIFIED DUDOPANA LUCER WITH PERFORATION 37.3 CHONIC OR UNSPECIFIED DUDOPANA LUCER WITH HEMORRHAGE AND PERFORATION 37.3 CHONIC OR UNSPECIFIED STEW WITH HEMORRHAGE AND PERFORATION 37.3 CHONIC OR UNSPECIFIED STEW WITH HEMORRHAGE AND PERFORATION 37.3 CHONIC OR UNSPECIFIED STEW WITH HEMORRHAGE AND PERFORATION 37.4 CHONIC OR UNSPECIFIED STEW WITH HEMORRHAGE AND PERFORATION 37.5 CHONIC OR UNSPECIFIED STEW WITH HEMORRHAGE WITHOUT OBSTRUCTION 37.4 CHONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE OR PERFORATI | | |
| ACUTE GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION 33.1.2 ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 33.1.3 ACUTE GASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 33.1.4 CHORNIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE OR PERFORATION 33.1.5 CHORNIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION 33.1.6 CHORNIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 33.1.7 CHORNIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 33.1.7 CHORNIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION 33.1.7 CHORNIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION 33.1.7 CHORNIC OR UNSPECIFIED SA EVENT OF HEMORRHAGE AND PERFORATION 33.1.7 CHORNIC OR UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 33.1.1 CHORNIC OR UNSPECIFIED SA EVENT OF CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 33.1.2 CHORNIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE OR PERFORATION 33.1.3 CHORNIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 33.2 CHORNIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 33.3 CHORNIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 33.3 CHORNIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 33.4 CHORNIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 33.5 CHORNIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 33.6 CHORNIC OR UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 33.7 CHORNIC OR UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 33.8 CHORNIC OR UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 33.9 CHORNIC OR UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 33.9 CHORNIC OR UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 33.1 CHORNIC OR UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 33.1 CHORNIC OR UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 33.1 CHORNIC OR UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 34.1 CHORNIC OR UNSPECIFIED S | | |
| ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 33.12 ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 33.13 ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 33.15 CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 33.16 CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 33.17 CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 33.17 CHRONIC GASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 33.19 ACUTE DUDOBENAL ULCER WITH HEMORRHAGE WITHOUT DESTRUCTION 33.21 ACUTE DUDOBENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 33.23 ACUTE DUDOBENAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 33.24 CHRONIC OR UNSPECIFIED DUDOBENAL ULCER WITH HEMORRHAGE OR PERFORATION 33.25 ACUTE DUDOBENAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 33.26 CHRONIC OR UNSPECIFIED DUDOBENAL ULCER WITH HEMORRHAGE OR PERFORATION 33.27 ACUTE PUDOBENAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 33.28 ACUTE PUDOBENAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 33.29 ACUTE PUDOBENAL ULCER WITHOUT MENTION OF HEMORRHAGE WITH OBSTRUCTION 33.20 ACUTE PUDOBENAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 33.31 ACUTE PEPTIC ULCER OF UNSPECIFIED SET WITH PERFORATION 33.32 ACUTE PEPTIC ULCER OF UNSPECIFIED SET WITH PERFORATION 33.34 ACUTE PEPTIC ULCER OF UNSPECIFIED SET WITH PERFORATION 33.4 ACUTE PEPTIC ULCER OF UNSPECIFIED SET WITH HEMORRHAGE WITH OBSTRUCTION 44 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 45 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 46 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 46 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE 46 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFI | | |
| ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION ACUTE GASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION CHRONIC GASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION CHRONIC GASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION ACUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION ACUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION ACUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION ACUTE DUODENAL ULCER WITHOUT MENTION OF HEMORRHAGE WITHOUT OBSTRUCTION ACUTE DUODENAL ULCER WITHOUT MENTION OF HEMORRHAGE WITHOUT OBSTRUCTION ACUTE DUODENAL ULCER WITHOUT MENTION OF HEMORRHAGE CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION CHRONIC OR UNSPECIFIED SPETIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION CHRONIC OR UNSPECIFIED SPETIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION CHRONIC OR UNSPECIFIED SPETIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED SPETIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE ACUTE GASTROILINAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED GASTROILINAL ULCER WITH HEMORRHAGE CHRO | | |
| ACUTE CASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE OR PERFORATION WITH OBSTRUCTION CHRONIC GASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION CHRONIC OR UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION ACUTE DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION ACUTE DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH PERFORATION CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH PERFORATION CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH PERFORATION CHRONIC OR UNSPECIFIED OWNER OF THE WITH HEMORRHAGE AND PERFORATION CHRONIC OR UNSPECIFIED SHE WITH HEMORRHAGE AND PERFORATION CHRONIC OR UNSPECIFIED SHE WITH HEMORRHAGE AND PERFORATION CHRONIC OR UNSPECIFIED PERFORMED SHE WITH HEMORRHAGE WITH DESTRUCTION CHRONIC OR UNSPECIFIED PERFORMED SHE WITH HEMORRHAGE WITH DESTRUCTION CHRONIC OR UNSPECIFIED PERFORMED CHARGE OR PERFORATION CHRONIC OR UNSPECIFIED PERFORMED CHARGE OR PERFORATION CHRONIC OR UNSPECIFIED PERFORMED CHARGE OR PERFORATION CHRONIC OR UNSPECIFIED SHE WITH HEMORRHAGE WITH HEMORRHAGE WITH DESTRUCTION CHRONIC OR UNSPECIFIED SHE WITH HEMORRHAGE CHRONIC OR UNSPECIFIED SHE WITH HEMORRHAGE WITH HEMORRHAGE OR PERFORATION CHRONIC OR UNSPECIFIED SASTROLEUMAL ULCER WITH HEMORRHAGE CHRONIC OR UNSPECIFIED GASTROLEUMAL ULCER WITH HEMORRHAGE CHRONIC OR UNSPECIFIED GASTROLEUMAL | | |
| CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION CHRONIC GASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE AND PERFORATION WITH OBSTRUCTION CHRONIC GASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION CHRONIC GASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION CHRONIC GASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION CHRONIC GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION ACUTE DUDOBNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED DUDOBNAL ULCER WITH HEMORRHAGE OR PERFORATION CHRONIC OR UNSPECIFIED DUDOBNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED DUDOBNAL ULCER WITH HEMORRHAGE WITHOUT MENTION OF HEMORRHAGE OR PERFORATION CHRONIC OR UNSPECIFIED DUDOBNAL ULCER WITH HEMORRHAGE WITHOUT MENTION OF HEMORRHAGE OR PERFORATION CHRONIC OR UNSPECIFIED DUDOBNAL ULCER WITH HEMORRHAGE WITHOUT MENTION OF HEMORRHAGE OR PERFORATION CHRONIC OR UNSPECIFIED DUDOBNAL ULCER WITH HEMORRHAGE WITHOUT MENTION OF HEMORRHAGE OR PERFORATION CHRONIC OR UNSPECIFIED DUSTE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH DESTRUCTION CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH DESTRUCTION CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE CH | | |
| 531.6 CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.6 CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.7 CHRONIC GASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 531.9 GASTRIC ULCER UNSPECIFIED ASSTRIC ULCER WITHOUT OR HEMORRHAGE OR PERFORATION 532.1 ACUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 532.1 ACUTE DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.2 ACUTE DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.3 ACUTE DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.4 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE OR PERFORATION 532.5 ACUTE DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.6 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.7 HORNIC OR UNSPECIFIED DUODENAL ULCER WITH PERFORATION 532.8 PRODENAL ULCER OF UNSPECIFIED DUODENAL ULCER WITH PERFORATION 533.1 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.2 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.3 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.4 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.5 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.6 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.7 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.8 PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 534.1 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 535.2 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 536.4 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE OR PERFORATION 537.6 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 538.4 CHRONIC OR UNSPECIFIED SITE WITH HEMORRH | | |
| 531.6 CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.7 CHRONIC GOATRIC ULCER WITHOUT MENTION OF HEMORRHAGE AND PERFORATION 531.7 CHRONIC GASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 532.1 CAUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 532.2 ACUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 532.3 ACUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 532.4 CHRONIC OR UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 532.5 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 532.6 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 532.5 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 533.1 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 533.2 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 533.3 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITHOUT STRUCTION 533.4 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.5 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.6 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.6 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 534.2 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 535.4 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 536.5 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 537.6 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 538.6 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 539.7 PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 530.7 PERFORATIO | | |
| 531.61 531.7 CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE ON PERFORATION WITH OBSTRUCTION 531.9 GASTRIC ULCER UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 532.0 532.0 ACUTE DUDDENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 32.1 ACUTE DUDDENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 32.2 ACUTE DUDDENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 32.3 ACUTE DUDDENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 32.4 CHRONIC OR UNSPECIFIED DUDDENAL ULCER WITH HEMORRHAGE OR PERFORATION 32.4 CHRONIC OR UNSPECIFIED DUDDENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.5 CHRONIC OR UNSPECIFIED DUDDENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.6 DUDDENAL ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.1 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.2 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.2 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.4 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH DESTRUCTION 533.5 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH DESTRUCTION 533.6 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 534.6 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 535.6 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 536.7 ACUTE GASTROJEUNAL ULCER WITH HEMORRHAGE 537.8 ACUTE GASTROJEUNAL ULCER WITH HEMORRHAGE 538.4 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 538.6 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE OR PERFORATION 539.6 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 530.7 ACUTE GASTROJEUNAL ULCER WITH HEMORRHAGE 530.7 ACUTE GASTROJEUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 530.7 CHRONIC OR UNSPECIFIED GASTROJEUNAL ULCER WITH HEMORRHAGE AND PERFORATION 530.7 | | |
| 531.7 531.8 531.7 532.8 532.8 532.1 532.1 532.1 532.1 532.1 532.3 532.1 532.3 532.3 532.3 532.3 532.4 532.4 532.4 532.4 532.5 532.5 532.5 532.5 532.5 532.5 532.5 532.6 532.7 532.8 533.8 | | |
| S31.9 GASTRIC ULCER UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 32.01 ACUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 32.1 ACUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 32.2 ACUTE DUODENAL ULCER WITH PERFORATION 32.3 ACUTE DUODENAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 32.4 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE 32.4 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE 32.4 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH PERFORATION 32.5 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH PERFORATION 33.6 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH PERFORATION 33.7 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 33.8 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 33.9 CAUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 33.1 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 33.4 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 33.5 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 33.9 PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 33.9 PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 33.1 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE OR PERFORATION 33.1 CHRONIC OR UNSPECIFIED SEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE ON PERFORATION 34.2 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE 35.4 CHRONIC OR UNSPECIFIED SACUTE WITH HEMORRHAGE 35.4 CHRONIC OR UNSPECIFIED SACUTE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 36.5 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 37.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE OR PERFORATION 37.7 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE OR PERFORATION 37.8 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE OR PERFORATION 37.9 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER | | |
| ACUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 532.1 ACUTE DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.1 ACUTE DUODENAL ULCER WITH HEPRORATION 532.3 ACUTE DUODENAL ULCER WITH HEPRORATION 532.4 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE OR PERFORATION 532.4 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.5 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.6 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 533.1 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 533.2 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 533.4 CHRONIC OR UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 533.4 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.4 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.5 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 534.6 CHRONIC OR UNSPECIFIED SITE ULCER OF UNSPECIFIED SITE WITH PERFORATION 535.6 CHRONIC OR UNSPECIFIED SITE ULCER OF UNSPECIFIED SITE WITH PERFORATION 536.6 CHRONIC OR UNSPECIFIED SITE ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 537.7 PEPTIC ULCER OF UNSPECIFIED SITE UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 538.4 CHRONIC OR UNSPECIFIED SITE UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 539.4 CHRONIC OR UNSPECIFIED SITE UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 539.4 CHRONIC OR UNSPECIFIED SHAD AUTH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 531.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 531.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 531.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 531.7 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 532.4 OTHER SPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 533.61 UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 535.61 UNSPECIFIED GASTRO | | |
| ACUTE DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 332.1 ACUTE DUODENAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 332.3 ACUTE DUODENAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 332.4 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 332.5 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 332.6 DUODENAL ULCER UNSPECIFIED SA CAUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 333.1 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 333.2 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 333.2 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 333.4 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 333.5 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 333.6 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 334.7 PEPTIC ULCER OF UNSPECIFIED SITE UNSPECIFIED SITE WITH PERFORATION 335.9 PEPTIC ULCER OF UNSPECIFIED SITE UNSPECIFIED SITE WITH PERFORATION 336.4 ACUTE GASTROIDIANAL ULCER WITH HEMORRHAGE AND PERFORATION 337.4 ACUTE GASTROIDIANAL ULCER WITH HEMORRHAGE AND PERFORATION 338.4 CHRONIC OR UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 339.4 ACUTE GASTROIDIANAL ULCER WITH HEMORRHAGE AND PERFORATION 340.4 CHRONIC OR UNSPECIFIED GASTROIDIANAL ULCER WITH HEMORRHAGE 341.4 CHRONIC OR UNSPECIFIED GASTROIDIANAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 342.5 CHRONIC OR UNSPECIFIED GASTROIDIANAL ULCER WITH HEMORRHAGE AND PERFORATION 343.6 CHRONIC OR UNSPECIFIED GASTROIDIANAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 344.6 CHRONIC OR UNSPECIFIED GASTROIDIANAL ULCER WITH HEMORRHAGE AND PERFORATION 351.6 CHRONIC OR UNSPECIFIED GASTROIDIANAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 352.7 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 353.5 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 353.5 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 353.6 UNDERTICULITIS OF SMAL | | |
| 532.1 ACUTE DUODENAL ULCER WITH PERFORATION 532.2 ACUTE DUODENAL ULCER WITHOUT MENTION OF HEMORRHAGE 532.4 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE 532.4 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.9 DUODENAL ULCER UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE OR PERFORATION 533.1 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 533.2 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.4 CHRONIC OR UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 533.4 CHRONIC OR UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 533.4 CHRONIC OR UNSPECIFIED SITE UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.5 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.6 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.6 CHRONIC OR UNSPECIFIED SEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.2 ACUTE GASTROJEJUNAL ULCER OF UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 534.4 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.4 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.5 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 535.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 536.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 537.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 537.7 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 538.1 ACCOHOLIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 539.7 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE 539.7 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE 539.7 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE 539.7 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE 539.7 ACUTE GASTROJEJUNAL ULCER WITH HEMOR | | |
| 532.3 ACUTE DUODENAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 532.4 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.5 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH PERFORATION 532.6 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH PERFORATION 533.7 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 533.1 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.2 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.4 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.5 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.6 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.7 PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.9 PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.2 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.4 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 535.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 535.1 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 536.2 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 537.4 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 538.4 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 535.1 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 535.1 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 535.1 ACUTE GASTRITIS WITH HEMORRHAGE 536.6 DUODENTIS WITH HEMORRHAGE 537.6 DUODENTIS WITH HEMORRHAGE 538.6 DUODENTIS WITH HEMORRHAGE 539.6 DUODENTIS WITH HEMORRHAGE 540.0 DIVERTICULTIS OF SMALL INTESTINE WITH HEMORRHAGE 550.1 DIVERTICULTIS OF SMALL INTESTINE WITH HEMORRHAGE 550.2 DIVERTICULTIS OF SMALL INTESTINE WITH HEMORRHAGE 550.2 DIVERTICUL | | |
| 532.41 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE 532.51 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.52 DUODENAL ULCER UNSPECIFIED DUODENAL ULCER WITH PERFORATION 533.63 DUODENAL ULCER OF UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 533.61 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.62 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 533.63 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.63 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.69 PEPTIC ULCER OF UNSPECIFIED SITE UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.60 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.71 ACUTE GASTROIEUNAL ULCER WITH HEMORRHAGE 534.72 ACUTE GASTROIEUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.61 CHRONIC OR UNSPECIFIED GASTROIEUNAL ULCER WITH HEMORRHAGE 534.62 CHRONIC OR UNSPECIFIED GASTROIEUNAL ULCER WITH HEMORRHAGE 535.61 CHRONIC OR UNSPECIFIED GASTROIEUNAL ULCER WITH HEMORRHAGE 536.61 CHRONIC OR UNSPECIFIED GASTROIEUNAL ULCER WITH HEMORRHAGE AND PERFORATION 536.61 CHRONIC OR UNSPECIFIED GASTROIEUNAL ULCER WITH HEMORRHAGE 537.61 CHRONIC OR UNSPECIFIED GASTROIEUNAL ULCER WITH HEMORRHAGE AND PERFORATION 538.61 CHRONIC OR UNSPECIFIED GASTROIEUNAL ULCER WITH HEMORRHAGE AND PERFORATION 539.71 (ARONIC OR UNSPECIFIED GASTROIEUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 539.71 (DATE SPECIFIED GASTROIEUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 539.71 (DATE SPECIFIED GASTROIEUNAL ULCER WITH HEMORRHAGE 539.71 (DOUDENTIS WITH HEMORRHAGE 549.72 (DOUDENTIS WITH HEMORRHAGE 549.73 (DOUDENTIS WITH HEMORRHAGE 549.74 (DOUDENTIS WITH HEMORRHAGE 549.75 (DOUDENTIS WITH HEMORRHAGE 549.75 (DOUDENTIS WITH HEMORRHAGE 549.75 (DOUDENTIS WITH HEMORRHAGE 549.75 (DOUDENTIS WITH HEMORRHAGE 549.75 (DOUDENTIS WITH HEMORRHAGE 550.75 | | |
| 532.41 532.42 532.53 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION 532.9 DUODENAL ULCER UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 533.1 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 533.2 CHRONIC OR UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.41 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH DUSTRUCTION 533.61 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.61 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 534.62 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.64 CHRONIC OR UNSPECIFIED SITE UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.65 CHRONIC OR UNSPECIFIED SITE UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.67 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.61 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.62 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.63 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.64 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 535.61 DUSCRIPPIN OF WITHOUT WISPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.61 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 535.91 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 536.61 DUSCRIPPIN OR WISPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 537.91 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 538.91 DUSCRIPPIN OR WITHOUT WITHOUT HEMORRHAGE 539.10 DUSCRIPPIN OR WITHOUT WITHOUT HEMORRHAGE 530.61 DUSCRIPPIN OR WITHOUT WITHOUT WITHOUT WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 539.71 DUS | | |
| 532.5 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH PERFORATION 533.1 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 533.2 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.21 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 533.41 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.51 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.6 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.7 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.8 CHRONIC OR UNSPECIFIED SITE UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.4 CUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.4 CUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.4 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.5 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.9 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 535.1 ATROPHIC GASTRITIS WITH HEMORRHAGE 535.5 LACOHOLIC GASTRITIS WITH HEMORRHAGE 535.5 LACOHOLIC GASTRITIS WITH HEMORRHAGE 535.5 LOUDENNITS WITH HEMORRHAGE 535.5 LOUDENNITS WITH HEMORRHAGE 535.5 LOUDENNITS WITH HEMORRHAGE 535.6 LOUDENNITS WITH HEMORRHAGE 535.6 LOUDENNITS WITH HEMORRHAGE 535.7 LOUR REPORT OF COLON (WITHOUT HEMORRHAGE) 536.7 LOUR REPORT OF COLON (WITHOUT HEMORRHAGE) 537.8 LOUDENTIS WITH HEMORRHAGE 538.8 LOUDENTIS WITH HEMORRHAGE 538.9 LOUDENTIS WITH HEMORRHAGE 539.1 GROSS HEMATURIA 539.1 GROSS HEMATURIA 539.1 GROSS HEMATURIA 539.1 LOUR REPORT OF COLON (WITHOUT HEMORRHAGE) 540.1 LOUR REPORT OF COLON (WITHOUT HEMORRHAGE) 551.1 CHRONIC OR UNSPECIFIED GASTROJEOUDENTIS WITH HEMORRHAGE 552.1 DIVERTICULITIS OF COLON WITHOUT HEMORRHAGE 553.1 LOUDENTIS WITH HEMORRHAGE 554.1 DIVERTICULITIS OF COLON WITHOUT HEM | | |
| 532.9 DUODENAL ULCER UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 533.21 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.41 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 533.41 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.61 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.62 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.64 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.75 CHRONIC OR UNSPECIFIED SITE UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.76 CHRONIC OR UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.77 CHRONIC OR UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.78 CHRONIC OR UNSPECIFIED SITE WITH HEMORRHAGE 534.40 CHRONIC OR UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.41 CHRONIC OR UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.42 CHRONIC OR UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.43 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.44 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.54 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 535.61 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 535.61 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 535.61 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 535.61 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE OR PERFORATION 535.61 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 535.61 DUSPECTICULTIS OF SMALL INTESTINE WITH HEMORRHAGE 535.61 DUSPECTICULTIS OF SMALL INTESTINE WITH HEMORRHAGE 536.62 DUSPECTICULTIS OF SMALL INTESTINE WITH HEMORRHAGE 536.61 DUSPECTICULTIS OF SMALL INTESTINE WITH HEMORRHAGE 536.62 DUSPECTICU | | |
| 533.1 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 533.21 CAUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 533.41 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.41 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.41 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 533.41 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.52 CHRONIC OR UNSPECIFIED SITE UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.61 CHRONIC OR UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.61 CHRONIC OR UNSPECIFIED SITE WITH HEMORRHAGE 534.42 CHIE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 534.61 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.62 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.63 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.64 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.96 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 535.11 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 535.11 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 535.11 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE OR PERFORATION 536.11 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 537.11 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 538.21 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 538.22 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 539.35 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 539.36 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 539.37 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 539.38 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 539.39 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 539.40 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 539.41 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 540.41 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 550.41 UNSPECIFIED GASTRITI | | |
| 533.21 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.41 CHRONIC OR UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 533.41 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.51 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 534.61 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.62 CHRONIC OR UNSPECIFIED SITE UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.61 CHRONIC OR UNSPECIFIED SITE UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 534.62 CHRONIC OR UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 534.64 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.65 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.66 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 535.11 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 535.40 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 535.41 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 535.41 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 536.40 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 537.41 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 538.41 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 538.42 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 539.41 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 540.41 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 550.40 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 550.40 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 550.40 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 550.40 UNSPECIFIED GASTRITIS WIT | | |
| 533.21 533.41 533.42 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.51 535.51 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.61 535.72 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.61 534.22 CHRONIC OR UNSPECIFIED SITE UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.41 534.42 CHRONIC OR UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 534.41 534.42 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.61 534.62 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT MENTION OF HEMORRHAGE OR PERFORATION UNSPECIFIED GASTRITIS WITH HEMORRHAGE 535.41 535.41 546.43 547.44 548.45 549.47 5 | | |
| 533.41 533.41 533.41 533.41 533.51 533.61 534.61 534.61 535.61 53 | | |
| 533.41 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION 533.51 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 533.61 533.61 533.72 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 534.73 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.74 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.75 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.61 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.61 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.62 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.63 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 535.41 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 536.53 ATROPHIC GASTRITIS WITH HEMORRHAGE 535.51 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 535.51 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 535.51 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 536.01 DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 536.01 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 5378.11 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 5378.11 GROSS HEMATURIA 539.71 CHRONIC OR UNSPECIFIED AS CUECA OF UNSPECIFIED SITE WITH HEMORRHAGE OF VAGINA | | |
| 533.5 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION 533.6 CHRONIC OR UNSPECIFIED SITE UNCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION 533.7 PEPTIC ULCER OF UNSPECIFIED SITE UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 534.2 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.2 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.4 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.5 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.7 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 534.9 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 535.11 ATROPHIC GASTRITIS WITH HEMORRHAGE 535.31 ALCOHOLIC GASTRITIS WITH HEMORRHAGE 535.31 AUCHOLIC GASTRITIS WITH HEMORRHAGE 535.31 UNSPECIFIED GASTRITIS (WITHOUT HEMORRHAGE) 535.31 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 535.31 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 536.41 DUODENITIS WITH HEMORRHAGE 540.20 DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 550.31 DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 550.32 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 562.33 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 563.84 DIVERTICULIOSIS OF COLON WITH HEMORRHAGE 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 569.87 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 569.87 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 569.87 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 569.88 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | | |
| 533.9 PEPTIC ULCER OF UNSPECIFIED SITE UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 534.4 CAUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.4 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.4 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 534.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.9 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.9 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.9 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 535.11 ATROPHIC GASTRITIS WITH HEMORRHAGE 535.11 ATROPHIC GASTRITIS WITH HEMORRHAGE 535.21 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 535.21 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 535.21 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 535.21 DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 536.20 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 536.21 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 5378.1 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 536.21 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 5378.1 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 538.8 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 539.71 GROSS HEMATURIA 539.71 GROSS HEMATURIA 539.71 GROSS HEMATURIA 539.71 GROSS HEMATURIA 539.71 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | | |
| 534.2 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.21 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 534.4 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.7 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 534.8 CASTROJEJUNAL ULCER UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 535.11 ATROPHIC GASTRITIS WITH HEMORRHAGE 535.11 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 535.5 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 535.6 DUDOENITIS WITH HEMORRHAGE 536.0 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 562.01 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 562.11 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 562.12 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 563.81 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 569.81 GROSS HEMATURIA 6623.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | 533.6 | CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION |
| 534.21 534.21 534.42 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.61 534.61 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.61 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.91 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.91 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 535.91 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 536.91 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 536.91 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 537.91 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 536.91 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 535.91 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 535.91 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 536.91 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 536.91 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 540.91 UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE 540.91 UNSPECIFIED GASTROJEJUNAL | 533.9 | PEPTIC ULCER OF UNSPECIFIED SITE UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION |
| 534.21 534.41 534.42 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.61 534.62 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.61 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.62 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 534.69 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 534.61 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 535.51 ATROPHIC GASTRITIS WITH HEMORRHAGE 535.51 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 535.51 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 535.51 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 540.01 DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 550.01 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 562.02 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 562.11 DIVERTICULIOSIS OF COLON WITH HEMORRHAGE 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 578.1 BLOOD IN STOOL GROSS HEMATURIA 678.28 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | 534 | ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE |
| 534.4 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION 534.9 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.9 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 534.9 GASTROJEJUNAL ULCER UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 535.11 ATROPHIC GASTRITIS WITH HEMORRHAGE 535.31 ACOHOLIC GASTRITIS WITH HEMORRHAGE 535.40 UNSPECIFIED GASTRITIS (WITHOUT HEMORRHAGE) 535.51 UNSPECIFIED GASTRITIS AND GASTRODUODENITIS WITH HEMORRHAGE 535.61 DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 562.01 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 562.02 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 562.03 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 562.04 DIVERTICULITIS OF COLON WITH HEMORRHAGE 563.8 BLOOD IN STOOL 569.75 AGROSS HEMATURIA 670.75 GROSS HEMATURIA 670.76 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | 534.2 | ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION |
| 534.4 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 534.9 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 534.9 CASTROJEJUNAL ULCER UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 535.11 ATROPHIC GASTRITIS WITH HEMORRHAGE 535.31 ALCOHOLIC GASTRITIS WITH HEMORRHAGE 535.41 UNSPECIFIED GASTRITIS (WITHOUT HEMORRHAGE) 535.51 UNSPECIFIED GASTRITIS AND GASTRODUODENITIS WITH HEMORRHAGE 502.01 DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 502.02 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 502.03 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 502.04 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 502.05 DIVERTICULITIS OF COLON WITH HEMORRHAGE 502.07 DIVERTICULOSIS OF COLON WITH HEMORRHAGE 509.07 GROSS HEMATURIA 603.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | 534.21 | ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION |
| 534.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION 534.9 CASTROJEJUNAL ULCER UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 535.11 ATROPHIC GASTRITIS WITH HEMORRHAGE 535.31 ALCOHOLIC GASTRITIS WITH HEMORRHAGE 535.41 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 535.51 UNSPECIFIED GASTRITIS WITH HEMORRHAGE 535.61 DUODENITIS WITH HEMORRHAGE 536.01 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 546.01 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 556.11 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 5578.11 DIVERTICULOSIS OF COLON WITH HEMORRHAGE 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 569.87 CROSS HEMATURIA 678.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | 534.4 | CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE |
| 534.6 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 534.9 GASTROJEJUNAL ULCER UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 535.11 ATROPHIC GASTRITIS WITH HEMORRHAGE 535.4 OTHER SPECIFIED GASTRITIS (WITHOUT HEMORRHAGE) 535.5 UNSPECIFIED GASTRITIS (WITHOUT HEMORRHAGE) 535.61 DUODENITIS WITH HEMORRHAGE 562.01 DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 562.03 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 562.11 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 562.12 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 578.1 BLOOD IN STOOL 579.71 GROSS HEMATURIA 672.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | 534.4 | CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION |
| 534.9 GASTROJEJUNAL ULCER UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 535.11 ATROPHIC GASTRITIS WITH HEMORRHAGE 535.41 UNSPECIFIED GASTRITIS WITH HEMORRHAGE) 535.51 UNSPECIFIED GASTRITIS (WITHOUT HEMORRHAGE) 535.61 DUODENITIS WITH HEMORRHAGE 502.01 DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 562.01 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 562.11 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 562.12 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 562.13 DIVERTICULITIS OF COLON WITH HEMORRHAGE 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 578.1 BLOOD IN STOOL 599.71 GROSS HEMATURIA 623.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | 534.6 | CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION |
| 535.11 ATROPHIC GASTRITIS WITH HEMORRHAGE 535.31 ALCOHOLIC GASTRITIS WITH HEMORRHAGE 535.31 OTHER SPECIFIED GASTRITIS (WITHOUT HEMORRHAGE) 535.51 UNSPECIFIED GASTRITIS AND GASTRODUODENITIS WITH HEMORRHAGE 502.01 DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 502.03 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 502.10 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 502.11 DIVERTICULOSIS OF COLON WITH HEMORRHAGE 509.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 578.1 BLOOD IN STOOL GROSS HEMATURIA 623.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | 534.6 | CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION |
| 535.31 535.4 535.4 535.5 535.51 UNSPECIFIED GASTRITIS (WITHOUT HEMORRHAGE) 535.61 DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 562.01 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 562.11 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 562.12 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 562.13 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 562.14 DIVERTICULOSIS OF COLON WITH HEMORRHAGE 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 578.1 BLOOD IN STOOL GROSS HEMATURIA 673.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | 534.9 | GASTROJEJUNAL ULCER UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION |
| 535.4 OTHER SPECIFIED GASTRITIS (WITHOUT HEMORRHAGE) 535.51 UNSPECIFIED GASTRITIS AND GASTRODUODENITIS WITH HEMORRHAGE 535.61 DUODENITIS WITH HEMORRHAGE 562.01 DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 562.11 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 562.12 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 562.13 DIVERTICULOSIS OF COLON WITH HEMORRHAGE 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 578.11 BLOOD IN STOOL 6ROSS HEMATURIA 673.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | | |
| 535.51 UNSPECIFIED GASTRITIS AND GASTRODUODENITIS WITH HEMORRHAGE 535.61 DUODENITIS WITH HEMORRHAGE 562.01 DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 562.03 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 562.12 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 562.12 DIVERTICULIS OF COLON (WITHOUT HEMORRHAGE) 562.12 DIVERTICULOSIS OF COLON WITH HEMORRHAGE 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 578.1 BLOOD IN STOOL 599.71 GROSS HEMATURIA 623.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | | |
| 535.61 DUODENITIS WITH HEMORRHAGE 562.01 DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 562.03 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 562.11 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 562.12 DIVERTICULOSIS OF COLON WITH HEMORRHAGE 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 578.1 BLOOD IN STOOL 599.71 GROSS HEMATURIA 623.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | | |
| 562.01 DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE) 562.03 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 562.11 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 562.12 DIVERTICULOSIS OF COLON WITH HEMORRHAGE 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 578.1 BLOOD IN STOOL 599.71 GROSS HEMATURIA 623.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | | |
| 562.03 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE 562.11 DIVERTICULOSIS OF COLON (WITHOUT HEMORRHAGE) 562.12 DIVERTICULOSIS OF COLON WITH HEMORRHAGE 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 578.1 BLOOD IN STOOL 599.71 GROSS HEMATURIA 623.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | | |
| 562.11 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE) 562.81 DIVERTICULOSIS OF COLON WITH HEMORRHAGE 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 578.11 BLOOD IN STOOL 579.71 GROSS HEMATURIA 623.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | | |
| 562.12 DIVERTICULOSIS OF COLON WITH HEMORRHAGE 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 578.1 BLOOD IN STOOL 599.71 GROSS HEMATURIA 623.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | | |
| 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE 578.1 BLOOD IN STOOL 599.71 GROSS HEMATURIA 623.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | | |
| 578.1 BLOOD IN STOOL 599.71 GROSS HEMATURIA 623.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | | |
| 599.71 GROSS HEMATURIA 623.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | | |
| 623.8 OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF VAGINA | | |
| | | OTHER DISORDERS OF MENSTRUATION AND OTHER ABNORMAL BLEEDING FROM FEMALE GENITAL TRACT |


| К6 | 4.8 | Other hemorrhoids |
|----|-----|-----------------------------------------------------|
| К9 | 2.2 | Gastrointestinal hemorrhage, unspecified |
| N8 | 9.8 | Other specified noninflammatory disorders of vagina |
| N9 | 3.9 | Abnormal uterine and vaginal bleeding, unspecified |
| R0 | 4.1 | Hemorrhage from throat |
| R0 | 4.2 | Hemoptysis |

#### **Inpatient, Primary Diagnosis: ICD-9 Codes**

- 280.0 IRON DEFICIENCY ANEMIA SECONDARY TO BLOOD LOSS (CHRONIC)
- 455.7 UNSPECIFIED THROMBOSED HEMORRHOIDS
- 459.0 HEMORRHAGE UNSPECIFIED
- 530.10 ESOPHAGITIS UNSPECIFIED
- 530.13 EOSINOPHILIC ESOPHAGITIS
- 531.0 ACUTE GASTRIC ULCER WITH HEMORRHAGE
- 531.1 ACUTE GASTRIC ULCER WITH PERFORATION
- 531.2 ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION
- 531.20 ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION
- 531.3 ACUTE GASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION
- 531.4 CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE
- 531.6 CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION
- 531.61 CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION
- 531.9 GASTRIC ULCER UNSPECIFIED AS ACUTE OR CHRONIC
- WITHOUT MENTION OF HEMORRHAGE OR PERFORATION
- 532.0 ACUTE DUODENAL ULCER WITH HEMORRHAGE
- 532.00 ACUTE DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION
- 532.01 ACUTE DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION
- 532.2 ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION
- 532.20 ACUTE DUODENAL ULCER WITH HEMORRHAGE AND
- PERFORATION WITHOUT OBSTRUCTION
- 532.3 ACUTE DUODENAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION

- 532.4 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE
- 532.41 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION
- 532.5 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH PERFORATION
- 532.61 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION
- 533.0 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE
- 533.00 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION
- 533.01 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION
- 533.1 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH PERFORATION
- 533.2 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION
- 533.20 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION
- 533.3 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITHOUT
- MENTION OF HEMORRHAGE AND PERFORATION
- 533.6 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF
- UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION
- 533.60 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF
- UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION
- 533.7 CHRONIC PEPTIC ULCER OF UNSPECIFIED SITE WITHOUT MENTION OF HEMORRHAGE OR PERFORATION
- 534.00 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION
- 534.01 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION
- 534.20 ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION
- 534.3 ACUTE GASTROJEJUNAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 534.40 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION
- 534.41 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE WITH OBSTRUCTION
- 534.61 CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 534.7 CHRONIC GASTROJEJUNAL ULCER WITHOUT MENTION OF
- 534.7 CHRONIC GASTROJEJUNAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION
- 534.9 GASTROJEJUNAL ULCER UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION
- 535.00 ACUTE GASTRITIS (WITHOUT HEMORRHAGE)
- 535.01 ACUTE GASTRITIS WITH HEMORRHAGE
- 535.10 ATROPHIC GASTRITIS (WITHOUT HEMORRHAGE)
- 535.20 GASTRIC MUCOSAL HYPERTROPHY (WITHOUT HEMORRHAGE)
- 535.21 GASTRIC MUCOSAL HYPERTROPHY WITH HEMORRHAGE
- 535.31 ALCOHOLIC GASTRITIS WITH HEMORRHAGE
- 535.40 OTHER SPECIFIED GASTRITIS (WITHOUT HEMORRHAGE)
- 535.41 OTHER SPECIFIED GASTRITIS WITH HEMORRHAGE
- 562.00 DIVERTICULOSIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE)
- 562.01 DIVERTICULITIS OF SMALL INTESTINE (WITHOUT HEMORRHAGE)
- 562.03 DIVERTICULITIS OF SMALL INTESTINE WITH HEMORRHAGE
- 562.11 DIVERTICULITIS OF COLON (WITHOUT HEMORRHAGE)
- 562.13 DIVERTICULITIS OF COLON WITH HEMORRHAGE
- 569.85 ANGIODYSPLASIA OF INTESTINE WITH HEMORRHAGE

| 578.0 - HEMATEMESIS 578.1 - BLOOD IN STOOL 578.9 - HEMORRHAGE OF GASTROINTESTINAL TRACT UNSPECIFIED 593.81 - VASCULAR DISORDERS OF KIDNEY 599.70 - HEMATURIA UNSPECIFIED 599.71 - GROSS HEMATURIA 623.6 - VAGINAL HEMATOMA 626.6 - METRORRHAGIA 784.7 - EPISTAXIS 784.8 - HEMORRHAGE FROM THROAT 786.31 - ACUTE IDIOPATHIC PULMONARY HEMORRHAGE IN INFANTS 285.1 - ACUTE POSTHEMORRHAGIC ANEMIA 455.1 - INTERNAL THROMBOSED HEMORRHOIDS |
|---|
| 455.2 - INTERNAL HEMORRHOIDS WITH OTHER COMPLICATION<br>455.4 - EXTERNAL THROMBOSED HEMORRHOIDS |
| 455.5 - EXTERNAL HEMORRHOIDS WITH OTHER COMPLICATION |
| 455.6 - UNSPECIFIED HEMORRHOIDS WITHOUT COMPLICATION |
| 455.8 - UNSPECIFIED HEMORRHOIDS WITH OTHER COMPLICATION 455.9 - RESIDUAL HEMORRHOIDAL SKIN TAGS 456.0 - ESOPHAGEAL VARICES WITH BLEEDING 456.20 - ESOPHAGEAL VARICES IN DISEASES CLASSIFIED ELSEWHERE WITH BLEEDING 530.1 - ESOPHAGITIS 530.11 - REFLUX ESOPHAGITIS 530.12 - ACUTE ESOPHAGITIS 530.19 - OTHER ESOPHAGITIS 530.7 - GASTROESOPHAGEAL LACERATION-HEMORRHAGE |
| SYNDROME |
| 530.82 - ESOPHAGEAL HEMORRHAGE |
| 330.02 - ESUFTIAGEAL HEINURKHAGE |

- 531.00 ACUTE GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION
- 531.01 ACUTE GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION
- 531.21 ACUTE GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION
- 531.40 CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION
- 531.41 CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE WITH OBSTRUCTION
- 531.5 CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH PERFORATION
- 531.60 CHRONIC OR UNSPECIFIED GASTRIC ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION
- 531.7 CHRONIC GASTRIC ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION
- 532.1 ACUTE DUODENAL ULCER WITH PERFORATION
- 532.21 ACUTE DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION
- 532.40 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE WITHOUT OBSTRUCTION
- 532.6 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION
- 532.60 CHRONIC OR UNSPECIFIED DUODENAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION 532.7 CHRONIC DUODENAL ULCER WITHOUT MENTION OF HEMORRHAGE OR PERFORATION
- 532.9 DUODENAL ULCER UNSPECIFIED AS ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION 533.21 ACUTE PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION 533.4 CHRONIC OR UNSPECIFIED PEPTIC ULCER OF UNSPECIFIED SITE WITH HEMORRHAGE

| 533.40 - CHRONIC | OR UNSPECIFIED PEPTIC ULCER OF |
|------------------|--------------------------------|

UNSPECIFIED SITE WITH HEMORRHAGE WITHOUT OBSTRUCTION

533.41 - CHRONIC OR UNSPECIFIED PEPTIC ULCER OF

UNSPECIFIED SITE WITH HEMORRHAGE WITH OBSTRUCTION

533.5 - CHRONIC OR UNSPECIFIED PEPTIC ULCER OF

UNSPECIFIED SITE WITH PERFORATION

533.61 - CHRONIC OR UNSPECIFIED PEPTIC ULCER OF

UNSPECIFIED SITE WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION

533.9 - PEPTIC ULCER OF UNSPECIFIED SITE UNSPECIFIED AS

ACUTE OR CHRONIC WITHOUT MENTION OF HEMORRHAGE OR PERFORATION

534.0 - ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE

534.1 - ACUTE GASTROJEJUNAL ULCER WITH PERFORATION

534.2 - ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION

534.21 - ACUTE GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITH OBSTRUCTION

534.4 - CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE

534.5 - CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH PERFORATION

534.6 - CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION

534.60 - CHRONIC OR UNSPECIFIED GASTROJEJUNAL ULCER WITH HEMORRHAGE AND PERFORATION WITHOUT OBSTRUCTION

535.11 - ATROPHIC GASTRITIS WITH HEMORRHAGE

535.30 - ALCOHOLIC GASTRITIS (WITHOUT HEMORRHAGE)

535.50 - UNSPECIFIED GASTRITIS AND GASTRODUODENITIS (WITHOUT HEMORRHAGE)

535.51 - UNSPECIFIED GASTRITIS AND GASTRODUODENITIS WITH HEMORRHAGE

535.60 - DUODENITIS (WITHOUT HEMORRHAGE)

535.61 - DUODENITIS WITH HEMORRHAGE 537.83 - ANGIODYSPLASIA OF STOMACH AND DUODENUM WITH **HEMORRHAGE** 562.02 - DIVERTICULOSIS OF SMALL INTESTINE WITH **HEMORRHAGE** 562.10 - DIVERTICULOSIS OF COLON (WITHOUT HEMORRHAGE) 562.12 - DIVERTICULOSIS OF COLON WITH HEMORRHAGE 569.3 - HEMORRHAGE OF RECTUM AND ANUS 623.8 - OTHER SPECIFIED NONINFLAMMATORY DISORDERS OF **VAGINA** 626.8 - OTHER DISORDERS OF MENSTRUATION AND OTHER ABNORMAL BLEEDING FROM FEMALE GENITAL TRACT 786.3 - HEMOPTYSIS 786.30 - HEMOPTYSIS UNSPECIFIED 786.39 - OTHER HEMOPTYSIS 285.9 - ANEMIA UNSPECIFIED 790.92 - ABNORMAL COAGULATION PROFILE 363.63 - CHOROIDAL RUPTURE 626.2 - EXCESSIVE OR FREQUENT MENSTRUATION 372.72 - CONJUNCTIVAL HEMORRHAGE Inpatient, Primary Diagnosis: ICD-10 Codes D50.0 - Iron deficiency anemia secondary to blood loss (chronic) D62 - Acute posthemorrhagic anemia 185.01 - Esophageal varices with bleeding 185.11 - Secondary esophageal varices with bleeding K20.0 - Eosinophilic esophagitis K20.8 - Other esophagitis K22.11 - Ulcer of esophagus with bleeding K22.6 - Gastro-esophageal laceration-hemorrhage syndrome K25.0 - Acute gastric ulcer with hemorrhage K25.1 - Acute gastric ulcer with perforation K25.2 - Acute gastric ulcer with both hemorrhage and perforation

- K25.4 Chronic or unspecified gastric ulcer with hemorrhage
- K25.5 Chronic or unspecified gastric ulcer with perforation
- K26.1 Acute duodenal ulcer with perforation
- K26.2 Acute duodenal ulcer with both hemorrhage and perforation
- K26.4 Chronic or unspecified duodenal ulcer with hemorrhage
- K27.1 Acute peptic ulcer, site unspecified, with perforation
- K27.2 Acute peptic ulcer, site unspecified, with both hemorrhage and perforation
- K27.5 Chronic or unspecified peptic ulcer, site unspecified, with perforation
- K27.6 Chronic or unspecified peptic ulcer, site unspecified, with both hemorrhage and perforation
- K28.0 Acute gastrojejunal ulcer with hemorrhage
- K28.4 Chronic or unspecified gastrojejunal ulcer with hemorrhage
- K28.6 Chronic or unspecified gastrojejunal ulcer with both hemorrhage and perforation
- K29.01 Acute gastritis with bleeding
- K29.31 Chronic superficial gastritis with bleeding
- K29.41 Chronic atrophic gastritis with bleeding
- K29.51 Unspecified chronic gastritis with bleeding
- K29.71 Gastritis, unspecified, with bleeding
- K57.11 Diverticulosis of small intestine without perforation or abscess with bleeding
- K57.21 Diverticulitis of large intestine with perforation and abscess with bleeding
- K57.41 Diverticulitis of both small and large intestine with perforation and abscess with bleeding
- K57.51 Diverticulosis of both small and large intestine without perforation or abscess with bleeding
- K57.81 Diverticulitis of intestine, part unspecified, with perforation and abscess with bleeding
- K57.91 Diverticulosis of intestine, part unspecified, without perforation or abscess with bleeding
- K57.93 Diverticulitis of intestine, part unspecified, without perforation or abscess with bleeding

- K62.5 Hemorrhage of anus and rectum
- K64.0 First degree hemorrhoids
- K64.5 Perianal venous thrombosis
- K64.8 Other hemorrhoids
- K64.9 Unspecified hemorrhoids
- K92.0 Hematemesis
- K92.2 Gastrointestinal hemorrhage, unspecified
- N89.7 Hematocolpos
- N93.8 Other specified abnormal uterine and vaginal bleeding
- R04.2 Hemoptysis
- R31.0 Gross hematuria
- K20 Esophagitis
- K20.9 Esophagitis, unspecified
- K21.0 Gastro-esophageal reflux disease with esophagitis
- K25.6 Chronic or unspecified gastric ulcer with both hemorrhage and perforation
- K26.0 Acute duodenal ulcer with hemorrhage
- K26.5 Chronic or unspecified duodenal ulcer with perforation
- K26.6 Chronic or unspecified duodenal ulcer with both hemorrhage and perforation
- K27.0 Acute peptic ulcer, site unspecified, with hemorrhage
- K27.4 Chronic or unspecified peptic ulcer, site unspecified, with hemorrhage
- K28.1 Acute gastrojejunal ulcer with perforation
- K28.2 Acute gastrojejunal ulcer with both hemorrhage and perforation
- K28.5 Chronic or unspecified gastrojejunal ulcer with perforation
- K29.21 Alcoholic gastritis with bleeding
- K29.61 Other gastritis with bleeding
- K29.81 Duodenitis with bleeding
- K29.91 Gastroduodenitis, unspecified, with bleeding
- K31.811 Angiodysplasia of stomach and duodenum with bleeding
- K55.21 Angiodysplasia of colon with hemorrhage

- K57.01 Diverticulitis of small intestine with perforation and abscess with bleeding
- K57.31 Diverticulosis of large intestine without perforation or abscess with bleeding
- K57.53 Diverticulitis of both small and large intestine without perforation or abscess with bleeding
- K64.1 Second degree hemorrhoids
- K64.2 Third degree hemorrhoids
- K64.3 Fourth degree hemorrhoids
- K64.4 Residual hemorrhoidal skin tags
- K92.1 Melena
- N89.8 Other specified noninflammatory disorders of vagina
- N93.9 Abnormal uterine and vaginal bleeding, unspecified
- R04.0 Epistaxis
- R04.1 Hemorrhage from throat
- R58 Hemorrhage, not elsewhere classified
- D64.9 Anemia, unspecified
- R79.1 Abnormal coagulation profile
- H11.30 Conjunctival hemorrhage, unspecified eye
- H11.31 Conjunctival hemorrhage, right eye
- H11.32 Conjunctival hemorrhage, left eye
- H11.33 Conjunctival hemorrhage, bilateral
- H31.321 Choroidal rupture, right eye
- H31.322 Choroidal rupture, left eye
- H31.323 Choroidal rupture, bilateral
- H31.329 Choroidal rupture, unspecified eye
- N92.1 Excessive and frequent menstruation with irregular cycle
- R31.1 Benign essential microscopic hematuria
- R31.2 Other microscopic hematuria
- R31.29 Other microscopic hematuria
- N92.0 Excessive and frequent menstruation with regular cycle
- R31.21 Asymptomatic microscopic hematuria
- R31.9 Hematuria, unspecified


TUMOR OF BONE

209.7 - SECONDARY NEUROENDOCRINE TUMORS

209.71 - SECONDARY NEUROENDOCRINE TUMOR OF DISTANT LYMPH NODES 209.73 - SECONDARY NEUROENDOCRINE

209.74 - SECONDARY NEUROENDOCRINE TUMOR OF PERITONEUM

C50.62 - Malignant neoplasm of axillary tail of breast, male C50.622 - Malignant neoplasm of axillary tail of left male breast

C50.8 - Malignant neoplasm of overlapping sites of breast C50.819 - Malignant neoplasm of overlapping sites of unspecified female breast

C50.82 - Malignant neoplasm of overlapping sites of breast, male

C50.821 - Malignant neoplasm of overlapping sites of right male breast

C50.822 - Malignant neoplasm of overlapping sites of left male breast

C50.9 - Malignant neoplasm of breast of unspecified site

C50.91 - Malignant neoplasm of breast of unspecified site, female

C50.911 - Malignant neoplasm of unspecified site of right female breast

C50.919 - Malignant neoplasm of unspecified site of unspecified female breast

C52 - Malignant neoplasm of vagina

C53 - Malignant neoplasm of cervix uteri

C53.1 - Malignant neoplasm of exocervix

C53.8 - Malignant neoplasm of overlapping sites of cervix uteri

C53.9 - Malignant neoplasm of cervix uteri, unspecified

C54 - Malignant neoplasm of corpus uteri

C54.0 - Malignant neoplasm of isthmus uteri

C54.8 - Malignant neoplasm of overlapping sites of corpus uteri

C54.9 - Malignant neoplasm of corpus uteri, unspecified

- C55 Malignant neoplasm of uterus, part unspecified
- C56.1 Malignant neoplasm of right ovary
- C56.2 Malignant neoplasm of left ovary
- C56.9 Malignant neoplasm of unspecified ovary
- C57 Malignant neoplasm of other and unspecified female genital organs
- C57.0 Malignant neoplasm of fallopian tube
- C57.01 Malignant neoplasm of right fallopian tube
- C57.10 Malignant neoplasm of unspecified broad ligament
- C57.2 Malignant neoplasm of round ligament
- C57.20 Malignant neoplasm of unspecified round ligament
- C57.21 Malignant neoplasm of right round ligament
- C57.22 Malignant neoplasm of left round ligament
- C57.3 Malignant neoplasm of parametrium
- C57.4 Malignant neoplasm of uterine adnexa, unspecified
- C57.7 Malignant neoplasm of other specified female genital organs
- C58 Malignant neoplasm of placenta
- C60 Malignant neoplasm of penis
- C60.2 Malignant neoplasm of body of penis
- C60.8 Malignant neoplasm of overlapping sites of penis
- C62 Malignant neoplasm of testis
- C62.0 Malignant neoplasm of undescended testis
- C62.1 Malignant neoplasm of descended testis
- C62.10 Malignant neoplasm of unspecified descended testis
- C62.11 Malignant neoplasm of descended right testis
- C62.91 Malignant neoplasm of right testis, unspecified whether descended or undescended

- C63 Malignant neoplasm of other and unspecified male genital organs
- C63.0 Malignant neoplasm of epididymis
- C63.00 Malignant neoplasm of unspecified epididymis
- C63.01 Malignant neoplasm of right epididymis
- C63.1 Malignant neoplasm of spermatic cord
- C63.10 Malignant neoplasm of unspecified spermatic cord
- C63.11 Malignant neoplasm of right spermatic cord
- C63.12 Malignant neoplasm of left spermatic cord
- C63.7 Malignant neoplasm of other specified male genital organs
- C63.9 Malignant neoplasm of male genital organ, unspecified
- C64.1 Malignant neoplasm of right kidney, except renal pelvis
- C64.9 Malignant neoplasm of unspecified kidney, except renal pelvis
- C65 Malignant neoplasm of renal pelvis
- C65.1 Malignant neoplasm of right renal pelvis
- C66.9 Malignant neoplasm of unspecified ureter
- C67.0 Malignant neoplasm of trigone of bladder
- C67.1 Malignant neoplasm of dome of bladder
- C67.4 Malignant neoplasm of posterior wall of bladder
- C67.5 Malignant neoplasm of bladder neck
- C67.7 Malignant neoplasm of urachus
- C67.8 Malignant neoplasm of overlapping sites of bladder
- C67.9 Malignant neoplasm of bladder, unspecified
- C68.0 Malignant neoplasm of urethra
- C68.1 Malignant neoplasm of paraurethral glands
- C68.8 Malignant neoplasm of overlapping sites of urinary organs

- C69 Malignant neoplasm of eye and adnexa
- C69.0 Malignant neoplasm of conjunctiva
- C69.00 Malignant neoplasm of unspecified conjunctiva
- C69.01 Malignant neoplasm of right conjunctiva
- C69.02 Malignant neoplasm of left conjunctiva
- C69.10 Malignant neoplasm of unspecified cornea
- C69.11 Malignant neoplasm of right cornea
- C69.2 Malignant neoplasm of retina
- C69.20 Malignant neoplasm of unspecified retina
- C69.22 Malignant neoplasm of left retina
- C69.31 Malignant neoplasm of right choroid
- C69.4 Malignant neoplasm of ciliary body
- C69.40 Malignant neoplasm of unspecified ciliary body
- C69.41 Malignant neoplasm of right ciliary body
- C69.42 Malignant neoplasm of left ciliary body
- C69.50 Malignant neoplasm of unspecified lacrimal gland and duct
- C69.6 Malignant neoplasm of orbit
- C69.61 Malignant neoplasm of right orbit
- C69.62 Malignant neoplasm of left orbit
- C69.8 Malignant neoplasm of overlapping sites of eye and adnexa
- C69.80 Malignant neoplasm of overlapping sites of unspecified eye and adnexa
- C69.9 Malignant neoplasm of unspecified site of eye
- C69.90 Malignant neoplasm of unspecified site of unspecified eye
- C71.0 Malignant neoplasm of cerebrum, except lobes and ventricles
- C71.1 Malignant neoplasm of frontal lobe
- C72.1 Malignant neoplasm of cauda equina
- C72.2 Malignant neoplasm of olfactory nerve

- C72.20 Malignant neoplasm of unspecified olfactory nerve
- C72.21 Malignant neoplasm of right olfactory nerve
- C72.22 Malignant neoplasm of left olfactory nerve
- C72.31 Malignant neoplasm of right optic nerve
- C72.42 Malignant neoplasm of left acoustic nerve
- C72.5 Malignant neoplasm of other and unspecified cranial nerves
- C74.0 Malignant neoplasm of cortex of adrenal gland
- C74.02 Malignant neoplasm of cortex of left adrenal gland
- C74.1 Malignant neoplasm of medulla of adrenal gland
- C74.11 Malignant neoplasm of medulla of right adrenal gland
- C74.12 Malignant neoplasm of medulla of left adrenal gland
- C74.9 Malignant neoplasm of unspecified part of adrenal gland
- C74.90 Malignant neoplasm of unspecified part of unspecified adrenal gland
- C74.91 Malignant neoplasm of unspecified part of right adrenal gland
- C75.1 Malignant neoplasm of pituitary gland
- C75.2 Malignant neoplasm of craniopharyngeal duct
- C75.3 Malignant neoplasm of pineal gland
- C75.5 Malignant neoplasm of aortic body and other paraganglia
- C76 Malignant neoplasm of other and ill-defined sites
- C76.0 Malignant neoplasm of head, face and neck
- C76.1 Malignant neoplasm of thorax
- C76.2 Malignant neoplasm of abdomen
- C76.3 Malignant neoplasm of pelvis

- C76.4 Malignant neoplasm of upper limb
- C77 Secondary and unspecified malignant neoplasm of lymph nodes
- C77.3 Secondary and unspecified malignant neoplasm of axilla and upper limb lymph nodes
- C77.4 Secondary and unspecified malignant neoplasm of inguinal and lower limb lymph nodes
- C77.5 Secondary and unspecified malignant neoplasm of intrapelvic lymph nodes
- C77.8 Secondary and unspecified malignant neoplasm of lymph nodes of multiple regions
- C78.0 Secondary malignant neoplasm of lung
- C78.01 Secondary malignant neoplasm of right lung
- C78.02 Secondary malignant neoplasm of left lung
- C78.3 Secondary malignant neoplasm of other and unspecified respiratory organs
- C78.4 Secondary malignant neoplasm of small intestine
- C78.8 Secondary malignant neoplasm of other and unspecified digestive organs
- C79 Secondary malignant neoplasm of other and unspecified sites
- C79.0 Secondary malignant neoplasm of kidney and renal pelvis
- C79.00 Secondary malignant neoplasm of unspecified kidney and renal pelvis
- C79.01 Secondary malignant neoplasm of right kidney and renal pelvis
- C79.1 Secondary malignant neoplasm of bladder and other and unspecified urinary organs
- C79.10 Secondary malignant neoplasm of unspecified urinary organs
- C79.19 Secondary malignant neoplasm of other urinary organs

- C79.32 Secondary malignant neoplasm of cerebral meninges
- C79.4 Secondary malignant neoplasm of other and unspecified parts of nervous system
- C79.40 Secondary malignant neoplasm of unspecified part of nervous system
- C79.49 Secondary malignant neoplasm of other parts of nervous system
- C79.51 Secondary malignant neoplasm of bone
- C79.52 Secondary malignant neoplasm of bone marrow C79.60 Secondary malignant neoplasm of unspecified ovary
- C79.61 Secondary malignant neoplasm of right ovary C79.71 Secondary malignant neoplasm of right adrenal gland
- C79.82 Secondary malignant neoplasm of genital organs C79.89 Secondary malignant neoplasm of other specified sites
- C80.0 Disseminated malignant neoplasm, unspecified
- C80.1 Malignant (primary) neoplasm, unspecified
- C80.2 Malignant neoplasm associated with transplanted organ
- C81.00 Nodular lymphocyte predominant Hodgkin lymphoma, unspecified site
- C81.03 Nodular lymphocyte predominant Hodgkin lymphoma, intra-abdominal lymph nodes
- C81.05 Nodular lymphocyte predominant Hodgkin lymphoma, lymph nodes of inguinal region and lower limb C81.08 Nodular lymphocyte predominant Hodgkin lymphoma, lymph nodes of multiple sites

- C81.10 Nodular sclerosis Hodgkin lymphoma, unspecified site
- C81.11 Nodular sclerosis Hodgkin lymphoma, lymph nodes of head, face, and neck
- C81.13 Nodular sclerosis Hodgkin lymphoma, intraabdominal lymph nodes
- C81.21 Mixed cellularity Hodgkin lymphoma, lymph nodes of head, face, and neck
- C81.23 Mixed cellularity Hodgkin lymphoma, intraabdominal lymph nodes
- C81.25 Mixed cellularity Hodgkin lymphoma, lymph nodes of inguinal region and lower limb
- C81.28 Mixed cellularity Hodgkin lymphoma, lymph nodes of multiple sites
- C81.29 Mixed cellularity Hodgkin lymphoma, extranodal and solid organ sites
- C81.3 Lymphocyte depleted Hodgkin lymphoma
- C81.32 Lymphocyte depleted Hodgkin lymphoma, intrathoracic lymph nodes
- C81.33 Lymphocyte depleted Hodgkin lymphoma, intraabdominal lymph nodes
- C81.35 Lymphocyte depleted Hodgkin lymphoma, lymph nodes of inguinal region and lower limb
- C81.37 Lymphocyte depleted Hodgkin lymphoma, spleen
- C81.39 Lymphocyte depleted Hodgkin lymphoma, extranodal and solid organ sites
- C81.40 Lymphocyte-rich Hodgkin lymphoma, unspecified site
- C81.45 Lymphocyte-rich Hodgkin lymphoma, lymph nodes of inquinal region and lower limb
- C81.46 Lymphocyte-rich Hodgkin lymphoma, intrapelvic lymph nodes
- C81.47 Lymphocyte-rich Hodgkin lymphoma, spleen

- C81.48 Lymphocyte-rich Hodgkin lymphoma, lymph nodes of multiple sites
- C81.49 Lymphocyte-rich Hodgkin lymphoma, extranodal and solid organ sites
- C81.74 Other Hodgkin lymphoma, lymph nodes of axilla and upper limb
- C81.76 Other Hodgkin lymphoma, intrapelvic lymph nodes
- C81.77 Other Hodgkin lymphoma, spleen
- C81.78 Other Hodgkin lymphoma, lymph nodes of multiple sites
- C81.9 Hodgkin lymphoma, unspecified
- C81.92 Hodgkin lymphoma, unspecified, intrathoracic lymph nodes
- C81.93 Hodgkin lymphoma, unspecified, intra-abdominal lymph nodes
- C81.95 Hodgkin lymphoma, unspecified, lymph nodes of inguinal region and lower limb
- C81.99 Hodgkin lymphoma, unspecified, extranodal and solid organ sites
- C82.0 Follicular lymphoma grade I
- C82.00 Follicular lymphoma grade I, unspecified site
- C82.01 Follicular lymphoma grade I, lymph nodes of head, face, and neck
- C82.02 Follicular lymphoma grade I, intrathoracic lymph nodes
- C82.03 Follicular lymphoma grade I, intra-abdominal lymph nodes
- C82.04 Follicular lymphoma grade I, lymph nodes of axilla and upper limb
- C82.10 Follicular lymphoma grade II, unspecified site
- C82.11 Follicular lymphoma grade II, lymph nodes of head, face, and neck

- C82.13 Follicular lymphoma grade II, intra-abdominal lymph nodes
- C82.16 Follicular lymphoma grade II, intrapelvic lymph nodes
- C82.17 Follicular lymphoma grade II, spleen
- C82.22 Follicular lymphoma grade III, unspecified, intrathoracic lymph nodes
- C82.23 Follicular lymphoma grade III, unspecified, intraabdominal lymph nodes
- C82.26 Follicular lymphoma grade III, unspecified, intrapelvic lymph nodes
- C82.27 Follicular lymphoma grade III, unspecified, spleen
- C82.3 Follicular lymphoma grade IIIa
- C82.30 Follicular lymphoma grade IIIa, unspecified site
- C82.31 Follicular lymphoma grade IIIa, lymph nodes of head, face, and neck
- C82.34 Follicular lymphoma grade IIIa, lymph nodes of axilla and upper limb
- C82.36 Follicular lymphoma grade IIIa, intrapelvic lymph nodes
- C82.37 Follicular lymphoma grade IIIa, spleen
- C82.38 Follicular lymphoma grade IIIa, lymph nodes of multiple sites
- C82.4 Follicular lymphoma grade IIIb
- C82.40 Follicular lymphoma grade IIIb, unspecified site
- C82.41 Follicular lymphoma grade IIIb, lymph nodes of head, face, and neck
- C82.42 Follicular lymphoma grade IIIb, intrathoracic lymph nodes
- C82.43 Follicular lymphoma grade IIIb, intra-abdominal lymph nodes
- C82.45 Follicular lymphoma grade IIIb, lymph nodes of inguinal region and lower limb
- C82.48 Follicular lymphoma grade IIIb, lymph nodes of multiple sites
- C82.49 Follicular lymphoma grade IIIb, extranodal and solid organ sites
- C82.5 Diffuse follicle center lymphoma
- C82.50 Diffuse follicle center lymphoma, unspecified site
- C82.53 Diffuse follicle center lymphoma, intra-abdominal lymph nodes
- C82.54 Diffuse follicle center lymphoma, lymph nodes of axilla and upper limb
- C82.57 Diffuse follicle center lymphoma, spleen
- C82.58 Diffuse follicle center lymphoma, lymph nodes of multiple sites
- C82.6 Cutaneous follicle center lymphoma
- C82.64 Cutaneous follicle center lymphoma, lymph nodes of axilla and upper limb
- C82.65 Cutaneous follicle center lymphoma, lymph nodes of inguinal region and lower limb
- C82.66 Cutaneous follicle center lymphoma, intrapelvic lymph nodes
- C82.67 Cutaneous follicle center lymphoma, spleen
- C82.81 Other types of follicular lymphoma, lymph nodes of head, face, and neck
- C82.82 Other types of follicular lymphoma, intrathoracic lymph nodes
- C82.83 Other types of follicular lymphoma, intraabdominal lymph nodes
- C82.84 Other types of follicular lymphoma, lymph nodes of axilla and upper limb
- C82.85 Other types of follicular lymphoma, lymph nodes of inguinal region and lower limb

C82.88 - Other types of follicular lymphoma, lymph nodes of multiple sites

C82.9 - Follicular lymphoma, unspecified

C82.90 - Follicular lymphoma, unspecified, unspecified site

C82.91 - Follicular lymphoma, unspecified, lymph nodes of head, face, and neck

C82.93 - Follicular lymphoma, unspecified, intra-abdominal lymph nodes

C82.94 - Follicular lymphoma, unspecified, lymph nodes of axilla and upper limb

C83 - Non-follicular lymphoma

C83.0 - Small cell B-cell lymphoma

C83.04 - Small cell B-cell lymphoma, lymph nodes of axilla and upper limb

C83.05 - Small cell B-cell lymphoma, lymph nodes of inguinal region and lower limb

C83.09 - Small cell B-cell lymphoma, extranodal and solid organ sites

C83.1 - Mantle cell lymphoma

C83.10 - Mantle cell lymphoma, unspecified site

C83.13 - Mantle cell lymphoma, intra-abdominal lymph nodes

C83.15 - Mantle cell lymphoma, lymph nodes of inguinal region and lower limb

C83.16 - Mantle cell lymphoma, intrapelvic lymph nodes

C83.3 - Diffuse large B-cell lymphoma

C83.32 - Diffuse large B-cell lymphoma, intrathoracic lymph nodes

C83.33 - Diffuse large B-cell lymphoma, intra-abdominal lymph nodes

C83.39 - Diffuse large B-cell lymphoma, extranodal and solid organ sites

- C83.51 Lymphoblastic (diffuse) lymphoma, lymph nodes of head, face, and neck
- C83.54 Lymphoblastic (diffuse) lymphoma, lymph nodes of axilla and upper limb
- C83.55 Lymphoblastic (diffuse) lymphoma, lymph nodes of inguinal region and lower limb
- C83.57 Lymphoblastic (diffuse) lymphoma, spleen
- C83.7 Burkitt lymphoma
- C83.70 Burkitt lymphoma, unspecified site
- C83.71 Burkitt lymphoma, lymph nodes of head, face, and neck
- C83.73 Burkitt lymphoma, intra-abdominal lymph nodes
- C83.74 Burkitt lymphoma, lymph nodes of axilla and upper limb
- C83.75 Burkitt lymphoma, lymph nodes of inguinal region and lower limb
- C83.78 Burkitt lymphoma, lymph nodes of multiple sites
- C83.81 Other non-follicular lymphoma, lymph nodes of head, face, and neck
- C83.82 Other non-follicular lymphoma, intrathoracic lymph nodes
- C83.85 Other non-follicular lymphoma, lymph nodes of inguinal region and lower limb
- C83.86 Other non-follicular lymphoma, intrapelvic lymph nodes
- C83.87 Other non-follicular lymphoma, spleen
- C83.88 Other non-follicular lymphoma, lymph nodes of multiple sites
- C83.91 Non-follicular (diffuse) lymphoma, unspecified, lymph nodes of head, face, and neck
- C83.94 Non-follicular (diffuse) lymphoma, unspecified, lymph nodes of axilla and upper limb

C83.96 - Non-follicular (diffuse) lymphoma, unspecified, intrapelvic lymph nodes

C83.97 - Non-follicular (diffuse) lymphoma, unspecified, spleen

C83.98 - Non-follicular (diffuse) lymphoma, unspecified, lymph nodes of multiple sites

C83.99 - Non-follicular (diffuse) lymphoma, unspecified, extranodal and solid organ sites

C84 - Mature T/NK-cell lymphomas

C84.0 - Mycosis fungoides

C84.00 - Mycosis fungoides, unspecified site

C84.01 - Mycosis fungoides, lymph nodes of head, face, and neck

C84.03 - Mycosis fungoides, intra-abdominal lymph nodes

C84.04 - Mycosis fungoides, lymph nodes of axilla and upper limb

C84.05 - Mycosis fungoides, lymph nodes of inguinal region and lower limb

C84.06 - Mycosis fungoides, intrapelvic lymph nodes

C84.08 - Mycosis fungoides, lymph nodes of multiple sites

C84.09 - Mycosis fungoides, extranodal and solid organ sites

C84.1 - Sezary disease

C84.10 - Sezary disease, unspecified site

C84.12 - Sezary disease, intrathoracic lymph nodes

C84.14 - Sezary disease, lymph nodes of axilla and upper limb

C84.16 - Sezary disease, intrapelvic lymph nodes

C84.19 - Sezary disease, extranodal and solid organ sites

C84.40 - Peripheral T-cell lymphoma, not classified, unspecified site

- C84.46 Peripheral T-cell lymphoma, not classified, intrapelvic lymph nodes
- C84.47 Peripheral T-cell lymphoma, not classified, spleen
- C84.6 Anaplastic large cell lymphoma, ALK-positive
- C84.60 Anaplastic large cell lymphoma, ALK-positive, unspecified site
- C84.62 Anaplastic large cell lymphoma, ALK-positive, intrathoracic lymph nodes
- C84.63 Anaplastic large cell lymphoma, ALK-positive, intra-abdominal lymph nodes
- C84.64 Anaplastic large cell lymphoma, ALK-positive, lymph nodes of axilla and upper limb
- C84.65 Anaplastic large cell lymphoma, ALK-positive, lymph nodes of inguinal region and lower limb
- C84.67 Anaplastic large cell lymphoma, ALK-positive, spleen
- C84.68 Anaplastic large cell lymphoma, ALK-positive, lymph nodes of multiple sites
- C84.69 Anaplastic large cell lymphoma, ALK-positive, extranodal and solid organ sites
- C84.70 Anaplastic large cell lymphoma, ALK-negative, unspecified site
- C84.72 Anaplastic large cell lymphoma, ALK-negative, intrathoracic lymph nodes
- C84.73 Anaplastic large cell lymphoma, ALK-negative, intra-abdominal lymph nodes
- C84.77 Anaplastic large cell lymphoma, ALK-negative, spleen
- C84.78 Anaplastic large cell lymphoma, ALK-negative, lymph nodes of multiple sites
- C84.90 Mature T/NK-cell lymphomas, unspecified, unspecified site

- C84.91 Mature T/NK-cell lymphomas, unspecified, lymph nodes of head, face, and neck
- C84.92 Mature T/NK-cell lymphomas, unspecified, intrathoracic lymph nodes
- C84.A0 Cutaneous T-cell lymphoma, unspecified, unspecified site
- C84.A1 Cutaneous T-cell lymphoma, unspecified lymph nodes of head, face, and neck
- C84.A2 Cutaneous T-cell lymphoma, unspecified, intrathoracic lymph nodes
- C84.A3 Cutaneous T-cell lymphoma, unspecified, intraabdominal lymph nodes
- C84.A5 Cutaneous T-cell lymphoma, unspecified, lymph nodes of inguinal region and lower limb
- C84.A7 Cutaneous T-cell lymphoma, unspecified, spleen
- C84.Z Other mature T/NK-cell lymphomas
- C84.Z1 Other mature T/NK-cell lymphomas, lymph nodes of head, face, and neck
- C84.Z4 Other mature T/NK-cell lymphomas, lymph nodes of axilla and upper limb
- C84.Z6 Other mature T/NK-cell lymphomas, intrapelvic lymph nodes
- C84.Z8 Other mature T/NK-cell lymphomas, lymph nodes of multiple sites
- C85.1 Unspecified B-cell lymphoma
- C85.12 Unspecified B-cell lymphoma, intrathoracic lymph nodes
- C85.13 Unspecified B-cell lymphoma, intra-abdominal lymph nodes
- C85.15 Unspecified B-cell lymphoma, lymph nodes of inguinal region and lower limb
- C85.17 Unspecified B-cell lymphoma, spleen
- C85.18 Unspecified B-cell lymphoma, lymph nodes of multiple sites

C85.19 - Unspecified B-cell lymphoma, extranodal and solid organ sites

C85.22 - Mediastinal (thymic) large B-cell lymphoma, intrathoracic lymph nodes

C85.26 - Mediastinal (thymic) large B-cell lymphoma, intrapelvic lymph nodes

C85.8 - Other specified types of non-Hodgkin lymphoma C85.80 - Other specified types of non-Hodgkin lymphoma,

unspecified site

C85.86 - Other specified types of non-Hodgkin lymphoma, intrapelvic lymph nodes

C85.87 - Other specified types of non-Hodgkin lymphoma, spleen

C85.89 - Other specified types of non-Hodgkin lymphoma, extranodal and solid organ sites

C85.91 - Non-Hodgkin lymphoma, unspecified, lymph nodes of head, face, and neck

C85.92 - Non-Hodgkin lymphoma, unspecified, intrathoracic lymph nodes

C85.93 - Non-Hodgkin lymphoma, unspecified, intraabdominal lymph nodes

C85.96 - Non-Hodgkin lymphoma, unspecified, intrapelvic lymph nodes

C85.97 - Non-Hodgkin lymphoma, unspecified, spleen

C85.98 - Non-Hodgkin lymphoma, unspecified, lymph nodes of multiple sites

C85.99 - Non-Hodgkin lymphoma, unspecified, extranodal and solid organ sites

C86 - Other specified types of T/NK-cell lymphoma

C86.0 - Extranodal NK/T-cell lymphoma, nasal type

C86.3 - Subcutaneous panniculitis-like T-cell lymphoma

C86.4 - Blastic NK-cell lymphoma

- C86.5 Angioimmunoblastic T-cell lymphoma
- C86.6 Primary cutaneous CD30-positive T-cell proliferations
- C88.0 Waldenstrom macroglobulinemia
- C88.2 Heavy chain disease
- C88.4 Extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue [MALT-lymphoma]
- C88.8 Other malignant immunoproliferative diseases
- C90 Multiple myeloma and malignant plasma cell neoplasms
- C90.00 Multiple myeloma not having achieved remission
- C90.02 Multiple myeloma in relapse
- C90.1 Plasma cell leukemia
- C90.10 Plasma cell leukemia not having achieved remission
- C90.12 Plasma cell leukemia in relapse
- C90.21 Extramedullary plasmacytoma in remission
- C90.22 Extramedullary plasmacytoma in relapse
- C90.31 Solitary plasmacytoma in remission
- C90.32 Solitary plasmacytoma in relapse
- C91 Lymphoid leukemia
- C91.01 Acute lymphoblastic leukemia, in remission
- C91.02 Acute lymphoblastic leukemia, in relapse
- C91.1 Chronic lymphocytic leukemia of B-cell type
- C91.10 Chronic lymphocytic leukemia of B-cell type not having achieved remission
- C91.12 Chronic lymphocytic leukemia of B-cell type in relapse
- C91.30 Prolymphocytic leukemia of B-cell type not having achieved remission
- C91.32 Prolymphocytic leukemia of B-cell type, in relapse

- C91.42 Hairy cell leukemia, in relapse
- C91.51 Adult T-cell lymphoma/leukemia (HTLV-1-associated), in remission
- C91.52 Adult T-cell lymphoma/leukemia (HTLV-1-associated), in relapse
- C91.62 Prolymphocytic leukemia of T-cell type, in relapse
- C91.9 Lymphoid leukemia, unspecified
- C91.90 Lymphoid leukemia, unspecified not having achieved remission
- C91.92 Lymphoid leukemia, unspecified, in relapse
- C91.A Mature B-cell leukemia Burkitt-type
- C91.A0 Mature B-cell leukemia Burkitt-type not having achieved remission
- C91.A2 Mature B-cell leukemia Burkitt-type, in relapse
- C91.Z0 Other lymphoid leukemia not having achieved remission
- C91.Z1 Other lymphoid leukemia, in remission
- C92 Myeloid leukemia
- C92.0 Acute myeloblastic leukemia
- C92.10 Chronic myeloid leukemia, BCR/ABL-positive, not having achieved remission
- C92.12 Chronic myeloid leukemia, BCR/ABL-positive, in relapse
- C92.2 Atypical chronic myeloid leukemia, BCR/ABL-negative
- C92.20 Atypical chronic myeloid leukemia, BCR/ABL-negative, not having achieved remission
- C92.22 Atypical chronic myeloid leukemia, BCR/ABL-negative, in relapse
- C92.31 Myeloid sarcoma, in remission
- C92.32 Myeloid sarcoma, in relapse
- C92.40 Acute promyelocytic leukemia, not having achieved remission

- C92.5 Acute myelomonocytic leukemia
- C92.50 Acute myelomonocytic leukemia, not having achieved remission
- C92.51 Acute myelomonocytic leukemia, in remission
- C92.52 Acute myelomonocytic leukemia, in relapse
- C92.6 Acute myeloid leukemia with 11q23-abnormality
- C92.62 Acute myeloid leukemia with 11q23-abnormality in relapse
- C92.92 Myeloid leukemia, unspecified in relapse
- C92.A Acute myeloid leukemia with multilineage dysplasia
- C92.Z1 Other myeloid leukemia, in remission
- C92.Z2 Other myeloid leukemia, in relapse
- C93 Monocytic leukemia
- C93.00 Acute monoblastic/monocytic leukemia, not having achieved remission
- C93.02 Acute monoblastic/monocytic leukemia, in relapse
- C93.10 Chronic myelomonocytic leukemia not having achieved remission
- C93.11 Chronic myelomonocytic leukemia, in remission
- C93.9 Monocytic leukemia, unspecified
- C93.91 Monocytic leukemia, unspecified in remission
- C93.Z0 Other monocytic leukemia, not having achieved remission
- C93.Z2 Other monocytic leukemia, in relapse
- C94 Other leukemias of specified cell type
- C94.00 Acute erythroid leukemia, not having achieved remission
- C94.01 Acute erythroid leukemia, in remission
- C94.02 Acute erythroid leukemia, in relapse

- C94.2 Acute megakaryoblastic leukemia
- C94.30 Mast cell leukemia not having achieved remission
- C94.31 Mast cell leukemia, in remission
- C94.32 Mast cell leukemia, in relapse
- C94.41 Acute panmyelosis with myelofibrosis, in remission
- C94.8 Other specified leukemias
- C94.80 Other specified leukemias not having achieved remission
- C94.81 Other specified leukemias, in remission
- C94.82 Other specified leukemias, in relapse
- C95.00 Acute leukemia of unspecified cell type not having achieved remission
- C95.01 Acute leukemia of unspecified cell type, in remission
- C95.02 Acute leukemia of unspecified cell type, in relapse
- C95.10 Chronic leukemia of unspecified cell type not having achieved remission
- C95.11 Chronic leukemia of unspecified cell type, in remission
- C95.12 Chronic leukemia of unspecified cell type, in relapse
- C95.9 Leukemia, unspecified
- C95.91 Leukemia, unspecified, in remission
- C96.0 Multifocal and multisystemic (disseminated) Langerhans-cell histiocytosis
- C96.2 Malignant mast cell neoplasm
- C96.29 Other malignant mast cell neoplasm
- C96.4 Sarcoma of dendritic cells (accessory cells)
- C96.5 Multifocal and unisystemic Langerhans-cell histiocytosis
- C96.6 Unifocal Langerhans-cell histiocytosis

 $\mbox{C96.9}$  - Malignant neoplasm of lymphoid, hematopoietic and related tissue, unspecified

C96.A - Histiocytic sarcoma

C96.Z - Other specified malignant neoplasms of lymphoid, hematopoietic and related tissue

#### **Dialysis Codes**

#### Codes include:

#### - ICD9 prox codes:

39.95, Hemodialysis

54.98, Peritoneal dialysis

#### - ICD9 dx codes:

585.5x, Chronic kidney disease, Stage V (for ESRD with no mention of dialysis)

585.6x, End stage renal disease (for ESRD with dialysis)

V56.0x, encounter for dialysis NOS

V56.8x, encounter for peritoneal dialysis

V45.1x, renal dialysis status

#### - CPT4 codes:

90957, 90960, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 4 or more face-to-face physician visits per month

90958, 90961, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 2-3 face-to-face physician visits per

90959, 90962, ESRD related services monthly, for patients 12-19 and 20 years of age and older; with 1 face-to-face physician visit per month

90920, 90921, ESRD related services per full month; for patients 12-19 and twenty years of age and over

90924, 90925, ESRD related services (less than full month), per day; for patients 12-19 and twenty years of age and over

90935, Hemodialysis procedure with single physician evaluation

90937, Hemodialysis procedure requiring repeated evaluation(s) with or without substantial revision of dialysis prescription

90945, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies), with single physician evaluation

90947, Dialysis procedure other than hemodialysis (eg, peritoneal dialysis, hemofiltration, or other continuous renal replacement therapies) requiring repeated physician evaluations, with or without substantial revision of dialysis prescription

90965, 90966, ESRD related services for home dialysis per full month, for patients 12-19 and 20 years of age and older

90969, 90970, ESRD related services for dialysis less than a full month of service, per day; for patients 12-19 and 20 years of age and older

90989, Dialysis training, patient, including helper where applicable, any mode, completed course

90993, Dialysis training, patient, including helper where applicable, any mode, course not completed, per training session

90999, Unlisted dialysis procedure, inpatient or outpatient

99512, Home visit for hemodialysis

#### - HCPCS codes:

G0257, Unscheduled or emergency dialysis treatment for ESRD patient in a hospital outpatient dept. that is not certified as an ESRD facility

G0314, G0317, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age an over to include monitoring for the adequacy of nutrition, etc. w/4 or more physician visit per month

G0315, G0318, ESRD related services during the course of treatment, for patients 12-19 and 20yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/2 or 3 physician visit per month

G0316, G0319, ESRD related services during the course of treatment, for patients 12-19 and 20 yrs of age and over to include monitoring for the adequacy of nutrition, etc. w/1 physician visit per month

G0322, G0323, ESRD related services for home dialysis patients per full month: for patients 12-19 and 20 yrs of age and over to include monitoring for adequacy of nutrition and etc.

G0326, G0327, ESRD related services for home dialysis (less than full month), per day; for patients 12-19 and 20 yrs of age and over S9335, Home therapy, hemodialysis; administrative services, professional pharmacy services, care coordination, and all necessary supplies and equipment (drugs and nursing services coded separately), per diem

S9339, Home therapy, peritoneal dialysis, administrative services, care coordination and all necessary supplies and equipment, per diem

#### OR

Kidney transplant, defined as either 1 inpatient or 1 outpatient code

Codes include:

#### -ICD9 dx codes:

V42.0x, Kidney transplant status

996.81 Complications of transplanted kidney

#### -ICD9 prox codes:

55.6x, Transplant of kidney (Exclude 55.61)

#### - CPT4 codes:

50360, Renal allotransplantation, implantation, graft, w/o donor & recipient nephrectomy

50365, Renal allotransplantation, implantation, graft, w/ donor & recipient nephrectomy

#### Liver Bypass ICD-10 Procedure Codes 06100Z5 - Bypass Inferior Vena Cava to Superior Mesenteric Vein, Open Approach 0610496 - Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach 06104K5 - Bypass Inferior Vena Cava to Superior Mesenteric Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach 06104Z5 - Bypass Inferior Vena Cava to Superior Mesenteric Vein, Percutaneous Endoscopic Approach 06104ZY - Bypass Inferior Vena Cava to Lower Vein, Percutaneous Endoscopic Approach 061107B - Bypass Splenic Vein to Left Renal Vein with Autologous Tissue Substitute, Open Approach 0611099 - Bypass Splenic Vein to Right Renal Vein with Autologous Venous Tissue, Open Approach 06110AY - Bypass Splenic Vein to Lower Vein with Autologous Arterial Tissue, Open Approach 06110J9 - Bypass Splenic Vein to Right Renal Vein with Synthetic Substitute, Open Approach 0611479 - Bypass Splenic Vein to Right Renal Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach 061147Y - Bypass Splenic Vein to Lower Vein with Autologous Tissue Substitute. Percutaneous Endoscopic Approach 06114J9 - Bypass Splenic Vein to Right Renal Vein with Synthetic Substitute, Percutaneous Endoscopic Approach 06120ZY - Bypass Gastric Vein to Lower Vein, Open Approach 06140AY - Bypass Hepatic Vein to Lower Vein with Autologous Arterial Tissue, Open Approach 061507Y - Bypass Superior Mesenteric Vein to Lower Vein with Autologous Tissue Substitute, Open Approach 061509Y - Bypass Superior Mesenteric Vein to Lower Vein with Autologous Venous Tissue, Open Approach 061549Y - Bypass Superior Mesenteric Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach 06154AY - Bypass Superior Mesenteric Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach 061647Y - Bypass Inferior Mesenteric Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach 061709Y - Bypass Colic Vein to Lower Vein with Autologous Venous Tissue, Open Approach O61807Y - Bypass Portal Vein to Lower Vein with Autologous Tissue Substitute, Open Approach 061809B - Bypass Portal Vein to Left Renal Vein with Autologous Venous Tissue, Open Approach 061809Y - Bypass Portal Vein to Lower Vein with Autologous Venous Tissue, Open Approach 06180J9 - Bypass Portal Vein to Right Renal Vein with Synthetic Substitute, Open Approach 06180Z9 - Bypass Portal Vein to Right Renal Vein, Open Approach 0618479 - Bypass Portal Vein to Right Renal Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach 061849B - Bypass Portal Vein to Left Renal Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach 06184AB - Bypass Portal Vein to Left Renal Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach 06184JB - Bypass Portal Vein to Left Renal Vein with Synthetic Substitute, Percutaneous Endoscopic Approach 06184ZB - Bypass Portal Vein to Left Renal Vein, Percutaneous Endoscopic Approach 06190ZY - Bypass Right Renal Vein to Lower Vein, Open Approach 061947Y - Bypass Right Renal Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach 061949Y - Bypass Right Renal Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach 061B0ZY - Bypass Left Renal Vein to Lower Vein, Open Approach 061B4AY - Bypass Left Renal Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach 061B4KY - Bypass Left Renal Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach 061J09Y - Bypass Left Hypogastric Vein to Lower Vein with Autologous Venous Tissue, Open Approach 061J0KY - Bypass Left Hypogastric Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach 06L30ZZ - Occlusion of Esophageal Vein, Open Approach 061007Y - Bypass Inferior Vena Cava to Lower Vein with Autologous Tissue Substitute, Open Approach 06100A5 - Bypass Inferior Vena Cava to Superior Mesenteric Vein with Autologous Arterial Tissue, Open Approach 06100J5 - Bypass Inferior Vena Cava to Superior Mesenteric Vein with Synthetic Substitute, Open Approach 06100K6 - Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Nonautologous Tissue Substitute, Open Approach 06110JB - Bypass Splenic Vein to Left Renal Vein with Synthetic Substitute, Open Approach 06110KB - Bypass Splenic Vein to Left Renal Vein with Nonautologous Tissue Substitute, Open Approach 06114JY - Bypass Splenic Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach 061207Y - Bypass Gastric Vein to Lower Vein with Autologous Tissue Substitute, Open Approach 061407Y - Bypass Hepatic Vein to Lower Vein with Autologous Tissue Substitute, Open Approach 061409Y - Bypass Hepatic Vein to Lower Vein with Autologous Venous Tissue, Open Approach

061449Y - Bypass Hepatic Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach 06144AY - Bypass Hepatic Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach 06150KY - Bypass Superior Mesenteric Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach 06154ZY - Bypass Superior Mesenteric Vein to Lower Vein, Percutaneous Endoscopic Approach 061607Y - Bypass Inferior Mesenteric Vein to Lower Vein with Autologous Tissue Substitute, Open Approach 06160ZY - Bypass Inferior Mesenteric Vein to Lower Vein, Open Approach 06164AY - Bypass Inferior Mesenteric Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach 061749Y - Bypass Colic Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach 06174AY - Bypass Colic Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach 06174KY - Bypass Colic Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach 0618099 - Bypass Portal Vein to Right Renal Vein with Autologous Venous Tissue, Open Approach 06180K9 - Bypass Portal Vein to Right Renal Vein with Nonautologous Tissue Substitute. Open Approach 06184J9 - Bypass Portal Vein to Right Renal Vein with Synthetic Substitute, Percutaneous Endoscopic Approach O6184JY - Bypass Portal Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach 06184Z9 - Bypass Portal Vein to Right Renal Vein, Percutaneous Endoscopic Approach 061909Y - Bypass Right Renal Vein to Lower Vein with Autologous Venous Tissue, Open Approach 061J4JY - Bypass Left Hypogastric Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach O6L34CZ - Occlusion of Esophageal Vein with Extraluminal Device, Percutaneous Endoscopic Approach 0610075 - Bypass Inferior Vena Cava to Superior Mesenteric Vein with Autologous Tissue Substitute, Open Approach 06100A6 - Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Autologous Arterial Tissue, Open Approach 06100K5 - Bypass Inferior Vena Cava to Superior Mesenteric Vein with Nonautologous Tissue Substitute, Open Approach 06100KY - Bypass Inferior Vena Cava to Lower Vein with Nonautologous Tissue Substitute, Open Approach 06100ZY - Bypass Inferior Vena Cava to Lower Vein, Open Approach 061049Y - Bypass Inferior Vena Cava to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach 06104A5 - Bypass Inferior Vena Cava to Superior Mesenteric Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach 06104A6 - Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach 06104JY - Bypass Inferior Vena Cava to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach 06104Z6 - Bypass Inferior Vena Cava to Inferior Mesenteric Vein, Percutaneous Endoscopic Approach 061107Y - Bypass Splenic Vein to Lower Vein with Autologous Tissue Substitute, Open Approach 06110KY - Bypass Splenic Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach 06110ZB - Bypass Splenic Vein to Left Renal Vein, Open Approach 061149Y - Bypass Splenic Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach 06114A9 - Bypass Splenic Vein to Right Renal Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach 06114AB - Bypass Splenic Vein to Left Renal Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach 06114AY - Bypass Splenic Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach 06114ZB - Bypass Splenic Vein to Left Renal Vein, Percutaneous Endoscopic Approach 06140KY - Bypass Hepatic Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach 06140ZY - Bypass Hepatic Vein to Lower Vein, Open Approach 06144ZY - Bypass Hepatic Vein to Lower Vein, Percutaneous Endoscopic Approach 06150AY - Bypass Superior Mesenteric Vein to Lower Vein with Autologous Arterial Tissue. Open Approach 06150ZY - Bypass Superior Mesenteric Vein to Lower Vein, Open Approach 061609Y - Bypass Inferior Mesenteric Vein to Lower Vein with Autologous Venous Tissue, Open Approach 061649Y - Bypass Inferior Mesenteric Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach 06164JY - Bypass Inferior Mesenteric Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach 06164KY - Bypass Inferior Mesenteric Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach 06164ZY - Bypass Inferior Mesenteric Vein to Lower Vein, Percutaneous Endoscopic Approach 06170KY - Bypass Colic Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach 061807B - Bypass Portal Vein to Left Renal Vein with Autologous Tissue Substitute, Open Approach 06180JB - Bypass Portal Vein to Left Renal Vein with Synthetic Substitute, Open Approach 06180KY - Bypass Portal Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach

06180ZY - Bypass Portal Vein to Lower Vein, Open Approach 061847Y - Bypass Portal Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach 06184DY - Bypass Portal Vein to Lower Vein with Intraluminal Device, Percutaneous Endoscopic Approach 06184KY - Bypass Portal Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach 06190AY - Bypass Right Renal Vein to Lower Vein with Autologous Arterial Tissue, Open Approach 06194JY - Bypass Right Renal Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach 061B07Y - Bypass Left Renal Vein to Lower Vein with Autologous Tissue Substitute, Open Approach 061B0AY - Bypass Left Renal Vein to Lower Vein with Autologous Arterial Tissue, Open Approach 061B4ZY - Bypass Left Renal Vein to Lower Vein, Percutaneous Endoscopic Approach 061J07Y - Bypass Left Hypogastric Vein to Lower Vein with Autologous Tissue Substitute, Open Approach 061J4ZY - Bypass Left Hypogastric Vein to Lower Vein, Percutaneous Endoscopic Approach 06L33DZ - Occlusion of Esophageal Vein with Intraluminal Device, Percutaneous Approach O6L34DZ - Occlusion of Esophageal Vein with Intraluminal Device, Percutaneous Endoscopic Approach 0610096 - Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Autologous Venous Tissue, Open Approach 061009Y - Bypass Inferior Vena Caya to Lower Vein with Autologous Venous Tissue. Open Approach 06100Z6 - Bypass Inferior Vena Cava to Inferior Mesenteric Vein, Open Approach 0610476 - Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach 06104AY - Bypass Inferior Vena Cava to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach 06104J5 - Bypass Inferior Vena Cava to Superior Mesenteric Vein with Synthetic Substitute, Percutaneous Endoscopic Approach 06104J6 - Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Synthetic Substitute, Percutaneous Endoscopic Approach 06104KY - Bypass Inferior Vena Cava to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach 06110JY - Bypass Splenic Vein to Lower Vein with Synthetic Substitute, Open Approach 06110K9 - Bypass Splenic Vein to Right Renal Vein with Nonautologous Tissue Substitute, Open Approach 06110ZY - Bypass Splenic Vein to Lower Vein, Open Approach 0611499 - Bypass Splenic Vein to Right Renal Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach 06114JB - Bypass Splenic Vein to Left Renal Vein with Synthetic Substitute, Percutaneous Endoscopic Approach 06114K9 - Bypass Splenic Vein to Right Renal Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach 06114KB - Bypass Splenic Vein to Left Renal Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach 06114KY - Bypass Splenic Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach 06114Z9 - Bypass Splenic Vein to Right Renal Vein, Percutaneous Endoscopic Approach 06114ZY - Bypass Splenic Vein to Lower Vein, Percutaneous Endoscopic Approach 06120KY - Bypass Gastric Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach 061247Y - Bypass Gastric Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach 061249Y - Bypass Gastric Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach 06124AY - Bypass Gastric Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach 06150JY - Bypass Superior Mesenteric Vein to Lower Vein with Synthetic Substitute, Open Approach 06154JY - Bypass Superior Mesenteric Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach 06160KY - Bypass Inferior Mesenteric Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach 061747Y - Bypass Colic Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach 06174ZY - Bypass Colic Vein to Lower Vein, Percutaneous Endoscopic Approach 0618079 - Bypass Portal Vein to Right Renal Vein with Autologous Tissue Substitute, Open Approach 06180AY - Bypass Portal Vein to Lower Vein with Autologous Arterial Tissue, Open Approach 06180JY - Bypass Portal Vein to Lower Vein with Synthetic Substitute, Open Approach 06180KB - Bypass Portal Vein to Left Renal Vein with Nonautologous Tissue Substitute, Open Approach 06180ZB - Bypass Portal Vein to Left Renal Vein, Open Approach 06183DY - Bypass Portal Vein to Lower Vein with Intraluminal Device, Percutaneous Approach 061847B - Bypass Portal Vein to Left Renal Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach 0618499 - Bypass Portal Vein to Right Renal Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach 06184AY - Bypass Portal Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach 06184K9 - Bypass Portal Vein to Right Renal Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach

06184ZY - Bypass Portal Vein to Lower Vein, Percutaneous Endoscopic Approach 061907Y - Bypass Right Renal Vein to Lower Vein with Autologous Tissue Substitute, Open Approach 06194ZY - Bypass Right Renal Vein to Lower Vein, Percutaneous Endoscopic Approach 061B0JY - Bypass Left Renal Vein to Lower Vein with Synthetic Substitute, Open Approach 061B0KY - Bypass Left Renal Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach 061B47Y - Bypass Left Renal Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach 061B4JY - Bypass Left Renal Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach 061J0AY - Bypass Left Hypogastric Vein to Lower Vein with Autologous Arterial Tissue, Open Approach 061J0ZY - Bypass Left Hypogastric Vein to Lower Vein, Open Approach 061J47Y - Bypass Left Hypogastric Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach 06L30CZ - Occlusion of Esophageal Vein with Extraluminal Device, Open Approach 06L30DZ - Occlusion of Esophageal Vein with Intraluminal Device, Open Approach O6L33CZ - Occlusion of Esophageal Vein with Extraluminal Device, Percutaneous Approach 06L33ZZ - Occlusion of Esophageal Vein, Percutaneous Approach 0610076 - Bypass Inferior Vena Caya to Inferior Mesenteric Vein with Autologous Tissue Substitute. Open Approach 0610095 - Bypass Inferior Vena Cava to Superior Mesenteric Vein with Autologous Venous Tissue, Open Approach 06100AY - Bypass Inferior Vena Cava to Lower Vein with Autologous Arterial Tissue, Open Approach 06100J6 - Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Synthetic Substitute, Open Approach 06100JY - Bypass Inferior Vena Cava to Lower Vein with Synthetic Substitute, Open Approach 0610475 - Bypass Inferior Vena Cava to Superior Mesenteric Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach 061047Y - Bypass Inferior Vena Cava to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach 0610495 - Bypass Inferior Vena Cava to Superior Mesenteric Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach 06104K6 - Bypass Inferior Vena Cava to Inferior Mesenteric Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach 0611079 - Bypass Splenic Vein to Right Renal Vein with Autologous Tissue Substitute, Open Approach 061109B - Bypass Splenic Vein to Left Renal Vein with Autologous Venous Tissue, Open Approach 061109Y - Bypass Splenic Vein to Lower Vein with Autologous Venous Tissue, Open Approach 06110A9 - Bypass Splenic Vein to Right Renal Vein with Autologous Arterial Tissue, Open Approach 06110AB - Bypass Splenic Vein to Left Renal Vein with Autologous Arterial Tissue, Open Approach 06110Z9 - Bypass Splenic Vein to Right Renal Vein, Open Approach 061147B - Bypass Splenic Vein to Left Renal Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach 061149B - Bypass Splenic Vein to Left Renal Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach 061209Y - Bypass Gastric Vein to Lower Vein with Autologous Venous Tissue, Open Approach 06120AY - Bypass Gastric Vein to Lower Vein with Autologous Arterial Tissue, Open Approach 06120JY - Bypass Gastric Vein to Lower Vein with Synthetic Substitute, Open Approach 06124JY - Bypass Gastric Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach 06124KY - Bypass Gastric Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach 06124ZY - Bypass Gastric Vein to Lower Vein, Percutaneous Endoscopic Approach 06140JY - Bypass Hepatic Vein to Lower Vein with Synthetic Substitute, Open Approach 061447Y - Bypass Hepatic Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach 06144JY - Bypass Hepatic Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach 06144KY - Bypass Hepatic Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach 061547Y - Bypass Superior Mesenteric Vein to Lower Vein with Autologous Tissue Substitute, Percutaneous Endoscopic Approach 06154KY - Bypass Superior Mesenteric Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach 06160AY - Bypass Inferior Mesenteric Vein to Lower Vein with Autologous Arterial Tissue, Open Approach 06160JY - Bypass Inferior Mesenteric Vein to Lower Vein with Synthetic Substitute, Open Approach 061707Y - Bypass Colic Vein to Lower Vein with Autologous Tissue Substitute, Open Approach 06170AY - Bypass Colic Vein to Lower Vein with Autologous Arterial Tissue, Open Approach 06170JY - Bypass Colic Vein to Lower Vein with Synthetic Substitute, Open Approach 06170ZY - Bypass Colic Vein to Lower Vein, Open Approach 06174JY - Bypass Colic Vein to Lower Vein with Synthetic Substitute, Percutaneous Endoscopic Approach

| 06180A9 · | <ul> <li>Bypass</li> </ul> | Porta | l Vein | to | Right | Renal | Vein | with | Autol | ogous | Arteria | al Tissue | , Open | Approa | acl |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | _ | | | | | | | | | | | | _ | | |

06180AB - Bypass Portal Vein to Left Renal Vein with Autologous Arterial Tissue, Open Approach

061849Y - Bypass Portal Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach

06184A9 - Bypass Portal Vein to Right Renal Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach

06184KB - Bypass Portal Vein to Left Renal Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach

06190JY - Bypass Right Renal Vein to Lower Vein with Synthetic Substitute, Open Approach

06190KY - Bypass Right Renal Vein to Lower Vein with Nonautologous Tissue Substitute, Open Approach

06194AY - Bypass Right Renal Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach

06194KY - Bypass Right Renal Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach

061B09Y - Bypass Left Renal Vein to Lower Vein with Autologous Venous Tissue, Open Approach

061B49Y - Bypass Left Renal Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach

061J0JY - Bypass Left Hypogastric Vein to Lower Vein with Synthetic Substitute, Open Approach

061J49Y - Bypass Left Hypogastric Vein to Lower Vein with Autologous Venous Tissue, Percutaneous Endoscopic Approach

061J4AY - Bypass Left Hypogastric Vein to Lower Vein with Autologous Arterial Tissue, Percutaneous Endoscopic Approach

061J4KY - Bypass Left Hypogastric Vein to Lower Vein with Nonautologous Tissue Substitute, Percutaneous Endoscopic Approach

06L34ZZ - Occlusion of Esophageal Vein, Percutaneous Endoscopic Approach

| <b>Procedure Codes</b> | Description |
|---|---|
| CPT-4 codes | |
| | Anesthesia for vaginal delivery only |
| | Anesthesia for cesarean delivery only |
| | Anesthesia for urgent hysterectomy following delivery |
| 1963 | Anesthesia for cesarean hysterectomy w/o any labor analgesia/anesthesia care |
| 1967 | Neuraxial labor analgesia/anesthesia, planned vaginal delivery |
| 1968 | Anesthesia for cesarean delivery following neuraxial labor analgesia/anesthesia |
| 1969 | Anes for cesarean hysterectomy following neuraxial labor analgesia/anesthesia |
| 59050 | Fetal monitoring in labor, physician w/written report; s & i |
| 59051 | Fetal monitoring in labor, physician w/written report; intrepretation only |
| 59400 | ROUTINE TOTAL OBSTETRIC CARE including antepartum care, vaginal delivery (with or without episiotomy, and/or forceps) and postpartum care. |
| 59409 | Vaginal delivery only (w/wo episiotomy &/or forceps) |
| 59410 | Vaginal delivery only (w/wo episiotomy &/or forceps); w/postpartum care |
| 59412 | Ext cephalic version, w/wo tocolysis |
| 59414 | Delivery of placenta (separate proc) |
| | Postpartum care only |
| 59510 | Routine obstetric care w/antepartum care, cesarean delivery, & postpartum care |
| 59514 | Cesarean delivery only |
| 59515 | Cesarean delivery only; w/postpartum care |
| 59525 | Subtotal/total hysterectomy after cesarean delivery |
| | Routine obstetric care including antepartum care, vaginal delivery (with or without episiotomy, and/or forceps) and postpartum care, after previous cesarean delivery |
| | Vaginal delivery only, after previous cesarean delivery (with or without episiotomy and/or forceps) |
| | Vaginal delivery only, previous cesarean delivery w/postpartum care |
| | Routine obstetric care including antepartum care, cesarean delivery, and postpartum care, following attempted vaginal delivery after previous cesarean delivery |
| | Cesarean delivery after failed vaginal delivery, previous cesarean delivery |
| | Cesarean delivery after failed vaginal delivery, previous cesarean delivery; w/postpartum care |
| | Attendance at delivery, at request of delivering physician, & stabilization of newborn |
| 99440 | Newborn resuscitation |
| ICD O | |
| ICD-9 procedure | |
| codes<br>72.xx | Forceps, vacuum, & breech |
| | Other including manual delivery |
| | Cesarean section |
| | Manual removal of placenta |
| 75.4X<br>ICD-10 | Manual Territoral of pracerita |
| procedure | |
| codes | |
| Normal | |
| Delivery | |
| | Delivery of Products of Conception, External Approach |
| C-Section | Sellery of Houseas of Conception, Exertian Approach |
| | Extraction of Products of Conception, High, Open Approach |
| | Extraction of Products of Conception, Low, Open Approach |
| | Extraction of Products of Conception, Extraperitoneal, Open Approach |
| | elivery (forceps, vacuum, internal version, other) |
| | Extraction of Products of Conception, Low Forceps, Via Natural or Artificial Opening |
| | Extraction of Products of Conception, Mid Forceps, Via Natural or Artificial Opening |
| | Extraction of Products of Conception, High Forceps, Via Natural or Artificial Opening |
| | Extraction of Products of Conception, Vacuum, Via Natural or Artificial Opening |
| | Extraction of Products of Conception, Internal Version, Via Natural or Artificial Opening |
| | Extraction of Products of Conception, Other, Via Natural or Artificial Opening |
| ICD-9 code | Definition Gestational Age |


# Dx codes:

009.XYZ Supervision of high risk pregnancy (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)

O10 Pre-existing hypertension complicating pregnancy, childbirth and the puerperium (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)

- O11 Pre-existing hypertension with pre-eclampsia (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O12 Gestational [pregnancy-induced] edema and proteinuria without hypertension (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O13 Gestational [pregnancy-induced] hypertension without significant proteinuria (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)

- O14 Pre-eclampsia (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O15 Eclampsia (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O16 Unspecified maternal hypertension (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O20 Hemorrhage in early pregnancy
- O21 Excessive vomiting in pregnancy (last digit refers to first/second/third/unspecified trimester)
- O22 Venous complications and hemorrhoids in pregnancy
- O23 Infections of genitourinary tract in pregnancy (last digit refers to first/second/third/unspecified trimester)
- O24 Diabetes mellitus in pregnancy, childbirth, and the puerperium (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O25 Malnutrition in pregnancy, childbirth and the puerperium (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O26 Maternal care for other conditions predominantly related to pregnancy (if last digit indicating first/second/third/unspecified trimester/unspecified as to time period)
- O28 Abnormal findings on antenatal screening of mother
- O29 Complications of anesthesia during pregnancy (last digit refers to first/second/third/unspecified trimester)
- O30 Multiple gestation (last digit refers to first/second/third/unspecified trimester)
- O31 Complications specific to multiple gestation (certain digit refers to first/second/third/unspecified trimester)
- O32 Maternal care for malpresentation of fetus
- O33 Maternal care for disproportion
- O34 Maternal care for abnormality of pelvic organs (most codes indicate first/second/third/unspecified trimester)
- O35 Maternal care for known or suspected fetal abnormality and damage
- O36 Maternal care for other fetal problems (codes indicate first/second/third/unspecified trimester)
- O40 Polyhydramnios (codes indicate first/second/third/unspecified trimester)
- O41 Other disorders of amniotic fluid and membranes (codes indicate first/second/third/unspecified trimester)
- O42.1 Premature rupture of membranes, onset of labor more than 24 hours following rupture
- O42.9 Premature rupture of membranes, unspecified as to length of time between rupture and onset of labor
- O43 Placental disorders (last digit refers to first/second/third/unspecified trimester)
- O44 Placenta previa (last digit refers to first/second/third/unspecified trimester)
- O45 Premature separation of placenta (last digit refers to first/second/third/unspecified trimester)
- O46 Antepartum hemorrhage, not elsewhere classified (last digit refers to first/second/third/unspecified trimester)
- O47 False labor
- O60.0 Preterm labor without delivery
- O61 Failed induction of labor
- O71.0 Rupture of uterus (spontaneous) before onset of labor
- O72 Postpartum hemorrhage
- O72.2 Delayed and secondary postpartum hemorrhage
- O72.3 Postpartum coagulation defects
- 073 Retained placenta and membranes, without hemorrhage
- O75 Other complications of labor and delivery, not elsewhere classified
- O94 Sequelae of complication of pregnancy, childbirth, and the puerperium
- O98 Maternal infectious and parasitic diseases classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates first trimester, second trimester, third trimester, unspecified, or nothing)
- O99 Other maternal diseases classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates first trimester, second trimester, third trimester, unspecified, or nothing)
- O9A Maternal malignant neoplasms, traumatic injuries and abuse classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates first trimester, second trimester, third trimester, unspecified, or nothing)
- Z32.01 Encounter for pregnancy test result positive
- Z33 Pregnant state
- Z34 Encounter for supervision of normal pregnancy
- Z36 Encounter for antenatal screening of mother
- Z39 Encounter for maternal postpartum care and examination
- Z39.1 Encounter for care and examination of lactating mother
- Z39.2 Encounter for routine postpartum follow-up
- Z3A Weeks of gestation

#### Proc codes:

- 102 Change
- 109 Drainage
- 10H Insertion
- 10J Inspection
- 10P Removal
- 10Q Repair

#### 10S Reposition

10Y Transplantation

ICD-10 CODES INDICATING DELIVERY (diagnostic codes that were not considered in the algorithm to identify deliveries)

#### Dx codes:

Use the following codes only if the last digit indicates childbirth or puerperium or labor

- O10 Pre-existing hypertension complicating pregnancy, childbirth and the puerperium
- O11 Pre-existing hypertension with pre-eclampsia
- O12 Gestational [pregnancy-induced] edema and proteinuria without hypertension
- O13 Gestational [pregnancy-induced] hypertension without significant proteinuria
- O14 Pre-eclampsia
- O15 Eclampsia
- O16 Unspecified maternal hypertension
- O24 Diabetes mellitus in pregnancy, childbirth, and the puerperium
- O25 Malnutrition in pregnancy, childbirth and the puerperium
- O26 Maternal care for other conditions predominantly related to pregnancy
- O42.0 Premature rupture of membranes, onset of labor within 24 hours of rupture, except 042.011 (first trimester)
- O48 Late pregnancy
- O60.1 Preterm labor with preterm delivery
- O60.2 Term delivery with preterm labor
- O62 Abnormalities of forces of labor
- O63 Long labor
- O64 Obstructed labor due to malposition and malpresentation of fetus
- O65 Obstructed labor due to maternal pelvic abnormality
- O66 Other obstructed labor
- O67 Labor and delivery complicated by intrapartum hemorrhage, not elsewhere classified
- O68 Labor and delivery complicated by abnormality of fetal acid-base balance
- O69 Labor and delivery complicated by umbilical cord complications
- O70 Perineal laceration during delivery
- O71.1 Rupture of uterus during labor
- O71.2 Postpartum inversion of uterus
- O71.3 Obstetric laceration of cervix
- O71.4 Obstetric high vaginal laceration alone
- O72.0 Third-stage hemorrhage
- O72.1 Other immediate postpartum hemorrhage
- O74 Complications of anesthesia during labor and delivery
- O76 Abnormality in fetal heart rate and rhythm complicating labor and delivery
- O77 Other fetal stress complicating labor and delivery
- O80 Encounter for full-term uncomplicated delivery
- O82 Encounter for cesarean delivery without indication
- O98 Maternal infectious and parasitic diseases classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates childbirth or puerperium)
- O99 Other maternal diseases classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates childbirth or puerperium)
- O9A Maternal malignant neoplasms, traumatic injuries and abuse classifiable elsewhere but complicating pregnancy, childbirth and the puerperium (if last digit indicates childbirth or puerperium)
- Z37 Outcome of delivery (For livebirth cohort, exclude Z37.1, Z37.4, Z37.7 all stillbirth codes)
- Z38 Liveborn infants according to place of birth and type of delivery
- Z39.0 Encounter for care and examination of mother immediately after delivery

#### ICD-10 CODES INDICATING PREGNANCY WITH ABORTIVE/NON-LIVE BIRTH OUTCOMES

#### Dx codes:

O00-O08 Pregnancy with abortive outcome

#### Proc codes:

- 10A Abortion
- 10D17Z9 Manual Extraction of Products of Conception, Retained, Via Natural or Artificial Opening
- 10D17ZZ Extraction of Products of Conception, Retained, Via Natural or Artificial Opening
- 10D18Z9 Manual Extraction of Products of Conception, Retained, Via Natural or Artificial Opening Endoscopic
- 10D18ZZ Extraction of Products of Conception, Retained, Via Natural or Artificial Opening Endoscopic

#### ICD-10 CODES INDICATING ECTOPIC PREGNANCY

10D27ZZ Extraction of Products of Conception, Ectopic, Via Natural or Artificial Opening

10D28ZZ Extraction of Products of Conception, Ectopic, Via Natural or Artificial Opening Endoscopic

10S2 Reposition Products of Conception, Ectopic

10T Resection (Ectopic)

| | | | | Unma | atched | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Optum | | | MarketScan | | | Medicare | | | Pooled | |
| Variable | Rivaroxaban | Apixaban | St. Diff | Rivaroxaban | Apixaban | St. Diff | Rivaroxaban | Apixaban | St. Diff | Rivaroxaban | Apixaban | St. Diff |
| Number of patients | 4,49 | 9 5,08 | 37 | 6,33 | 9 4,78 | 1 | 12,78 | 5 8,32 | 9 | 23,624 | 18,197 | |
| Age<br>mean (sd) | 61.83 (16.97) | 69.01 (15.57) | -0.44 | 53.93 (15.65) | 57.11 (15.97) | -0.20 | 70.91 (13.02) | 74.18 (12.37) | -0.26 | 64.62 (14.57) | 68.25 (14.31) | -0.25 |
| mean (sɑ)<br>median (IQR) | 64.00 [51.00, 75.00] | | -0.49 | | 57.11 (15.97)<br>0] 57.00 [47.00, 66.00] | | | 74.18 (12.37)<br>0] 75.00 [68.00, 83.0 | | 65.91 (14.57) | 69.43 (14.31) | -0.25<br>-0.24 |
| Age categories | 64.00 [51.00, 75.00] | 72.00 [61.00, 81.00] | -0.49 | 55.00 [44.00, 63.0 | 0] 57.00 [47.00, 66.00] | -0.13 | 72.00 [66.00, 80.00 | ıj 75.00 [68.00, 83.0 | 00-0.24 | 05.91 (14.57) | 09.43 (14.31) | -0.24 |
| 18 - 54: n (%) | 1.386 (30.8%) | 883 (17.4%) | 0.32 | 3.104 (49.0%) | 1.981 (41.4%) | 0.15 | 1.412 (11.0%) | 592 (7.1%) | 0.14 | 5,902 (25.0%) | 3.456 (19.0%) | 0.15 |
| 55 - 64: n (%) | 865 (19.2%) | 676 (13.3%) | 0.16 | 1,888 (29.8%) | 1,536 (32.1%) | -0.05 | 1,202 (9.4%) | 619 (7.4%) | 0.07 | 3,955 (16.7%) | 2,831 (15.6%) | 0.03 |
| 65 - 74: n (%) | 1,095 (24.3%) | 1,341 (26.4%) | -0.05 | 723 (11.4%) | 552 (11.5%) | 0.00 | 4,839 (37.8%) | 2,798 (33.6%) | 0.09 | 6,657 (28.2%) | 4,691 (25.8%) | 0.05 |
| >= 75; n (%) | 1,153 (25.6%) | 2,187 (43.0%) | -0.37 | 624 (9.8%) | 712 (14.9%) | -0.16 | 5,333 (41.7%) | 4,320 (51.9%) | -0.21 | 7,110 (30.1%) | 7,219 (39.7%) | -0.20 |
| Calendar Year (2014-2020) | | | | | | | | | | | | |
| 2014; n (%) | 295 (6.6%) | 23 (0.5%) | 0.33 | 837 (13.2%) | 69 (1.4%) | 0.47 | 1,392 (10.9%) | 175 (2.1%) | 0.36 | 2,524 (10.7%) | 267 (1.5%) | 0.39 |
| 2015; n (%) | 761 (16.9%) | 193 (3.8%) | 0.44 | 1,592 (25.1%) | 465 (9.7%) | 0.41 | 3,619 (28.3%) | 1,581 (19.0%) | 0.22 | 5,972 (25.3%) | 2,239 (12.3%) | 0.34 |
| 2016; n (%) | 834 (18.5%) | 513 (10.1%) | 0.24 | 1,424 (22.5%) | 893 (18.7%) | 0.09 | 3,778 (29.5%) | 3,246 (39.0%) | -0.20 | 6,036 (25.6%) | 4,652 (25.6%) | 0.00 |
| .2017; n (%) | 793 (17.6%) | 774 (15.2%) | 0.06 | 1,032 (16.3%) | 1,069 (22.4%) | -0.15 | 3,997 (31.3%) | 3,327 (39.9%) | -0.18 | 5,822 (24.6%) | 5,170 (28.4%) | -0.09 |
| 2018; n (%) | 869 (19.3%) | 1,276 (25.1%) | -0.14 | 823 (13.0%) | 1,079 (22.6%) | -0.25 | 0 (0.0%) | 0 (0.0%) | 0.00 | 1,692 (7.2%) | 2,355 (12.9%) | -0.19 |
| .2019; n (%) | 727 (16.2%) | 1,514 (29.8%) | -0.33 | 631 (10.0%) | 1,206 (25.2%) | -0.41 | 0 (0.0%) | 0 (0.0%) | 0.00 | 1,358 (5.7%) | 2,720 (14.9%) | -0.31 |
| .2020; n (%) | 220 (4.9%) | 794 (15.6%) | -0.36 | 0 (0.0%) | 0 (0.0%) | 0.00 | 0 (0.0%) | 0 (0.0%) | 0.00 | 220 (0.9%) | 794 (4.4%) | -0.22 |
| ace | | | | | | | | | | | | |
| .White; n (%) | 3,257 (72.4%) | 3,455 (67.9%) | 0.10 | 0 (0.0%) | 0 (0.0%) | 0.00 | 10,471 (81.9%) | 6,881 (82.6%) | -0.02 | 13,728 (58.1%) | 10,336 (56.8%) | 0.03 |
| Asian; n (%) | 79 (1.8%) | 73 (1.4%) | 0.03 | 0 (0.0%) | 0 (0.0%) | 0.00 | 100 (0.8%) | 76 (0.9%) | -0.01 | 179 (0.8%) | 149 (0.8%) | 0.00 |
| .Black; n (%) | 635 (14.1%) | 822 (16.2%) | -0.06 | 0 (0.0%) | 0 (0.0%) | 0.00 | 1,661 (13.0%) | 1,086 (13.0%) | 0.00 | 2,296 (9.7%) | 1,908 (10.5%) | -0.03 |
| Hispanic; n (%) | 336 (7.5%) | 453 (8.9%) | -0.05 | 0 (0.0%) | 0 (0.0%) | 0.00 | 234 (1.8%) | 123 (1.5%) | 0.02 | 570 (2.4%) | 576 (3.2%) | -0.05 |
| North American Native; n (%) | 0 (0.0%) | 0 (0.0%) | 0.00 | 0 (0.0%) | 0 (0.0%) | 0.00 | 68 (0.5%) | 22 (0.3%) | 0.03 | 68 (0.3%) | 22 (0.1%) | 0.04 |
| .Other; n (%) | 0 (0.0%) | 0 (0.0%) | 0.00 | 0 (0.0%) | 0 (0.0%) | 0.00 | 101 (0.8%) | 63 (0.8%) | 0.00 | 101 (0.4%) | 63 (0.3%) | 0.02 |
| .Unknown/Missing; n (%) | 192 (4.3%) | 284 (5.6%) | -0.06 | 0 (0.0%) | 0 (0.0%) | 0.00 | 151 (1.2%) | 78 (0.9%) | 0.03 | 343 (1.5%) | 362 (2.0%) | -0.04 |
| ender | | | | | | | | | | | | |
| .Males; n (%) | 2,247 (49.9%) | 2,172 (42.7%) | 0.14 | 3,418 (53.9%) | 2,483 (51.9%) | 0.04 | 5,549 (43.4%) | 3,206 (38.5%) | 0.10 | 11,214 (47.5%) | 7,861 (43.2%) | 0.09 |
| .Females; n (%) | 2,252 (50.1%) | 2,915 (57.3%) | -0.14 | 2,921 (46.1%) | 2,298 (48.1%) | -0.04 | 7,237 (56.6%) | 5,123 (61.5%) | -0.10 | 12,410 (52.5%) | 10,336 (56.8%) | -0.09 |
| egion | | | | | | | | | | | | |
| .Northeast; n (%) | 528 (11.7%) | 544 (10.7%) | 0.03 | 1,311 (20.7%) | 962 (20.1%) | 0.01 | 2,384 (18.6%) | 1,613 (19.4%) | -0.02 | 4,223 (17.9%) | 3,119 (17.1%) | 0.02 |
| South; n (%) | 1,870 (41.6%) | 2,524 (49.6%) | -0.16 | 2,549 (40.2%) | 2,236 (46.8%) | -0.13 | 5,001 (39.1%) | 3,826 (45.9%) | -0.14 | 9,420 (39.9%) | 8,586 (47.2%) | -0.15 |
| .Midwest; n (%) | 1,082 (24.0%) | 996 (19.6%) | 0.11 | 1,625 (25.6%) | 1,028 (21.5%) | 0.10 | 3,191 (25.0%) | 1,720 (20.7%) | 0.10 | 5,898 (25.0%) | 3,744 (20.6%) | 0.11 |
| .West; n (%) | 1,004 (22.3%) | 1,016 (20.0%) | 0.06 | 825 (13.0%) | 544 (11.4%) | 0.05 | 2,200 (17.2%) | 1,162 (14.0%) | 0.09 | 4,029 (17.1%) | 2,722 (15.0%) | 0.06 |
| .Unknown+missing; n (%) | 15 (0.3%) | 7 (0.1%) | 0.04 | 29 (0.5%) | 11 (0.2%) | 0.05 | | | | | | |
| Combined comorbidity score, 180 days Copy | | | | | | | | | | | | |
| .mean (sd) | 2.62 (2.34) | 3.65 (2.64) | -0.41 | 1.61 (1.72) | 2.19 (1.89) | -0.32 | 2.17 (2.08) | 2.74 (2.27) | -0.26 | 2.11 (2.04) | 2.85 (2.29) | -0.34 |
| .median [IQR] | 2.00 [1.00, 4.00] | 3.00 [2.00, 5.00] | -0.40 | 1.00 [0.00, 3.00] | 2.00 [1.00, 3.00] | 0.00 | 2.00 [1.00, 3.00] | 2.00 [1.00, 4.00] | 0.00 | 1.73 (2.04) | 2.28 (2.29) | -0.25 |
| ifestyle Factors | | | | | | | | | | | | |
| ifestyle - Smoking ; n (%) | 1,587 (35.3%) | 1,929 (37.9%) | -0.05 | 1,226 (19.3%) | 925 (19.3%) | 0.00 | 5,433 (42.5%) | 3,322 (39.9%) | 0.05 | 8,246 (34.9%) | 6,176 (33.9%) | 0.02 |
| festyle - Drug abuse or dependence; n (%) | 220 (4.9%) | 274 (5.4%) | -0.02 | 180 (2.8%) | 135 (2.8%) | 0.00 | 605 (4.7%) | 300 (3.6%) | 0.06 | 1,005 (4.3%) | 709 (3.9%) | 0.02 |
| festyle - Alcohol abuse or dependence ; n (%) | 190 (4.2%) | 193 (3.8%) | 0.02 | 166 (2.6%) | 127 (2.7%) | -0.01 | 465 (3.6%) | 241 (2.9%) | 0.04 | 821 (3.5%) | 561 (3.1%) | 0.02 |
| omorbidities | 40 (0 00) | 00 (4 500) | 0.05 | 22 (2 52() | 22 (2 70) | 0.00 | 440 (0.000) | 00 (4 400) | 0.00 | 407 (0.00) | 204 (4 400) | 0.00 |
| M - Diabetic Retinopathy; n (%) | 42 (0.9%) | 83 (1.6%) | -0.06 | 33 (0.5%) | 32 (0.7%) | -0.03 | 112 (0.9%) | 89 (1.1%) | -0.02 | 187 (0.8%) | 204 (1.1%) | -0.03 |
| M - Diabetic Neuropathy; n (%) | 211 (4.7%) | 361 (7.1%) | -0.10 | 156 (2.5%) | 163 (3.4%) | -0.05 | 589 (4.6%) | 440 (5.3%) | -0.03 | 956 (4.0%) | 964 (5.3%) | -0.06 |
| M - Diabetic Nephropathy; n (%) | 144 (3.2%) | 381 (7.5%) | -0.19 | 80 (1.3%) | 105 (2.2%) | -0.07 | 299 (2.3%) | 364 (4.4%) | -0.12 | 523 (2.2%) | 850 (4.7%) | -0.14 |
| M - Diabetes with peripheral circulatory disorders; n (%) | 9 (0.2%) | 11 (0.2%) | 0.00 | 20 (0.3%) | 7 (0.1%) | 0.04 | 64 (0.5%) | 27 (0.3%) | 0.03 | 93 (0.4%) | 45 (0.2%) | 0.04 |
| M - Diabetes with peripheral circulatory disorders and lower extremity amputation; n (%) | 46 (1.0%) | 61 (1.2%) | -0.02 | 34 (0.5%) | 20 (0.4%) | 0.01 | 199 (1.6%) | 107 (1.3%) | 0.03 | 279 (1.2%) | 188 (1.0%) | 0.02 |
| M - Diabetes with unspecified complications; n (%) | 58 (1.3%) | 146 (2.9%) | -0.11 | 879 (13.9%) | 768 (16.1%) | -0.06 | 174 (1.4%) | 124 (1.5%) | -0.01 | 1,111 (4.7%) | 1,038 (5.7%) | -0.05 |
| M - Diabetes mellitus without mention of complications; n (%) | 780 (17.3%) | 1,249 (24.6%) | -0.18 | 68 (1.1%) | 75 (1.6%) | -0.04 | 2,920 (22.8%) | 1,979 (23.8%) | -0.02 | 3,768 (15.9%) | 3,303 (18.2%) | -0.06 |
| V - Hypertension; n (%) | 2,622 (58.3%) | 3,588 (70.5%) | -0.26 | 2,922 (46.1%) | 2,632 (55.1%) | -0.18 | 9,714 (76.0%) | 6,715 (80.6%) | -0.11 | 15,258 (64.6%) | 12,935 (71.1%) | -0.14 |
| V - Hyperlipidemia; n (%) | 1,932 (42.9%) | 2,645 (52.0%) | -0.18 | 2,051 (32.4%) | 1,737 (36.3%) | -0.08 | 6,823 (53.4%) | 4,603 (55.3%) | -0.04 | 10,806 (45.7%) | 8,985 (49.4%) | -0.07 |
| V -Acute MI; n (%) | 207 (4.6%) | 313 (6.2%) | -0.07 | 226 (3.6%) | 215 (4.5%) | -0.05 | 507 (4.0%) | 466 (5.6%) | -0.07 | 940 (4.0%) | 994 (5.5%) | -0.07 |
| V - ACS/unstable angina; n (%) | 130 (2.9%) | 232 (4.6%) | -0.09<br>-0.08 | 147 (2.3%) | 151 (3.2%) | -0.06<br>-0.02 | 442 (3.5%) | 308 (3.7%) | -0.01 | 719 (3.0%) | 691 (3.8%) | -0.04<br>-0.04 |
| V - Old MI; n (%) | 158 (3.5%) | 258 (5.1%)<br>165 (3.2%) | -0.08<br>-0.07 | 104 (1.6%)<br>107 (1.7%) | 92 (1.9%) | | 602 (4.7%)<br>277 (2.2%) | 454 (5.5%) | -0.04<br>-0.04 | 864 (3.7%)<br>480 (2.0%) | 804 (4.4%)<br>514 (2.8%) | |
| V - Stable angina; n (%) | 96 (2.1%) | | | | 109 (2.3%) | -0.04 | , , | 240 (2.9%) | | | | -0.05 |
| V - Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) | 603 (13.4%) | 976 (19.2%) | -0.16<br>-0.02 | 539 (8.5%) | 482 (10.1%) | -0.06<br>0.00 | 2,387 (18.7%) | 1,832 (22.0%) | -0.08<br>0.01 | 3,529 (14.9%) | 3,290 (18.1%) | -0.09<br>0.00 |
| V - Other atherosclerosis; n (%) | 41 (0.9%) | 58 (1.1%)<br>304 (6.0%) | -0.02<br>-0.09 | 26 (0.4%)<br>99 (1.6%) | 21 (0.4%)<br>64 (1.3%) | 0.00 | 128 (1.0%)<br>888 (6.9%) | 74 (0.9%)<br>663 (8.0%) | 0.01<br>-0.04 | 195 (0.8%)<br>1,171 (5.0%) | 153 (0.8%)<br>1.031 (5.7%) | -0.03 |
| | | | -0.09<br>-0.14 | 99 (1.6%)<br>230 (3.6%) | 64 (1.3%)<br>227 (4.7%) | -0.06 | 888 (6.9%)<br>830 (6.5%) | 663 (8.0%)<br>685 (8.2%) | -0.04<br>-0.07 | 1,171 (5.0%)<br>1,299 (5.5%) | 1,031 (5.7%) | -0.03<br>-0.08 |
| V - Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) | 184 (4.1%) | AAC (0.00/\ | -0.14 | 23U (3.b%) | ZZ/ (4./%) | | , | 685 (8.2%)<br>16 (0.2%) | -0.07<br>0.00 | 1,299 (5.5%)<br>34 (0.1%) | 1,358 (7.5%) | -0.08 |
| / - Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%)<br>/ - Ischemic stroke; n (%) | 239 (5.3%) | 446 (8.8%) | 0.04 | E (O 19/) | 2 (0.09/) | | | | | 34 (U.1%) | 38 (U.2%) | -0.03 |
| / - Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) / - Ischemic stroke; n (%) / - Hemorrhagic stroke; n (%) | 239 (5.3%)<br>8 (0.2%) | 20 (0.4%) | -0.04 | 5 (0.1%) | 2 (0.0%) | 0.04 | 21 (0.2%) | | | 357 /1 50/\ | 271 /2 09/1 | -0.04 |
| / - Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) /- Ischemic stroke; n (%) /- Hemorrhagic stroke; n (%) /- TIA; n (%) | 239 (5.3%)<br>8 (0.2%)<br>72 (1.6%) | 20 (0.4%)<br>118 (2.3%) | -0.05 | 69 (1.1%) | 77 (1.6%) | -0.04 | 216 (1.7%) | 176 (2.1%) | -0.03 | 357 (1.5%) | 371 (2.0%) | -0.04 |
| /- Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) /- Ischemic stroke; n (%) /- Hemorrhagic stroke; n (%) /- TIA; n (%) /- Other cerebrovascular disease; n (%) | 239 (5.3%)<br>8 (0.2%)<br>72 (1.6%)<br>122 (2.7%) | 20 (0.4%)<br>118 (2.3%)<br>246 (4.8%) | -0.05<br>-0.11 | 69 (1.1%)<br>93 (1.5%) | 77 (1.6%)<br>124 (2.6%) | -0.04<br>-0.08 | 216 (1.7%)<br>365 (2.9%) | 176 (2.1%)<br>302 (3.6%) | -0.03<br>-0.04 | 580 (2.5%) | 672 (3.7%) | -0.07 |
| /- Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) - Ischemic stroke; n (%) - Hemorrhagic stroke; n (%) - TIA; n (%) / - Other cerebrovascular disease; n (%) - Late effects of cerebrovascular disease; n (%) | 239 (5.3%)<br>8 (0.2%)<br>72 (1.6%)<br>122 (2.7%)<br>94 (2.1%) | 20 (0.4%)<br>118 (2.3%)<br>246 (4.8%)<br>203 (4.0%) | -0.05<br>-0.11<br>-0.11 | 69 (1.1%)<br>93 (1.5%)<br>67 (1.1%) | 77 (1.6%)<br>124 (2.6%)<br>59 (1.2%) | -0.04<br>-0.08<br>-0.01 | 216 (1.7%)<br>365 (2.9%)<br>375 (2.9%) | 176 (2.1%)<br>302 (3.6%)<br>273 (3.3%) | -0.03<br>-0.04<br>-0.02 | 580 (2.5%)<br>536 (2.3%) | 672 (3.7%)<br>535 (2.9%) | -0.07<br>-0.04 |
| /- Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) /- Ischemic stroke; n (%) /- Hemorrhagic stroke; n (%) /- TIA; n (%) /- TIA; n (%) /- Other cerebrovascular disease; n (%) /- Late effects of cerebrovascular disease; n (%) /- Heart failure (CHF); n (%) | 239 (5.3%)<br>8 (0.2%)<br>72 (1.6%)<br>122 (2.7%)<br>94 (2.1%)<br>538 (12.0%) | 20 (0.4%)<br>118 (2.3%)<br>246 (4.8%)<br>203 (4.0%)<br>974 (19.1%) | -0.05<br>-0.11<br>-0.11<br>0.00 | 69 (1.1%)<br>93 (1.5%)<br>67 (1.1%)<br>462 (7.3%) | 77 (1.6%)<br>124 (2.6%)<br>59 (1.2%)<br>511 (10.7%) | -0.04<br>-0.08<br>-0.01<br>-0.12 | 216 (1.7%)<br>365 (2.9%)<br>375 (2.9%)<br>1,842 (14.4%) | 176 (2.1%)<br>302 (3.6%)<br>273 (3.3%)<br>1,573 (18.9%) | -0.03<br>-0.04<br>-0.02<br>-0.12 | 580 (2.5%)<br>536 (2.3%)<br>2,842 (12.0%) | 672 (3.7%)<br>535 (2.9%)<br>3,058 (16.8%) | -0.07<br>-0.04<br>-0.14 |
| /- Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) /- Ischemic stroke; n (%) /- Hemorrhagic stroke; n (%) /- TIA; n (%) /- Other cerebrovascular disease; n (%) /- Late effects of cerebrovascular disease; n (%) /- Late effects of cerebrovascular disease; n (%) /- Heart failure (CHF); n (%) /- Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) | 239 (5.3%)<br>8 (0.2%)<br>72 (1.6%)<br>122 (2.7%)<br>94 (2.1%)<br>538 (12.0%)<br>371 (8.2%) | 20 (0.4%)<br>118 (2.3%)<br>246 (4.8%)<br>203 (4.0%)<br>974 (19.1%)<br>525 (10.3%) | -0.05<br>-0.11<br>-0.11<br>0.00<br>-0.07 | 69 (1.1%)<br>93 (1.5%)<br>67 (1.1%)<br>462 (7.3%)<br>301 (4.7%) | 77 (1.6%)<br>124 (2.6%)<br>59 (1.2%)<br>511 (10.7%)<br>247 (5.2%) | -0.04<br>-0.08<br>-0.01<br>-0.12<br>-0.02 | 216 (1.7%)<br>365 (2.9%)<br>375 (2.9%)<br>1,842 (14.4%)<br>1,056 (8.3%) | 176 (2.1%)<br>302 (3.6%)<br>273 (3.3%)<br>1,573 (18.9%)<br>803 (9.6%) | -0.03<br>-0.04<br>-0.02<br>-0.12<br>-0.05 | 580 (2.5%)<br>536 (2.3%)<br>2,842 (12.0%)<br>1,728 (7.3%) | 672 (3.7%)<br>535 (2.9%)<br>3,058 (16.8%)<br>1,575 (8.7%) | -0.07<br>-0.04<br>-0.14<br>-0.05 |
| /- Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) /- Ischemic stroke; n (%) /- Hemorrhagic stroke; n (%) /- TIA; n (%) /- Late effects of cerebrovascular disease; n (%) /- Late effects of cerebrovascular disease; n (%) /- Heart failure (CHF); n (%) /- Petripheral Vascular Disease (PVD) or PVD Surgery; n (%) /- Other cardiac dysrhythmia; n (%) | 239 (5.3%)<br>8 (0.2%)<br>72 (1.6%)<br>122 (2.7%)<br>94 (2.1%)<br>538 (12.0%)<br>371 (8.2%)<br>651 (14.5%) | 20 (0.4%)<br>118 (2.3%)<br>246 (4.8%)<br>203 (4.0%)<br>974 (19.1%)<br>525 (10.3%)<br>904 (17.8%) | -0.05<br>-0.11<br>-0.11<br>0.00<br>-0.07<br>-0.09 | 69 (1.1%)<br>93 (1.5%)<br>67 (1.1%)<br>462 (7.3%)<br>301 (4.7%)<br>773 (12.2%) | 77 (1.6%)<br>124 (2.6%)<br>59 (1.2%)<br>511 (10.7%)<br>247 (5.2%)<br>653 (13.7%) | -0.04<br>-0.08<br>-0.01<br>-0.12<br>-0.02<br>-0.04 | 216 (1.7%)<br>365 (2.9%)<br>375 (2.9%)<br>1,842 (14.4%)<br>1,056 (8.3%)<br>1,963 (15.4%) | 176 (2.1%)<br>302 (3.6%)<br>273 (3.3%)<br>1,573 (18.9%)<br>803 (9.6%)<br>1,347 (16.2%) | -0.03<br>-0.04<br>-0.02<br>-0.12<br>-0.05<br>-0.02 | 580 (2.5%)<br>536 (2.3%)<br>2,842 (12.0%)<br>1,728 (7.3%)<br>3,387 (14.3%) | 672 (3.7%)<br>535 (2.9%)<br>3,058 (16.8%)<br>1,575 (8.7%)<br>2,904 (16.0%) | -0.07<br>-0.04<br>-0.14<br>-0.05<br>-0.05 |
| /- Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) /- Ischemic stroke; n (%) /- Hemorrhagic stroke; n (%) /- TIA; n (%) /- TIA; n (%) /- Other cerebrovascular disease; n (%) /- Heart failure (CHF); n (%) /- Heart failure (CHF); n (%) /- Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) /- Other cardiac dysrhythmia; n (%) /- Cardiac conduction disorders; n (%) | 239 (5.3%)<br>8 (0.2%)<br>72 (1.6%)<br>122 (2.7%)<br>94 (2.1%)<br>538 (12.0%)<br>371 (8.2%)<br>651 (14.5%)<br>330 (7.3%) | 20 (0.4%)<br>118 (2.3%)<br>246 (4.8%)<br>203 (4.0%)<br>974 (19.1%)<br>525 (10.3%)<br>904 (17.8%)<br>538 (10.6%) | -0.05<br>-0.11<br>-0.11<br>0.00<br>-0.07<br>-0.09<br>-0.12 | 69 (1.1%)<br>93 (1.5%)<br>67 (1.1%)<br>462 (7.3%)<br>301 (4.7%)<br>773 (12.2%)<br>311 (4.9%) | 77 (1.6%)<br>124 (2.6%)<br>59 (1.2%)<br>511 (10.7%)<br>247 (5.2%)<br>653 (13.7%)<br>266 (5.6%) | -0.04<br>-0.08<br>-0.01<br>-0.12<br>-0.02<br>-0.04<br>-0.03 | 216 (1.7%)<br>365 (2.9%)<br>375 (2.9%)<br>1,842 (14.4%)<br>1,056 (8.3%)<br>1,963 (15.4%)<br>1,008 (7.9%) | 176 (2.1%)<br>302 (3.6%)<br>273 (3.3%)<br>1,573 (18.9%)<br>803 (9.6%)<br>1,347 (16.2%)<br>777 (9.3%) | -0.03<br>-0.04<br>-0.02<br>-0.12<br>-0.05<br>-0.02<br>-0.05 | 580 (2.5%)<br>536 (2.3%)<br>2,842 (12.0%)<br>1,728 (7.3%)<br>3,387 (14.3%)<br>1,649 (7.0%) | 672 (3.7%)<br>535 (2.9%)<br>3,058 (16.8%)<br>1,575 (8.7%)<br>2,904 (16.0%)<br>1,581 (8.7%) | -0.07<br>-0.04<br>-0.14<br>-0.05<br>-0.05<br>-0.06 |
| /- Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) /- Ischemic stroke; n (%) /- Henorrhagic stroke; n (%) /- TIA; n (%) /- Other cerebrovascular disease; n (%) Late effects of cerebrovascular disease; n (%) /- Heart failure (CHF); n (%) /- Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) /- Other cardiac dysrhythmia; n (%) /- Cardiac conduction disorders; n (%) /- Other CVD; n (%) | 239 (5.3%)<br>8 (0.2%)<br>72 (1.6%)<br>122 (2.7%)<br>94 (2.1%)<br>538 (12.0%)<br>371 (8.2%)<br>651 (14.5%)<br>330 (7.3%)<br>1,268 (28.2%) | 20 (0.4%)<br>118 (2.3%)<br>246 (4.8%)<br>203 (4.0%)<br>974 (19.1%)<br>525 (10.3%)<br>904 (17.8%)<br>538 (10.6%)<br>1,764 (34.7%) | -0.05<br>-0.11<br>-0.11<br>0.00<br>-0.07<br>-0.09<br>-0.12<br>-0.14 | 69 (1.1%)<br>93 (1.5%)<br>67 (1.1%)<br>462 (7.3%)<br>301 (4.7%)<br>773 (12.2%)<br>311 (4.9%)<br>1,420 (22.4%) | 77 (1.6%)<br>124 (2.6%)<br>59 (1.2%)<br>511 (10.7%)<br>247 (5.2%)<br>653 (13.7%)<br>266 (5.6%)<br>1,311 (27.4%) | -0.04<br>-0.08<br>-0.01<br>-0.12<br>-0.02<br>-0.04<br>-0.03<br>-0.12 | 216 (1.7%)<br>365 (2.9%)<br>375 (2.9%)<br>1,842 (14.4%)<br>1,056 (8.3%)<br>1,963 (15.4%)<br>1,008 (7.9%)<br>3,183 (24.9%) | 176 (2.1%)<br>302 (3.6%)<br>273 (3.3%)<br>1,573 (18.9%)<br>803 (9.6%)<br>1,347 (16.2%)<br>777 (9.3%)<br>2,346 (28.2%) | -0.03<br>-0.04<br>-0.02<br>-0.12<br>-0.05<br>-0.02<br>-0.05<br>-0.05 | 580 (2.5%)<br>536 (2.3%)<br>2,842 (12.0%)<br>1,728 (7.3%)<br>3,387 (14.3%)<br>1,649 (7.0%)<br>5,871 (24.9%) | 672 (3.7%)<br>535 (2.9%)<br>3,058 (16.8%)<br>1,575 (8.7%)<br>2,904 (16.0%)<br>1,581 (8.7%)<br>5,421 (29.8%) | -0.07<br>-0.04<br>-0.14<br>-0.05<br>-0.05<br>-0.06 |
| /- Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) /- Ischemic stroke; n (%) /- TIA; n (%) /- TIA; n (%) /- Late effects of cerebrovascular disease; n (%) /- Late effects of cerebrovascular disease; n (%) /- Heart failure (CHF); n (%) /- Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) /- Other Cardiac dysrhythmia; n (%) /- Cardiac conduction disorders; n (%) /- Other CVD; n (%) /- Medications - ACE inhibitors; n (%) | 239 (5.3%)<br>8 (0.2%)<br>72 (1.6%)<br>122 (2.7%)<br>94 (2.1%)<br>538 (12.0%)<br>371 (8.2%)<br>651 (14.5%)<br>330 (7.3%)<br>1,268 (28.2%)<br>919 (20.4%) | 20 (0.4%)<br>118 (2.3%)<br>246 (4.8%)<br>203 (4.0%)<br>974 (19.1%)<br>525 (10.3%)<br>904 (17.8%)<br>538 (10.6%)<br>1,764 (24.7%)<br>1,236 (24.3%) | -0.05<br>-0.11<br>-0.11<br>0.00<br>-0.07<br>-0.09<br>-0.12<br>-0.14<br>-0.09 | 69 (1.1%)<br>93 (1.5%)<br>67 (1.1%)<br>462 (7.3%)<br>301 (4.7%)<br>773 (12.2%)<br>311 (4.9%)<br>1,420 (22.4%)<br>1,077 (17.0%) | 77 (1.6%)<br>124 (2.6%)<br>59 (1.2%)<br>511 (10.7%)<br>247 (5.2%)<br>653 (13.7%)<br>266 (5.6%)<br>1,311 (27.4%)<br>937 (19.6%) | -0.04<br>-0.08<br>-0.01<br>-0.12<br>-0.02<br>-0.04<br>-0.03<br>-0.12<br>-0.07 | 216 (1.7%)<br>365 (2.9%)<br>375 (2.9%)<br>1,842 (14.4%)<br>1,056 (8.3%)<br>1,963 (15.4%)<br>1,008 (7.9%)<br>3,183 (24.9%)<br>3,436 (26.9%) | 176 (2.1%)<br>302 (3.6%)<br>273 (3.3%)<br>1,573 (18.9%)<br>803 (9.6%)<br>1,347 (16.2%)<br>777 (9.3%)<br>2,346 (28.2%)<br>2,317 (27.8%) | -0.03<br>-0.04<br>-0.02<br>-0.12<br>-0.05<br>-0.02<br>-0.05<br>-0.07<br>-0.02 | 580 (2.5%)<br>536 (2.3%)<br>2,842 (12.0%)<br>1,728 (7.3%)<br>3,387 (14.3%)<br>1,649 (7.0%)<br>5,871 (24.9%)<br>5,432 (23.0%) | 672 (3.7%)<br>535 (2.9%)<br>3,058 (16.8%)<br>1,575 (8.7%)<br>2,904 (16.0%)<br>1,581 (8.7%)<br>5,421 (29.8%)<br>4,490 (24.7%) | -0.07<br>-0.04<br>-0.14<br>-0.05<br>-0.05<br>-0.06<br>-0.11<br>-0.04 |
| /- Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) /- Ischemic stroke; n (%) /- Hemorrhagic stroke; n (%) /- TIA; n (%) /- Other cerebrovascular disease; n (%) /- Late effects of cerebrovascular disease; n (%) /- Late effects of cerebrovascular disease; n (%) /- Lear failure (CHF); n (%) /- Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) /- Other cardiac dysrhythmia; n (%) /- Cardiac conduction disorders; n (%) /- Other CVD; n (%) /- Other CVD; n (%) /- Medications - ACE inhibitors; n (%) /- Medications - ARE; n (%) | 239 (5.3%)<br>8 (0.2%)<br>72 (1.6%)<br>122 (2.7%)<br>94 (2.1%)<br>538 (12.0%)<br>371 (8.2%)<br>651 (14.5%)<br>330 (7.3%)<br>1,268 (28.2%)<br>919 (20.4%)<br>601 (13.4%) | 20 (0.4%)<br>118 (2.3%)<br>246 (4.8%)<br>203 (4.0%)<br>974 (19.1%)<br>525 (10.3%)<br>904 (17.8%)<br>538 (10.6%)<br>1,764 (34.7%)<br>1,236 (24.3%)<br>882 (17.3%) | -0.05<br>-0.11<br>-0.11<br>-0.00<br>-0.07<br>-0.09<br>-0.12<br>-0.14<br>-0.09<br>-0.11 | 69 (1.1%)<br>93 (1.5%)<br>67 (1.1%)<br>462 (7.3%)<br>301 (4.7%)<br>773 (12.2%)<br>311 (4.9%)<br>1,420 (22.4%)<br>1,077 (17.0%)<br>720 (11.4%) | 77 (1.6%)<br>124 (2.6%)<br>59 (1.2%)<br>511 (10.7%)<br>247 (5.2%)<br>653 (13.7%)<br>266 (5.6%)<br>1,311 (27.4%)<br>937 (19.6%)<br>659 (13.8%) | -0.04<br>-0.08<br>-0.01<br>-0.12<br>-0.02<br>-0.04<br>-0.03<br>-0.12<br>-0.07 | 216 (1.7%)<br>365 (2.9%)<br>375 (2.9%)<br>1,842 (14.4%)<br>1,056 (8.3%)<br>1,963 (15.4%)<br>1,008 (7.9%)<br>3,183 (24.9%)<br>3,436 (26.9%)<br>2,108 (16.5%) | 176 (2.1%)<br>302 (3.6%)<br>273 (3.3%)<br>1,573 (18.9%)<br>803 (9.6%)<br>1,347 (16.2%)<br>777 (9.3%)<br>2,346 (28.2%)<br>2,317 (27.8%)<br>1,547 (18.6%) | -0.03<br>-0.04<br>-0.02<br>-0.12<br>-0.05<br>-0.02<br>-0.05<br>-0.07<br>-0.02<br>-0.06 | 580 (2.5%)<br>536 (2.3%)<br>2,842 (12.0%)<br>1,728 (7.3%)<br>3,337 (14.3%)<br>1,649 (7.0%)<br>5,871 (24.9%)<br>5,432 (23.0%)<br>3,429 (14.5%) | 672 (3.7%)<br>535 (2.9%)<br>3,058 (16.8%)<br>1,575 (8.7%)<br>2,904 (16.0%)<br>1,581 (8.7%)<br>5,421 (29.8%)<br>4,490 (24.7%)<br>3,088 (17.0%) | -0.07<br>-0.04<br>-0.14<br>-0.05<br>-0.05<br>-0.06<br>-0.11<br>-0.04<br>-0.07 |
| /- Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) /- Ischemic stroke; n (%) /- Henorrhagic stroke; n (%) /- TLA; n (%) /- TLA; n (%) /- Other cerebrovascular disease; n (%) /- Late effects of cerebrovascular disease; n (%) /- Heart failure (CHF); n (%) /- Peripheral Yascular Disease (PVD) or PVD Surgery; n (%) /- Other cardiac dysrhythmia; n (%) /- Other Cardiac conduction disorders; n (%) /- Other CVD; n (%) /- Medications - ACE inhibitors; n (%) /- Medications - ARS; n (%) /- Medications - Apha blockers; n (%) | 239 (5.3%)<br>8 (0.2%)<br>72 (1.6%)<br>122 (2.7%)<br>94 (2.1%)<br>538 (12.0%)<br>371 (8.2%)<br>651 (14.5%)<br>330 (7.3%)<br>1268 (28.2%)<br>919 (20.4%)<br>601 (13.4%)<br>319 (7.1%) | 20 (0.4%)<br>118 (2.3%)<br>246 (4.8%)<br>203 (4.0%)<br>974 (19.1%)<br>525 (10.3%)<br>904 (17.8%)<br>1,764 (34.7%)<br>1,236 (24.3%)<br>882 (17.3%)<br>480 (9.4%) | -0.05<br>-0.11<br>-0.11<br>-0.11<br>-0.00<br>-0.07<br>-0.09<br>-0.12<br>-0.14<br>-0.09<br>-0.11 | 69 (1.1%)<br>93 (1.5%)<br>67 (1.1%)<br>462 (7.3%)<br>301 (4.7%)<br>773 (12.2%)<br>311 (4.9%)<br>1,420 (22.4%)<br>1,077 (17.0%)<br>720 (11.4%)<br>333 (5.3%) | 77 (1.6%) 124 (2.6%) 59 (1.2%) 511 (10.7%) 247 (5.2%) 653 (13.7%) 266 (5.6%) 1,311 (27.4%) 937 (19.6%) 639 (19.6%) 929 (6.3%) | -0.04<br>-0.08<br>-0.01<br>-0.12<br>-0.02<br>-0.04<br>-0.03<br>-0.12<br>-0.07<br>-0.07 | 216 (1.7%)<br>365 (2.9%)<br>375 (2.9%)<br>1,842 (14.4%)<br>1,056 (8.3%)<br>1,063 (15.4%)<br>1,008 (7.9%)<br>3,183 (24.9%)<br>3,436 (26.9%)<br>2,108 (16.5%)<br>1,308 (10.2%) | 176 (2.1%)<br>302 (3.6%)<br>273 (3.3%)<br>1,573 (18.9%)<br>803 (9.6%)<br>1,347 (16.2%)<br>777 (9.3%)<br>2,346 (28.2%)<br>2,317 (27.8%)<br>1,547 (18.6%)<br>845 (10.1%) | -0.03<br>-0.04<br>-0.02<br>-0.12<br>-0.05<br>-0.02<br>-0.07<br>-0.07<br>-0.06<br>0.00 | 580 (2.5%)<br>536 (2.3%)<br>2,842 (12.0%)<br>1,728 (7.3%)<br>3,387 (14.3%)<br>1,649 (7.0%)<br>5,871 (24.9%)<br>5,432 (23.0%)<br>3,429 (14.5%)<br>1,960 (8.3%) | 672 (3.7%)<br>535 (2.9%)<br>3,058 (16.8%)<br>1,575 (8.7%)<br>2,904 (16.0%)<br>1,581 (8.7%)<br>5,421 (29.8%)<br>4,490 (24.7%)<br>3,088 (17.0%)<br>1,624 (8.9%) | -0.07<br>-0.04<br>-0.14<br>-0.05<br>-0.05<br>-0.06<br>-0.11<br>-0.04<br>-0.07<br>-0.02 |
| /- Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) /- Ischemic stroke; n (%) /- Ischemic stroke; n (%) /- IHchmorrhagic stroke; n (%) /- TIA; n (%) /- Other cerebrovascular disease; n (%) /- Late effects of cerebrovascular disease; n (%) /- Late effects of cerebrovascular disease; n (%) /- Heart failure (CHF); n (%) /- Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) /- Other cardiac dysrhythmia; n (%) /- Other cardiac dysrhythmia; n (%) /- Cardiac conduction disorders; n (%) /- Cother CVD; n (%) /- Wedications - ACBS; n (%) /- Medications - ARBS; n (%) /- Medications - Alpha blockers; n (%) /- Medications - Alpha blockers; n (%) /- Medications - Beta blockers; n (%) | 239 (5.3%)<br>8 (0.2%)<br>72 (1.6%)<br>122 (2.7%)<br>94 (2.1%)<br>538 (12.0%)<br>371 (8.2%)<br>1,268 (28.2%)<br>919 (20.4%)<br>601 (13.4%)<br>319 (7.1%) | 20 (0.4%)<br>118 (2.3%)<br>246 (4.8%)<br>203 (4.0%)<br>974 (19.1%)<br>525 (10.3%)<br>904 (17.8%)<br>538 (10.6%)<br>1,764 (34.7%)<br>1,236 (24.3%)<br>882 (17.3%)<br>882 (17.3%)<br>1,496 (29.4%) | -0.05<br>-0.11<br>-0.11<br>-0.11<br>-0.00<br>-0.07<br>-0.09<br>-0.12<br>-0.14<br>-0.09<br>-0.11<br>-0.08<br>-0.19 | 69 (1.1%)<br>93 (1.5%)<br>67 (1.1%)<br>462 (7.3%)<br>301 (4.7%)<br>773 (12.2%)<br>311 (4.9%)<br>1,420 (22.4%)<br>1,077 (17.0%)<br>720 (11.4%)<br>333 (5.3%)<br>1,112 (17.5%) | 77 (1.6%) 124 (2.6%) 59 (1.2%) 511 (10.7%) 5247 (5.2%) 653 (13.7%) 266 (5.6%) 1,311 (27.4%) 937 (19.6%) 659 (13.8%) 1,052 (22.0%) | -0.04<br>-0.08<br>-0.01<br>-0.12<br>-0.02<br>-0.04<br>-0.03<br>-0.12<br>-0.07<br>-0.07<br>-0.07 | 216 (1.7%)<br>365 (2.9%)<br>375 (2.9%)<br>1,842 (14.4%)<br>1,056 (8.3%)<br>1,963 (15.4%)<br>1,008 (7.9%)<br>3,183 (24.9%)<br>3,436 (26.9%)<br>2,108 (16.5%)<br>1,308 (10.2%)<br>3,972 (31.1%) | 176 (2.1%) 302 (3.6%) 1,573 (18.9%) 803 (9.6%) 1,347 (16.2%) 777 (9.3%) 2,346 (28.2%) 2,317 (27.8%) 1,547 (18.6%) 845 (10.1%) 3,007 (36.1%) | -0.03<br>-0.04<br>-0.02<br>-0.05<br>-0.05<br>-0.05<br>-0.07<br>-0.07<br>-0.02<br>-0.06<br>0.00 | 580 (2.5%)<br>536 (2.3%)<br>2,842 (12.0%)<br>1,728 (7.3%)<br>3,387 (14.3%)<br>1,649 (7.0%)<br>5,871 (24.9%)<br>5,432 (23.0%)<br>3,429 (14.5%)<br>1,960 (8.3%)<br>6,029 (25.5%) | 672 (3.7%)<br>535 (2.9%)<br>3,058 (16.8%)<br>1,575 (8.7%)<br>2,904 (16.0%)<br>1,581 (8.7%)<br>5,421 (29.8%)<br>4,490 (24.7%)<br>3,088 (17.0%)<br>1,624 (8.9%)<br>5,555 (30.5%) | -0.07<br>-0.04<br>-0.14<br>-0.05<br>-0.05<br>-0.06<br>-0.11<br>-0.04<br>-0.07<br>-0.02 |
| V - Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) V - Ischemic stroke; n (%) V - Henorrhagis stroke; n (%) V - TIA; n (%) V - TIA; n (%) V - Other cerebrovascular disease; n (%) V - Late effects of cerebrovascular disease; n (%) V - Late effects of cerebrovascular disease; n (%) V - Letaer failure (CHF); n (%) V - Peripheral Vascular Diseases (PVD) or PVD Surgery; n (%) V - Other cardiac dysrhythmia; n (%) V - Other cardiac odsrchythmia; n (%) V - Other CVD; n (%) V Medications - ACE inhibitors; n (%) V Medications - ARBs; n (%) V Medications - Alpha blockers; n (%) V Medications - Loop Diuretics; n (%) V Medications - Loop Diuretics; n (%) V Medications - Loop Diuretics; n (%) | 239 (5.3%)<br>8 (0.2%)<br>72 (1.6%)<br>122 (2.7%)<br>94 (2.1%)<br>538 (12.0%)<br>371 (8.2%)<br>651 (14.5%)<br>330 (7.3%)<br>1268 (28.2%)<br>919 (20.4%)<br>319 (7.1%)<br>945 (21.0%)<br>442 (9.3%) | 20 (0.4%)<br>118 (2.3%)<br>246 (4.8%)<br>203 (4.0%)<br>974 (19.1%)<br>525 (10.3%)<br>904 (17.8%)<br>538 (10.6%)<br>1,764 (34.7%)<br>1,236 (24.3%)<br>882 (17.3%)<br>480 (9.4%)<br>1,496 (29.4%)<br>750 (14.7%) | -0.05 -0.11 -0.11 -0.11 -0.00 -0.07 -0.09 -0.12 -0.14 -0.09 -0.11 -0.08 -0.19 -0.15 | 69 (1.1%) 93 (1.5%) 67 (1.1%) 462 (7.3%) 301 (4.7%) 773 (12.2%) 311 (4.9%) 1,420 (22.4%) 1,077 (17.0%) 720 (11.4%) 333 (5.3%) 1,112 (17.5%) 373 (5.9%) | 77 (1.6%) 124 (2.6%) 59 (1.2%) 511 (10.7%) 247 (5.2%) 653 (13.7%) 266 (5.6%) 1,311 (27.4%) 937 (19.6%) 659 (13.8%) 299 (6.3%) 1,052 (22.0%) 435 (9.1%) | -0.04<br>-0.08<br>-0.01<br>-0.12<br>-0.02<br>-0.04<br>-0.03<br>-0.12<br>-0.07<br>-0.07<br>-0.04<br>-0.11 | 216 (1.7%)<br>365 (2.9%)<br>375 (2.9%)<br>1,842 (14.4%)<br>1,056 (8.3%)<br>1,008 (7.9%)<br>3,183 (24.9%)<br>2,108 (16.5%)<br>1,308 (10.2%)<br>3,972 (31.1%)<br>1,913 (15.0%) | 176 (2.1%) 302 (3.6%) 273 (3.3%) 1,573 (18.9%) 803 (9.6%) 1,347 (16.2%) 777 (9.3%) 2,346 (28.2%) 2,317 (27.8%) 1,547 (18.6%) 845 (10.1%) 3,007 (36.1%) 1,613 (19.4%) | -0.03<br>-0.04<br>-0.02<br>-0.12<br>-0.05<br>-0.02<br>-0.05<br>-0.07<br>-0.02<br>-0.06<br>0.00<br>-0.11 | 580 (2.5%)<br>536 (2.3%)<br>2,842 (12.0%)<br>1,728 (7.3%)<br>3,387 (14.3%)<br>1,649 (7.0%)<br>5,871 (24.9%)<br>5,432 (23.0%)<br>3,429 (14.5%)<br>1,960 (8.3%)<br>6,029 (25.5%)<br>2,728 (11.5%) | 672 (3.7%)<br>535 (2.9%)<br>3,058 (16.8%)<br>1,575 (8.7%)<br>2,904 (16.0%)<br>1,581 (8.7%)<br>5,421 (29.8%)<br>4,490 (24.7%)<br>3,088 (17.0%)<br>1,624 (8.9%)<br>5,555 (30.5%)<br>2,798 (15.4%) | -0.07<br>-0.04<br>-0.14<br>-0.05<br>-0.05<br>-0.06<br>-0.11<br>-0.04<br>-0.07<br>-0.02<br>-0.11<br>-0.11 |
| V - Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) V - Ischemic stroke; n (%) V - Hemorrhagic stroke; n (%) V - TIA; n (%) V - TIA; n (%) V - Other cerebrovascular disease; n (%) V - Late effects of cerebrovascular disease; n (%) V - Lette failure (CHF); n (%) V - Peripheral Vascular Diseases (PVD) or PVD Surgery; n (%) V - Peripheral Vascular Diseases (PVD) or PVD Surgery; n (%) V - Cardiac conduction disorders; n (%) V - Cardiac conduction disorders; n (%) V - Medications - AEB; n (%) V Medications - ABB; n (%) V Medications - Beta blockers; n (%) V Medications - Beta blockers; n (%) V Medications - Deta Diuretics; n (%) V Medications - Other diuretics; n (%) V Medications - Other diuretics; n (%) | 239 (5.3%)<br>8 (0.2%)<br>72 (1.6%)<br>122 (2.7%)<br>94 (2.1%)<br>538 (12.0%)<br>371 (8.2%)<br>651 (14.5%)<br>330 (7.3%)<br>1,268 (28.2%)<br>919 (20.4%)<br>601 (13.4%)<br>319 (7.1%)<br>945 (21.0%)<br>442 (9.8%)<br>99 (2.2%) | 20 (0.4%), 118 (2.3%) 246 (4.8%) 203 (4.0%) 974 (19.1%) 525 (10.3%) 904 (17.8%) 538 (10.6%) 1,764 (34.7%) 1,236 (24.3%) 882 (17.3%) 480 (9.4%) 1,496 (29.4%) 1,591 (14.7%) 159 (3.1%) | -0.05<br>-0.11<br>-0.11<br>-0.00<br>-0.07<br>-0.09<br>-0.12<br>-0.14<br>-0.09<br>-0.11<br>-0.08<br>-0.19<br>-0.15<br>-0.06 | 69 (1.1%) 93 (1.5%) 67 (1.1%) 462 (7.3%) 301 (4.7%) 773 (12.2%) 311 (4.9%) 1,077 (17.0%) 720 (11.4%) 333 (5.3%) 1,112 (17.5%) 373 (5.9%) 125 (2.0%) | 77 (1.6%) 124 (2.6%) 59 (1.2%) 511 (10.7%) 511 (10.7%) 653 (13.7%) 266 (5.6%) 1,311 (27.4%) 937 (19.6%) 659 (13.8%) 1,052 (22.0%) 435 (9.1%) 120 (2.5%) | -0.04<br>-0.08<br>-0.01<br>-0.12<br>-0.02<br>-0.04<br>-0.03<br>-0.12<br>-0.07<br>-0.07<br>-0.04<br>-0.11<br>-0.12<br>-0.03 | 216 (1.7%)<br>365 (2.9%)<br>375 (2.9%)<br>1,842 (14.4%)<br>1,056 (8.3%)<br>1,063 (15.4%)<br>1,008 (7.9%)<br>3,183 (42.9%)<br>3,436 (26.9%)<br>2,108 (16.5%)<br>1,308 (10.2%)<br>3,972 (31.13%)<br>1,913 (15.0%)<br>346 (2.7%) | 176 (2.1%)<br>302 (3.6%)<br>273 (3.3%)<br>1,573 (18.9%)<br>803 (9.6%)<br>1,347 (16.2%)<br>777 (9.3%)<br>2,346 (28.2%)<br>2,347 (27.8%)<br>4,547 (18.6%)<br>845 (10.1%)<br>3,007 (36.1%)<br>1,613 (19.4%)<br>277 (3.3%) | -0.03<br>-0.04<br>-0.02<br>-0.12<br>-0.05<br>-0.02<br>-0.05<br>-0.07<br>-0.02<br>-0.06<br>0.00<br>-0.11<br>-0.12 | 580 (2.5%)<br>536 (2.3%)<br>2,842 (12.0%)<br>1,728 (7.3%)<br>3,387 (14.3%)<br>1,649 (7.0%)<br>5,432 (23.0%)<br>3,429 (14.5%)<br>1,960 (8.3%)<br>6,029 (25.5%)<br>2,728 (11.5%)<br>570 (2.4%) | 672 (3.7%)<br>535 (2.9%)<br>3,058 (16.8%)<br>1,575 (8.7%)<br>2,904 (16.0%)<br>1,581 (8.7%)<br>5,421 (29.8%)<br>4,490 (24.7%)<br>3,088 (17.0%)<br>1,624 (8.9%)<br>5,555 (30.5%)<br>2,798 (15.4%)<br>556 (3.1%) | -0.07<br>-0.04<br>-0.14<br>-0.05<br>-0.05<br>-0.06<br>-0.11<br>-0.04<br>-0.07<br>-0.02<br>-0.11<br>-0.11 |
| V - Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) V - Ischemic stroke; n (%) V - Hemorrhagic stroke; n (%) V - TIA; n (%) V - TIA; n (%) V - TIA; n (%) V - Late effects of cerebrovascular disease; n (%) V - Late effects of cerebrovascular disease; n (%) V - Hemorrhagic (CHF); n (%) V - Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) V - Other cardiac dysrhythmia; n (%) V - Cardiac conduction disorders; n (%) V - Cardiac conduction disorders; n (%) V - Medications - AEBs, n (%) V Medications - ABBs, n (%) V Medications - Beta blockers; n (%) V Medications - Other diuretics; n (%) V Medications - Other diuretics; n (%) V Medications - Other diuretics; n (%) V Medications - Use of statins; n (%) V Medications - Use of statins; n (%) | 239 (5.3%)<br>8 (0.2%)<br>72 (1.6%)<br>122 (2.7%)<br>94 (2.1%)<br>538 (12.0%)<br>371 (8.2%)<br>651 (14.5%)<br>330 (7.3%)<br>1268 (28.2%)<br>919 (20.4%)<br>319 (7.1%)<br>945 (21.0%)<br>442 (9.3%) | 20 (0.4%)<br>118 (2.3%)<br>246 (4.8%)<br>203 (4.0%)<br>974 (19.1%)<br>525 (10.3%)<br>904 (17.8%)<br>538 (10.6%)<br>1,764 (34.7%)<br>1,236 (24.3%)<br>882 (17.3%)<br>480 (9.4%)<br>1,496 (29.4%)<br>750 (14.7%) | -0.05 -0.11 -0.11 -0.11 -0.00 -0.07 -0.09 -0.12 -0.14 -0.09 -0.11 -0.08 -0.19 -0.15 | 69 (1.1%) 93 (1.5%) 67 (1.1%) 462 (7.3%) 301 (4.7%) 773 (12.2%) 311 (4.9%) 1,420 (22.4%) 1,077 (17.0%) 720 (11.4%) 333 (5.3%) 1,112 (17.5%) 373 (5.9%) | 77 (1.6%) 124 (2.6%) 59 (1.2%) 511 (10.7%) 247 (5.2%) 653 (13.7%) 266 (5.6%) 1,311 (27.4%) 937 (19.6%) 659 (13.8%) 299 (6.3%) 1,052 (22.0%) 435 (9.1%) | -0.04<br>-0.08<br>-0.01<br>-0.12<br>-0.02<br>-0.04<br>-0.03<br>-0.12<br>-0.07<br>-0.07<br>-0.04<br>-0.11 | 216 (1.7%)<br>365 (2.9%)<br>375 (2.9%)<br>1,842 (14.4%)<br>1,056 (8.3%)<br>1,008 (7.9%)<br>3,183 (24.9%)<br>2,108 (16.5%)<br>1,308 (10.2%)<br>3,972 (31.1%)<br>1,913 (15.0%) | 176 (2.1%) 302 (3.6%) 273 (3.3%) 1,573 (18.9%) 803 (9.6%) 1,347 (16.2%) 777 (9.3%) 2,346 (28.2%) 2,317 (27.8%) 1,547 (18.6%) 845 (10.1%) 3,007 (36.1%) 1,613 (19.4%) | -0.03<br>-0.04<br>-0.02<br>-0.12<br>-0.05<br>-0.02<br>-0.05<br>-0.07<br>-0.02<br>-0.06<br>0.00<br>-0.11 | 580 (2.5%)<br>536 (2.3%)<br>2,842 (12.0%)<br>1,728 (7.3%)<br>3,387 (14.3%)<br>1,649 (7.0%)<br>5,871 (24.9%)<br>5,432 (23.0%)<br>3,429 (14.5%)<br>1,960 (8.3%)<br>6,029 (25.5%)<br>2,728 (11.5%) | 672 (3.7%)<br>535 (2.9%)<br>3,058 (16.8%)<br>1,575 (8.7%)<br>2,904 (16.0%)<br>1,581 (8.7%)<br>5,421 (29.8%)<br>4,490 (24.7%)<br>3,088 (17.0%)<br>1,624 (8.9%)<br>5,555 (30.5%)<br>2,798 (15.4%) | -0.07<br>-0.04<br>-0.14<br>-0.05<br>-0.05<br>-0.06<br>-0.11<br>-0.04<br>-0.07<br>-0.02 |

| CV Medications - calcium channel blockers; n (%) | 765 (17.0%) | 1,232 (24.2%) | -0.18 | 835 (13.2%) | 821 (17.2%) | -0.11 | 2,960 (23.2%) | 2,243 (26.9%) | -0.09 | 4,560 (19.3%) | 4,296 (23.6%) | -0.10 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| CV Medications - Use of Low Weight Molecular Heparins; n (%) | 90 (2.0%) | 102 (2.0%) | 0.00 | 162 (2.6%) | 97 (2.0%) | 0.04 | 217 (1.7%) | 158 (1.9%) | -0.02 | 469 (2.0%) | 357 (2.0%) | 0.00 |
| Other Comorbidity - Osteoporosis; n (%) | 345 (7.7%) | 603 (11.9%) | -0.14 | 184 (2.9%) | 156 (3.3%) | -0.02 | 1,464 (11.5%) | 1,109 (13.3%) | -0.05 | 1,993 (8.4%) | 1,868 (10.3%) | -0.07 |
| Other Comorbidity - Dementia; n (%) | 494 (11.0%) | 958 (18.8%) | -0.22 | 223 (3.5%) | 255 (5.3%) | -0.09 | 1,816 (14.2%) | 1,646 (19.8%) | -0.15 | 2,533 (10.7%) | 2,859 (15.7%) | -0.15 |
| Other Comorbidity - Hyperthyroidism + Hypothyroidism + Other disorders of thyroid gland; n | | 1,184 (23.3%) | -0.11 | 863 (13.6%) | 770 (16.1%) | -0.07 | 1,487 (11.6%) | 743 (8.9%) | 0.09 | 3,203 (13.6%) | 2,697 (14.8%) | -0.03 |
| Other Comorbidity - Edema; n (%) | 941 (20.9%) | 1,268 (24.9%) | -0.10 | 986 (15.6%) | 810 (16.9%) | -0.04 | 2,150 (16.8%) | 1,563 (18.8%) | -0.05 | 4,077 (17.3%) | 3,641 (20.0%) | -0.07 |
| Other Comorbidity - Depression; n (%) | 836 (18.6%) | 1,020 (20.1%) | -0.04 | 816 (12.9%) | 635 (13.3%) | -0.01 | 2,678 (20.9%) | 1,758 (21.1%) | 0.00 | 4,330 (18.3%) | 3,413 (18.8%) | -0.01 |
| Other Comorbidity - Anxiety; n (%) | 908 (20.2%) | 1,163 (22.9%) | -0.07 | 921 (14.5%) | 827 (17.3%) | -0.08 | 2,675 (20.9%) | 1,732 (20.8%) | 0.00 | 4,504 (19.1%) | 3,722 (20.5%) | -0.04 |
| Other Comorbidity - Pneumonia; n (%) | 719 (16.0%) | 1,105 (21.7%) | -0.15 | 833 (13.1%) | 729 (15.2%) | -0.06 | 2,169 (17.0%) | 1,518 (18.2%) | -0.03 | 3,721 (15.8%) | 3,352 (18.4%) | -0.07 |
| Other Comorbidity - COPD; n (%) | 772 (17.2%) | 1,163 (22.9%) | -0.14 | 585 (9.2%) | 496 (10.4%) | -0.04 | 2,910 (22.8%) | 2,061 (24.7%) | -0.04 | 4,267 (18.1%) | 3,720 (20.4%) | -0.06 |
| Other Comorbidity - Asthma; n (%) | 479 (10.6%) | 557 (10.9%) | -0.01 | 639 (10.1%) | 489 (10.2%) | 0.00 | 1,573 (12.3%) | 980 (11.8%) | 0.02 | 2,691 (11.4%) | 2,026 (11.1%) | 0.01 |
| Other Comorbidity - Acute renal disease; n (%) | 493 (11.0%) | 960 (18.9%) | -0.22 | 456 (7.2%) | 478 (10.0%) | -0.10 | 1,430 (11.2%) | 1,371 (16.5%) | -0.15<br>0.00 | 2,379 (10.1%) | 2,809 (15.4%) | -0.16<br>-0.02 |
| Other Comorbidity CKD Stage 1; n (%) | 14 (0.3%) | 15 (0.3%) | 0.00 | 11 (0.2%) | 4 (0.1%) | 0.03 | 33 (0.3%) | 28 (0.3%) | | 58 (0.2%) | 47 (0.3%) | |
| Other Comorbidity - CKD Stage 2; n (%) | 88 (2.0%) | 142 (2.8%)<br>712 (14.0%) | -0.05<br>-0.25 | 40 (0.6%) | 46 (1.0%) | -0.04<br>-0.11 | 177 (1.4%) | 168 (2.0%)<br>980 (11.8%) | -0.05<br>-0.20 | 305 (1.3%) | 356 (2.0%)<br>1.895 (10.4%) | -0.05<br>-0.19 |
| Other Comorbidity - CKD Stage 3; n (%) Other Comorbidity - Occurrence of chronic renal insufficiency w/o CKD; n (%) | 295 (6.6%) | 712 (14.0%)<br>473 (9.3%) | -0.25<br>-0.15 | 147 (2.3%)<br>127 (2.0%) | 203 (4.2%) | | 796 (6.2%)<br>679 (5.3%) | 726 (8.7%) | -0.20<br>-0.13 | 1,238 (5.2%)<br>1,051 (4.4%) | 1,384 (7.6%) | -0.19<br>-0.14 |
| Other Comorbidity - Occurrence of chronic renal insufficiency w/o CkD; n (%) Other Comorbidity - Occurrence of miscellaneous renal insufficiency; n (%) | 245 (5.4%) | | -0.15 | | 185 (3.9%) | -0.11<br>-0.05 | | | -0.13 | | | -0.14 |
| Other Comorbidity - Occurrence of miscenaneous renal insufficiency; n (%) Other Comorbidity - Hypertensive nephropathy; n (%) | 385 (8.6%)<br>333 (7.4%) | 553 (10.9%)<br>739 (14.5%) | -0.23 | 324 (5.1%)<br>162 (2.6%) | 301 (6.3%)<br>257 (5.4%) | -0.14 | 905 (7.1%)<br>1,056 (8.3%) | 764 (9.2%)<br>1,275 (15.3%) | -0.22 | 1,614 (6.8%)<br>1,551 (6.6%) | 1,618 (8.9%)<br>2,271 (12.5%) | -0.20 |
| Other Comorbidity - Obstructive sleep apnea; n (%) | 387 (8.6%) | 442 (8.7%) | 0.00 | 626 (9.9%) | 533 (11.1%) | -0.14 | 897 (7.0%) | 602 (7.2%) | -0.22 | 1,910 (8.1%) | 1,577 (8.7%) | -0.02 |
| Other Comorbidity - Osteoarthritis: n (%) | 1.152 (25.6%) | 1,658 (32.6%) | -0.15 | 1.178 (18.6%) | 964 (20.2%) | -0.04 | 4.067 (31.8%) | 2,876 (34.5%) | -0.06 | 6.397 (27.1%) | 5,498 (30.2%) | -0.02 |
| Other Comorbidity - Osteoartinitis, in (%) Other Comorbidity - Other arthritis, arthropathies and musculoskeletal pain; n (%) | 3,025 (67.2%) | 3,460 (68.0%) | -0.13 | 4,026 (63.5%) | 2,894 (60.5%) | 0.06 | 8,043 (62.9%) | 5,180 (62.2%) | 0.01 | 15,094 (63.9%) | 11,534 (63.4%) | 0.01 |
| Other Comorbidity - Other artifitis, artifitopathies and musculoskeletal pain, if (%) | 1.513 (33.6%) | 1.835 (36.1%) | -0.02 | 1,815 (28.6%) | 1,452 (30.4%) | -0.04 | 4,377 (34.2%) | 2.780 (33.4%) | 0.02 | 7.705 (32.6%) | 6,067 (33.3%) | -0.01 |
| Other Comorbidity - Fractures; n (%) | 472 (10.5%) | 647 (12.7%) | -0.03 | 487 (7.7%) | 391 (8.2%) | -0.02 | 1,209 (9.5%) | 845 (10.1%) | -0.02 | 2,168 (9.2%) | 1,883 (10.3%) | -0.01 |
| Other Comorbidity - Fractures, II (%) Other Comorbidity - Falls: n (%) | 502 (11.2%) | 897 (12.7%) | -0.18 | 263 (4.1%) | 243 (5.1%) | -0.02 | 602 (4.7%) | 453 (5.4%) | -0.02 | 1.367 (5.8%) | 1,593 (10.5%) | -0.12 |
| Other Comorbidity - Pais, if (%) Other Comorbidity - Sleep Disorder; n (%) | 217 (4.8%) | 171 (3.4%) | 0.07 | 379 (6.0%) | 159 (3.3%) | 0.13 | 670 (5.2%) | 291 (3.5%) | 0.08 | 1.266 (5.4%) | 621 (3.4%) | 0.10 |
| Other Comorbidity - Delirium: n (%) | 257 (5.7%) | 466 (9.2%) | -0.13 | 142 (2.2%) | 144 (3.0%) | -0.05 | 754 (5.9%) | 646 (7.8%) | -0.08 | 1.153 (4.9%) | 1.256 (6.9%) | -0.08 |
| Other Comorbidity - Psychosis; n (%) | 149 (3.3%) | 191 (3.8%) | -0.03 | 80 (1.3%) | 60 (1.3%) | 0.00 | 775 (6.1%) | 401 (4.8%) | 0.06 | 1,004 (4.2%) | 652 (3.6%) | 0.03 |
| Procedures | () | () | | () | () | | (2/0) | ( | | _, (-,, | (0/0) | |
| Procedure - Hip Surgery; n (%) | 38 (0.8%) | 74 (1.5%) | -0.07 | 55 (0.9%) | 36 (0.8%) | -0.01 | 139 (1.1%) | 87 (1.0%) | 0.01 | 232 (1.0%) | 197 (1.1%) | -0.01 |
| Medications | | | | | | | | | | | | |
| DM Medications - Meglitinides; n (%) | 5 (0.1%) | 6 (0.1%) | 0.00 | 4 (0.1%) | 7 (0.1%) | 0.00 | 35 (0.3%) | 20 (0.2%) | 0.02 | 44 (0.2%) | 33 (0.2%) | 0.00 |
| DM Medications - AGIs; n (%) | 3 (0.1%) | 0 (0.0%) | 0.04 | 1 (0.0%) | 2 (0.0%) | 0.00 | - | | | | | |
| DM Medications - Insulin; n (%) | 176 (3.9%) | 299 (5.9%) | -0.09 | 32 (0.5%) | 26 (0.5%) | 0.00 | 505 (3.9%) | 362 (4.3%) | -0.02 | 713 (3.0%) | 687 (3.8%) | -0.04 |
| DM Medications - Glitazones; n (%) | 20 (0.4%) | 34 (0.7%) | -0.04 | 210 (3.3%) | 221 (4.6%) | -0.07 | 93 (0.7%) | 49 (0.6%) | 0.01 | 323 (1.4%) | 304 (1.7%) | -0.02 |
| DM Medications - 1st and 2nd Generation SUs; n (%) | 176 (3.9%) | 292 (5.7%) | -0.08 | 201 (3.2%) | 194 (4.1%) | -0.05 | 640 (5.0%) | 466 (5.6%) | -0.03 | 1,017 (4.3%) | 952 (5.2%) | -0.04 |
| DM Medications - DPP-4 Inhibitors; n (%) | 63 (1.4%) | 116 (2.3%) | -0.07 | 97 (1.5%) | 115 (2.4%) | -0.07 | 279 (2.2%) | 219 (2.6%) | -0.03 | 439 (1.9%) | 450 (2.5%) | -0.04 |
| DM Medications - GLP-1 RA; n (%) | 27 (0.6%) | 56 (1.1%) | -0.05 | 53 (0.8%) | 54 (1.1%) | -0.03 | 58 (0.5%) | 47 (0.6%) | -0.01 | 138 (0.6%) | 157 (0.9%) | -0.03 |
| DM Medications - SGLT-2 Inhibitors ; n (%) | 37 (0.8%) | 48 (0.9%) | -0.01 | 68 (1.1%) | 57 (1.2%) | -0.01 | 59 (0.5%) | 40 (0.5%) | 0.00 | 164 (0.7%) | 145 (0.8%) | -0.01 |
| DM Medications - Metformin; n (%) | 362 (8.0%) | 615 (12.1%) | -0.14 | 509 (8.0%) | 438 (9.2%) | -0.04 | 1,357 (10.6%) | 841 (10.1%) | 0.02 | 2,228 (9.4%) | 1,894 (10.4%) | -0.03 |
| DM Medciations - All antidiabetic medications except Insulin; n (%) | 465 (10.3%) | 808 (15.9%) | -0.17 | 645 (10.2%) | 576 (12.0%) | -0.06 | 1,775 (13.9%) | 1,188 (14.3%) | -0.01 | 2,885 (12.2%) | 2,572 (14.1%) | -0.06 |
| Other Medications - Use of NSAIDs; n (%) | 887 (19.7%) | 936 (18.4%) | 0.03 | 1,479 (23.3%) | 1,054 (22.0%) | 0.03 | 2,647 (20.7%) | 1,646 (19.8%) | 0.02 | 5,013 (21.2%) | 3,636 (20.0%) | 0.03 |
| Other Medications - Use of other hypertension drugs; n (%) | 174 (3.9%) | 296 (5.8%) | -0.09 | 178 (2.8%) | 161 (3.4%) | -0.03 | 747 (5.8%) | 554 (6.7%) | -0.04 | 1,099 (4.7%) | 1,011 (5.6%) | -0.04 |
| Other Medications - Digoxin; n (%) | 17 (0.4%) | 18 (0.4%) | 0.00 | 12 (0.2%) | 19 (0.4%) | -0.04 | 83 (0.6%) | 56 (0.7%) | -0.01 | 112 (0.5%) | 93 (0.5%) | 0.00 |
| Other Medications - Use of Anti-arrhythmics; n (%) | 17 (0.4%) | 27 (0.5%) | -0.01 | 19 (0.3%) | 30 (0.6%) | -0.04 | 57 (0.4%) | 53 (0.6%) | -0.03 | 93 (0.4%) | 110 (0.6%) | -0.03 |
| Other Medications - Use of antipsychotics; n (%) | 263 (5.8%) | 357 (7.0%) | -0.05 | 230 (3.6%) | 214 (4.5%) | -0.05 | 1,436 (11.2%) | 864 (10.4%) | 0.03 | 1,929 (8.2%) | 1,435 (7.9%) | 0.01 |
| Other Medications - Use of dementia meds; n (%) | 210 (4.7%) | 386 (7.6%) | -0.12 | 94 (1.5%) | 105 (2.2%) | -0.05 | 936 (7.3%) | 800 (9.6%) | -0.08 | 1,240 (5.2%) | 1,291 (7.1%) | -0.08 |
| Other Medications - Use of antiparkinsonian meds; n (%) | 148 (3.3%) | 193 (3.8%) | -0.03 | 139 (2.2%) | 118 (2.5%) | -0.02 | 722 (5.6%) | 493 (5.9%) | -0.01 | 1,009 (4.3%) | 804 (4.4%) | 0.00 |
| Other Medications - Use of anxiolytics/hypnotics; n (%) | 291 (6.5%) | 330 (6.5%) | 0.00 | 443 (7.0%) | 362 (7.6%) | -0.02 | 1,091 (8.5%) | 679 (8.2%) | 0.01 | 1,825 (7.7%) | 1,371 (7.5%) | 0.01 |
| Other Medications - Use of anticonvulsants; n (%) | 738 (16.4%) | 1,036 (20.4%) | -0.10 | 844 (13.3%) | 718 (15.0%) | -0.05 | 2,968 (23.2%) | 1,871 (22.5%) | 0.02 | 4,550 (19.3%) | 3,625 (19.9%) | -0.02 |
| Other Medications - Use of antidepressants; n (%) | 1,187 (26.4%) | 1,520 (29.9%) | -0.08 | 1,443 (22.8%) | 1,205 (25.2%) | -0.06 | 4,303 (33.7%) | 2,949 (35.4%) | -0.04 | 6,933 (29.3%) | 5,674 (31.2%) | -0.04 |
| Other Medications - Use of lithium; n (%) | 13 (0.3%) | 14 (0.3%) | 0.00 | 21 (0.3%) | 15 (0.3%) | 0.00 | 79 (0.6%) | 40 (0.5%) | 0.01 | 113 (0.5%) | 69 (0.4%) | 0.01 |
| Other Medications - Use of Benzos; n (%) | 686 (15.2%) | 792 (15.6%) | -0.01 | 929 (14.7%) | 734 (15.4%) | -0.02 | 2,714 (21.2%) | 1,762 (21.2%) | 0.00 | 4,329 (18.3%) | 3,288 (18.1%) | 0.01 |
| Other Medication - Use of CNS stimulants; n (%) | 39 (0.9%) | 47 (0.9%) | 0.00 | 100 (1.6%) | 75 (1.6%) | 0.00 | 94 (0.7%) | 49 (0.6%) | 0.01 | 233 (1.0%) | 171 (0.9%) | 0.01 |
| Other Medications - Use of opioids; n (%) | 1,901 (42.3%) | 1,922 (37.8%) | 0.09 | 3,029 (47.8%) | 2,095 (43.8%) | 0.08 | 5,620 (44.0%) | 3,499 (42.0%) | 0.04 | 10,550 (44.7%) | 7,516 (41.3%) | 0.07 |
| Other Medications - Use of COPD/asthma meds; n (%) | 728 (16.2%) | 1,062 (20.9%) | -0.12 | 1,010 (15.9%) | 803 (16.8%) | -0.02 | 2,991 (23.4%) | 1,969 (23.6%) | 0.00 | 4,729 (20.0%) | 3,834 (21.1%) | -0.03 |
| Other Medications - Use of oral corticosteroids; n (%) | 1,204 (26.8%) | 1,433 (28.2%) | -0.03 | 1,628 (25.7%) | 1,307 (27.3%) | -0.04 | 3,906 (30.5%) | 2,715 (32.6%) | | 6,738 (28.5%) | 5,455 (30.0%) | -0.03 |
| Other Medications - Use of Sympatomimetic agents; n (%) | 68 (1.5%) | 58 (1.1%) | 0.04 | 156 (2.5%) | 135 (2.8%) | -0.02 | 143 (1.1%) | 73 (0.9%) | 0.02 | 367 (1.6%) | 266 (1.5%) | 0.01 |
| Other Medications - Use of bisphosphonates; n (%) Other Medications - Use of thiazide; n (%) | 121 (2.7%)<br>329 (7.3%) | 188 (3.7%)<br>448 (8.8%) | -0.06<br>-0.06 | 67 (1.1%)<br>363 (5.7%) | 49 (1.0%)<br>362 (7.6%) | 0.01<br>-0.08 | 502 (3.9%)<br>1,249 (9.8%) | 337 (4.0%)<br>831 (10.0%) | -0.01<br>-0.01 | 690 (2.9%)<br>1,941 (8.2%) | 574 (3.2%)<br>1,641 (9.0%) | -0.02<br>-0.03 |
| Other Medications - Use of thiazide; n (%) Other Medications - Use of estrogens, progestins, androgens; n (%) | 329 (7.3%)<br>388 (8.6%) | 448 (8.8%)<br>281 (5.5%) | 0.12 | 363 (5.7%)<br>872 (13.8%) | 362 (7.6%)<br>617 (12.9%) | -0.08 | 1,249 (9.8%)<br>578 (4.5%) | 831 (10.0%)<br>371 (4.5%) | -0.01 | 1,941 (8.2%) | 1,641 (9.0%) | -0.03 |
| Other Medications - Use of estrogens, progestins, androgens; n (%) Healthcare Utilization | J00 (0.U/b) | 201 (3.3%) | J.12 | 3/2 (13.876) | 01/ (12.370) | 0.05 | 3/0 (4.3%) | 3/1 (4.370) | 0.00 | 1,000 (7.8%) | 1,203 (7.0%) | V.U3 |
| HU - Bone mineral density; n (%) | 120 (2.7%) | 164 (3.2%) | -0.03 | 86 (1.4%) | 73 (1.5%) | -0.01 | 490 (3.8%) | 331 (4.0%) | -0.01 | 696 (2.9%) | 568 (3.1%) | -0.01 |
| HU - Occurrence of creatinine tests ordered ; n (%) | 250 (5.6%) | 330 (6.5%) | -0.03 | 264 (4.2%) | 203 (4.2%) | 0.00 | 490 (3.8%)<br>878 (6.9%) | 586 (7.0%) | 0.00 | 1,392 (5.9%) | 1,119 (6.1%) | -0.01 |
| HU - Occurrence of creatinine tests ordered ; n (%) HU - Number of D-dimer tests | 230 (3.0/6) | JJU (U.J/b) | -0.04 | 204 (4.276) | دان (۱۹۰۵/۱۰) | 0.00 | 3/0 (0.3%) | JOU (1.U%) | 0.00 | 1,374 (3.9%) | 1,117 (0.1%) | -0.01 |
| mean (sd) | 0.11 (0.35) | 0.11 (0.35) | 0.00 | 0.13 (0.38) | 0.12 (0.38) | 0.03 | 0.11 (0.35) | 0.10 (0.33) | 0.03 | 0.12 (0.36) | 0.11 (0.35) | 0.03 |
| median (IOR) | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.12 (0.38) | 0.03 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.03 | 0.12 (0.36) | 0.00 (0.35) | 0.03 |
| HU - Number of CRP, high-sensitivity CRP tests | 00 [0.00, 0.00] | 2.00 [0.00, 0.00] | 3.00 | 3.00 [0.00, 0.00] | 2.00 [0.00, 0.00] | 5.00 | 5.55 [5.55, 6.50] | 2.00 [0.00, 0.00] | | 0.00 (0.50) | 0.00 (0.33) | 2.00 |
| mean (sd) | 0.12 (0.55) | 0.12 (0.52) | 0.00 | 0.10 (0.47) | 0.11 (0.58) | -0.02 | 0.15 (0.59) | 0.16 (0.64) | -0.02 | 0.13 (0.55) | 0.14 (0.59) | -0.02 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.55) | 0.00 (0.59) | 0.00 |
| HU - Colonoscopy; n (%) | 157 (3.5%) | 172 (3.4%) | 0.01 | 223 (3.5%) | 200 (4.2%) | -0.04 | 475 (3.7%) | 282 (3.4%) | 0.02 | 855 (3.6%) | 654 (3.6%) | 0.00 |
| HU - Flu vaccine; n (%) | 641 (14.2%) | 728 (14.3%) | 0.00 | 615 (9.7%) | 472 (9.9%) | -0.01 | 3,737 (29.2%) | 2,445 (29.4%) | 0.00 | 4,993 (21.1%) | 3,645 (20.0%) | 0.03 |
| HU - Mammogram; n (%) | 346 (7.7%) | 422 (8.3%) | -0.02 | 453 (7.1%) | 379 (7.9%) | -0.03 | 1,175 (9.2%) | 733 (8.8%) | 0.01 | 1.974 (8.4%) | 1.534 (8.4%) | 0.00 |
| HU - PSA test or Prostate exam for DRE; n (%) | 387 (8.6%) | 401 (7.9%) | 0.03 | 562 (8.9%) | 412 (8.6%) | 0.01 | 1,144 (8.9%) | 729 (8.8%) | 0.00 | 2,093 (8.9%) | 1,542 (8.5%) | 0.01 |
| HU - Pap smear; n (%) | 186 (4.1%) | 140 (2.8%) | 0.03 | 417 (6.6%) | 267 (5.6%) | 0.01 | 349 (2.7%) | 185 (2.2%) | 0.03 | 952 (4.0%) | 592 (3.3%) | 0.01 |
| | 912 (20.3%) | 1,104 (21.7%) | -0.03 | 661 (10.4%) | 640 (13.4%) | -0.09 | 3,585 (28.0%) | 2,718 (32.6%) | -0.10 | 5,158 (21.8%) | 4,462 (24.5%) | -0.06 |
| HU - Pneumonia vaccine; n (%) | | , | | | | | ,, | , | | -, (, | , . ,/ | |
| Frailty Score: Empirical Version 365 days (ICD-9 and ICD-10) V2mean (sd) | 0.19 (0.07) | 0.21 (0.08) | -0.27 | 0.16 (0.05) | 0.17 (0.06) | -0.18 | 0.21 (0.07) | 0.22 (0.08) | -0.13 | 0.19 (0.07) | 0.20 (0.08) | -0.13 |
| Frailty Score: Empirical Version 365 days (ICD-9 and ICD-10) V2mean (sd) | 0.19 (0.07) | | | | | -0.18<br>-0.18 | | | | | | -0.13<br>-0.13 |
| Frailty Score: Empirical Version 365 days (ICD-9 and ICD-10) V2mean (sd)median [IQR] | | 0.21 (0.08)<br>0.20 [0.15, 0.26] | -0.27<br>-0.40 | 0.16 (0.05)<br>0.15 [0.12, 0.18] | 0.17 (0.06)<br>0.16 [0.13, 0.19] | | 0.21 (0.07)<br>0.19 [0.15, 0.25] | 0.22 (0.08)<br>0.20 [0.16, 0.26] | -0.13<br>-0.13 | 0.19 (0.07)<br>0.18 (0.07) | 0.20 (0.08)<br>0.19 (0.08) | |
| Frailty Score: Empirical Version 365 days (ICD-9 and ICD-10) V2mean (sd) | 0.19 (0.07) | | | | | | | | | | | |
| Frailty Score: Empirical Version 365 days (ICD-9 and ICD-10) V2mean [cd]median [lQR] CHADS2 score, 180 days | 0.19 (0.07)<br>0.17 [0.14, 0.22] | 0.20 [0.15, 0.26] | -0.40 | 0.15 [0.12, 0.18] | 0.16 [0.13, 0.19] | -0.18 | 0.19 [0.15, 0.25] | 0.20 [0.16, 0.26] | -0.13 | 0.18 (0.07) | 0.19 (0.08) | -0.13 |
| Frailty Score: Empirical Version 365 days (ICD-9 and ICD-10) V2mean (sd)median [IQR] CHADS2 Score, 180 daysmean (sd) | 0.19 (0.07)<br>0.17 [0.14, 0.22]<br>0.80 (1.04) | 0.20 [0.15, 0.26]<br>1.18 (1.20) | -0.40 | 0.15 [0.12, 0.18]<br>0.60 (0.91) | 0.16 [0.13, 0.19]<br>0.66 (0.98) | -0.18 | 0.19 [0.15, 0.25]<br>0.90 (1.03) | 0.20 [0.16, 0.26] | -0.13 | 0.18 (0.07) | 0.19 (0.08)<br>0.87 (1.01) | -0.13<br>-0.07 |

| 4.0 | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| .mean (sd)<br>.median [IQR] | 1.18 (0.55)<br>1.00 [1.00, 1.00] | 1.25 (0.66)<br>1.00 [1.00, 1.00] | -0.12<br>0.00 | 1.13 (0.41)<br>1.00 [1.00, 1.00] | 1.15 (0.46)<br>1.00 [1.00, 1.00] | -0.05<br>0.00 | 1.30 (0.73)<br>1.00 [1.00, 1.00] | 1.31 (0.67)<br>1.00 [1.00, 1.00] | -0.01<br>0.00 | 1.23 (0.63)<br>1.00 (0.63) | 1.25 (0.62)<br>1.00 (0.62) | -0.03<br>0.00 |
| IU - Number of hospital days | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.00 | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.00 | 1.00 [1.00, 1.00] | 1.00 [1.00, 1.00] | 0.00 | 1.00 (0.03) | 1.00 (0.02) | 0.00 |
| .mean (sd) | 5.54 (7.53) | 7.01 (9.17) | -0.18 | 4.83 (6.87) | 5.47 (8.41) | -0.08 | 6.63 (8.92) | 6.78 (7.60) | -0.02 | 5.94 (8.16) | 6.50 (8.28) | -0.07 |
| .median [IQR] | 4.00 [3.00, 6.00] | 4.00 [3.00, 7.00] | 0.00 | | 4.00 [2.00, 5.00] | -0.13 | | 4.00 [3.00, 7.00] | 0.00 | 3.73 (8.16) | 4.00 (8.28) | -0.03 |
| IU - Number of Emergency Department (ED) visits | 4.00 [5.00, 6.00] | 4.00 [5.00, 7.00] | 0.00 | 3.00 [2.00, 3.00] | 4.00 [2.00, 5.00] | 0.13 | 4.00 [5.00, 7.00] | 4.00 [5.00, 7.00] | 0.00 | 5.75 (0.20) | 4.00 (0.20) | 0.03 |
| .mean (sd) | 1.66 (2.41) | 1.83 (2.28) | -0.07 | 3.07 (4.52) | 3.35 (5.71) | -0.05 | 2.26 (8.21) | 2.12 (3.30) | 0.02 | 2.36 (6.56) | 2.36 (3.87) | 0.00 |
| .median [IQR] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 0.00 | 2.00 [0.00, 4.00] | 2.00 [0.00, 4.00] | 0.00 | 1.00 [1.00, 3.00] | 1.00 [1.00, 3.00] | 0.00 | 1.27 (6.56) | 1.26 (3.87) | 0.00 |
| IU - Number of internal medicine/family medicine visits | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 0.00 | 2.00 [0.00, 4.00] | 2.00 [0.00, 4.00] | 0.00 | 1.00 [1.00, 3.00] | 1.00 [1.00, 3.00] | 0.00 | 1.27 (0.30) | 1.20 (3.07) | 0.00 |
| .mean (sd) | 9.55 (14.11) | 12.64 (16.03) | -0.20 | 5.11 (7.96) | 5.61 (9.10) | -0.06 | 10.96 (11.24) | 11.46 (10.71) | -0.05 | 9.12 (11.10) | 10.25 (12.09) | -0.10 |
| .median [IQR] | | | -0.20 | | 3.00 [1.00, 7.00] | 0.00 | | 9.00 [5.00, 15.00] | | | | -0.10 |
| | 5.00 [2.00, 12.00] | 8.00 [3.00, 16.00] | -0.20 | 3.00 [1.00, 6.00] | 3.00 [1.00, 7.00] | 0.00 | 8.00 [4.00, 14.00] | 9.00 [5.00, 15.00] | -0.09 | 6.09 (11.10) | 7.14 (12.09) | -0.09 |
| IU - Number of different/distinct medication prescriptions | 7.05 (5.27) | 0.00 (5.40) | -0.21 | 7.55 (5.10) | 0.25 (5.22) | -0.13 | 0.54 (5.35) | 10.03 (5.31) | 0.00 | 0.70 (5.20) | 0.20 (5.20) | -0.11 |
| .mean (sd) | 7.95 (5.27) | 9.08 (5.48) | | 7.55 (5.18) | 8.25 (5.32) | | 9.54 (5.35) | 10.02 (5.31) | -0.09 | 8.70 (5.29) | 9.29 (5.36) | |
| median [IQR] | 7.00 [4.00, 11.00] | 8.00 [5.00, 12.00] | -0.19 | 6.00 [4.00, 10.00] | 7.00 [4.00, 11.00] | -0.19 | 9.00 [6.00, 12.00] | 9.00 [6.00, 13.00] | 0.00 | 7.81 (5.29) | 8.19 (5.36) | -0.07 |
| U Total N distinct ICD9/ICD10 diagnoses at the 3rd digit level | | | | | | | | | | | | |
| .mean (sd) | 12.59 (13.28) | 18.31 (15.13) | -0.40 | 8.39 (9.96) | 11.92 (11.17) | -0.33 | 14.89 (13.11) | 17.85 (13.14) | -0.23 | 12.71 (12.38) | 16.42 (13.26) | -0.29 |
| .median [IQR] | 9.00 [1.00, 19.00] | 15.00 [7.00, 26.00] | -0.42 | 5.00 [0.00, 14.00] | 11.00 [2.00, 18.00] | -0.57 | 13.00 [4.00, 22.00] | 16.00 [8.00, 25.00] | -0.23 | 10.09 (12.38) | 14.41 (13.26) | -0.34 |
| U - Number of Office visits | | | | | | | | | | | | |
| mean (sd) | 4.38 (4.11) | 4.56 (4.04) | -0.04 | 4.32 (4.06) | 4.47 (4.13) | -0.04 | 11.38 (13.70) | 11.16 (11.88) | 0.02 | 8.15 (10.45) | 7.56 (8.58) | 0.06 |
| median [IQR] | 3.00 [1.00, 6.00] | 4.00 [2.00, 6.00] | -0.25 | 3.00 [1.00, 6.00] | 4.00 [2.00, 6.00] | -0.24 | 8.00 [3.00, 15.00] | 8.00 [3.00, 15.00] | 0.00 | 5.71 (10.45) | 5.83 (8.58) | -0.01 |
| U - Number of Cardiologist visits | | | | | | | | | | | | |
| mean (sd) | 2.32 (3.74) | 2.91 (4.20) | -0.15 | 0.61 (1.84) | 0.74 (2.03) | -0.07 | 2.52 (3.93) | 2.83 (4.43) | -0.07 | 1.97 (3.45) | 2.30 (3.87) | -0.09 |
| median [IQR] | 1.00 [0.00, 3.00] | 1.00 [0.00, 4.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 1.00] | 0.00 | 1.00 [0.00, 3.00] | 1.00 [0.00, 4.00] | 0.00 | 0.73 (3.45) | 0.74 (3.87) | 0.00 |
| U - Number electrocardiograms | | | | | | | | | | | | |
| mean (sd) | 1.79 (1.98) | 2.06 (2.21) | -0.13 | 0.75 (1.19) | 0.80 (1.23) | -0.04 | 1.93 (2.08) | 1.99 (1.96) | -0.03 | 1.59 (1.86) | 1.70 (1.88) | -0.06 |
| median [IQR] | 1.00 [1.00, 2.00] | 2.00 [1.00, 3.00] | -0.48 | 0.00 [0.00, 1.00] | 0.00 [0.00, 1.00] | 0.00 | 1.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | -0.49 | 0.73 (1.86) | 1.47 (1.88) | -0.40 |
| U - Number of echocardiograms | | | | | | | | | | | | |
| mean (sd) | 1.07 (3.06) | 1.16 (3.08) | -0.03 | 0.61 (0.71) | 0.70 (0.77) | -0.12 | 0.73 (0.93) | 0.80 (0.97) | -0.07 | 0.76 (1.54) | 0.87 (1.80) | -0.07 |
| median (IQR) | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.00 | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.00 | 1.00 [0.00, 1.00] | 1.00 [0.00, 1.00] | 0.00 | 1.00 (1.54) | 1.00 (1.80) | 0.00 |
| U - Number of neurologist visits | | (,, | | | | | () | () | | () | () | |
| mean (sd) | 0.53 (2.11) | 0.71 (2.70) | -0.07 | 0.30 (1.41) | 0.43 (2.85) | -0.06 | 0.51 (2.05) | 0.59 (2.52) | -0.03 | 0.46 (1.91) | 0.58 (2.66) | -0.05 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (1.91) | 0.00 (2.66) | 0.00 |
| U - Fecal occult blood (FOB) test; n (%) U - Number of PT or aPTTt tests | 122 (2.7%) | 114 (2.2%) | 0.03 | 176 (2.8%) | 124 (2.6%) | 0.01 | 308 (2.4%) | 221 (2.7%) | -0.02 | 606 (2.6%) | 459 (2.5%) | 0.00 |
| | 0.44(4.45) | 0.54 (4.05) | 0.00 | 0.40(4.04) | 0.45 (4.40) | 0.00 | 0.05 (0.55) | 0.05 (0.65) | 0.00 | 0.04 (0.00) | 0.00 (4.00) | |
| .mean (sd) | 0.44 (1.15) | 0.51 (1.26) | -0.06 | 0.43 (1.04) | 0.45 (1.18) | -0.02 | 0.26 (0.65) | 0.25 (0.65) | 0.02 | 0.34 (0.88) | 0.38 (1.00) | -0.04 |
| median [IQR] | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.00] | 0.00 | 0.00 (0.88) | 0.00 (1.00) | 0.00 |
| l of days in database anytime prior | | | | | | | | | | | | |
| .mean (sd) | 1,791.06 (1,353.03) | 1,916.04 (1,463.00) | -0.09 | | ) 2,298.62 (1,602.77) | -0.09 | 715.30 (383.18) | 742.93 (368.81) | -0.07 | 1309.06 (1023.95) | | |
| .median [IQR] | 1,406.00 [684.00, 2,6 | 3. 1,475.00 [741.00, 2,7 | 99 -0.05 | 1,847.00 [812.00, 3 | 3, 2,022.00 [872.50, 3,4 | 2 -0.11 | 644.00 [486.00, 830 | 675.00 [518.00, 89 | (-0.08 | 1111.92 (1023.95) | 1252.55 (1155.63) | -0.13 |
| ocioeconomic Status Proxy Variables | | | | | | | | | | | | |
| ES - Mean Copay for per prescription cost (charges in U.S. \$) | | | | | | | | | | | | |
| mean (sd) | 18.46 (26.31) | 18.38 (27.06) | 0.00 | 12.27 (21.28) | 11.83 (19.16) | 0.02 | 18.70 (36.80) | 19.70 (48.22) | -0.02 | 16.93 (31.41) | 17.26 (36.95) | -0.01 |
| median [IQR] | 12.11 [4.29, 24.08] | 10.72 [4.02, 23.29] | 17.55 | 7.50 [0.96, 15.55] | 7.30 [1.00, 15.00] | 0.01 | | 9.93 [2.88, 24.06] | | 9.23 (31.41) | 9.46 (36.95) | -0.01 |
| Missing; n (%) | 479 (10.6%) | 370 (7.3%) | 0.12 | 1,021 (16.1%) | 1,094 (22.9%) | -0.17 | 1,930 (15.1%) | 453 (5.4%) | 0.32 | 3,430 (14.5%) | 1,917 (10.5%) | 0.12 |
| S - Copay: pharmacy cost | | | | | | | | | | | | |
| mean (sd) | 161.56 (270.51) | 184.68 (336.22) | -0.08 | 99.03 (224.48) | 91.21 (179.55) | 0.04 | 181.04 (376.97) | 226.18 (755.70) | -0.08 | 155.32 (323.07) | 179.12 (549.07) | -0.05 |
| median [IQR] | 65.00 [8.28, 207.12] | 72.61 [14.35, 228.00] | -0.02 | 24.78 [0.00, 117.74 | [ 16.90 [0.00, 107.17] | 0.04 | 55.69 [2.93, 202.24 | 79.75 [17.63, 254. | 7 -0.04 | 49.17 (323.07) | 61.24 (549.07) | -0.03 |
| S - Business type: Commercial vs Medicare | | | | | | | | | | | | |
| Commerical; n (%) | 2,178 (48.4%) | 1,399 (27.5%) | 0.44 | 4,978 (78.5%) | 3,523 (73.7%) | 0.11 | 0 (0.0%) | 0 (0.0%) | 0.00 | 7,156 (30.3%) | 4,922 (27.0%) | 0.07 |
| Medicare; n (%) | 2,321 (51.6%) | 3,688 (72.5%) | -0.44 | 1,361 (21.5%) | 1,258 (26.3%) | -0.11 | 0 (0.0%) | 0 (0.0%) | 0.00 | 3,682 (15.6%) | 4,946 (27.2%) | -0.29 |
| ES - Low income indicator; n (%) | 615 (13.7%) | 931 (18.3%) | -0.13 | 0 (0.0%) | 0 (0.0%) | 0.00 | 0 (0.0%) | 0 (0.0%) | 0.00 | 615 (2.6%) | 931 (5.1%) | -0.13 |
| S - Urban vs Rural (MSA variable) | 013 (13.770) | 332 (10.3/0) | 0.13 | 5 (0.070) | 5 (5.070) | 0.00 | J (J.0/0) | 5 (5.0/0) | 0.00 | 513 (2.0/0) | 332 (3.1/0) | 3.13 |
| Urban; n (%) | 0 (0.0%) | 0 (0.0%) | 0.00 | 4,492 (70.9%) | 3,008 (62.9%) | 0.17 | 0 (0.0%) | 0 (0.0%) | 0.00 | 4,492 (19.0%) | 3,008 (16.5%) | 0.07 |
| | | | | | | | | | | | | 0.07 |
| Rural; n (%) | 0 (0.0%) | 0 (0.0%) | 0.00 | 407 (6.4%) | 557 (11.7%) | -0.19 | 0 (0.0%) | 0 (0.0%) | 0.00 | 4,492 (19.0%) | 557 (3.1%) | |
| Unknown/Missing; n (%) | 0 (0.0%) | 0 (0.0%) | 0.00 | 1,440 (22.7%) | 1,216 (25.4%) | -0.06 | 0 (0.0%) | 0 (0.0%) | 0.00 | 1,440 (6.1%) | 1,216 (6.7%) | -0.02 |
| S - Dual Status; n (%) | 0 (0.0%) | 0 (0.0%) | 0.00 | 0 (0.0%) | 0 (0.0%) | 0.00 | 4,066 (31.8%) | 2,524 (30.3%) | 0.03 | 4,066 (17.2%) | 2,524 (13.9%) | 0.09 |
| S - Generic name prescription - unique value | | | | | | | | | | | | |
| mean (sd) | 7.95 (5.27) | 9.08 (5.48) | -0.21 | 7.55 (5.18) | 8.25 (5.32) | -0.13 | 9.54 (5.35) | 10.02 (5.31) | -0.09 | 8.70 (5.29) | 9.29 (5.36) | -0.11 |
| median [IQR] | 7.00 [4.00, 11.00] | 8.00 [5.00, 12.00] | -0.19 | 6.00 [4.00, 10.00] | 7.00 [4.00, 11.00] | -0.19 | 9.00 [6.00, 12.00] | 9.00 [6.00, 13.00] | 0.00 | 7.81 (5.29) | 8.19 (5.36) | -0.07 |
| S - Brand name prescription - unique value | | | | | | | | | | | | |
| | | | 0.04 | | 0.04 (5.40) | -0.13 | 0.65 (5.46) | 10 12 (5 41) | -0.09 | 8.80 (5.40) | 9.39 (5.46) | -0.11 |
| .mean (sd) | 8.04 (5.38) | 9.17 (5.59) | -0.21 | 7.64 (5.28) | 8.34 (5.42) | -0.13 | 9.65 (5.46) | 10.13 (5.41) | -0.09 | 0.00 (3.40) | | |

| | | Ontro | Matched | l | NA wheat com | | | Madiana | | | Dealed | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Optum | | | MarketScar | | | Medicare | | | Pooled | |
| Variable Number of patients | Rivaroxaban<br>3.03 | Apixaban<br>2 3.03 | St. Diff | Rivaroxaban<br>3.69 | Apixaban<br>3.69 | St. Diff | Rivaroxaban<br>7.47 | Apixaban<br>76 7.47 | St. Diff | Rivaroxaban<br>14.202 | Apixaban<br>14.202 | St. Diff |
| Age | 3,03 | 2 3,03 | 2 | 3,01 | 3,09 | | 7,4. | 7,47 | | 14,202 | 14,202 | |
| mean (sd) | 65.10 (16.13) | 65.21 (16.49) | -0.006743918 | 55.41 (15.52) | 55.52 (15.87) | -0.007008166 | 73.18 (12.05) | 73.20 (12.34) | -0.0016399 | 66.83 (13.95) | 66.90 (14.27) | -0.004960702 |
| median [IQR] Age categories | 68.00 [56.00, 77.00] | 68.00 [55.00, 78.00] | 0 | 56.00 [46.00, 64.0 | 00] 56.00 [45.00, 64.00] | 0 | 74.00 [68.00, 81.0 | 0] 74.00 [68.00, 82. | 00 0 | 68.04 (13.95) | 68.04 (14.27) | 0 |
| 18 - 54; n (%) | 704 (23.2%) | 740 (24.4%) | -0.028181129 | 1,653 (44.7%) | 1,662 (45.0%) | -0.00603211 | 601 (8.0%) | 586 (7.8%) | 0.007414632 | 2,958 (20.8%) | 2,988 (21.0%) | -0.004918922 |
| 55 - 64; n (%) | 521 (17.2%) | 498 (16.4%) | 0.021399249 | 1,191 (32.2%) | 1,170 (31.7%) | 0.010723258 | 576 (7.7%) | 604 (8.1%) | -0.01482957 | 2,288 (16.1%) | 2,272 (16.0%) | 0.002724285 |
| 65 - 74; n (%)<br>>=75; n (%) | 834 (27.5%)<br>973 (32.1%) | 784 (25.9%)<br>1,010 (33.3%) | 0.036172905<br>-0.025582051 | 407 (11.0%)<br>443 (12.0%) | 408 (11.0%)<br>454 (12.3%) | 0<br>-0.009182624 | 2,648 (35.4%)<br>3,651 (48.8%) | 2,668 (35.7%)<br>3,618 (48.4%) | -0.006267468<br>0.008003202 | 3,889 (27.4%)<br>5,067 (35.7%) | 3,860 (27.2%)<br>5,082 (35.8%) | 0.004489341<br>-0.002086535 |
| Calendar Year (2014-2020) | 373 (32.170) | 1,010 (33.376) | -0.023382031 | 443 (12.0%) | 434 (12.3%) | -0.009182024 | 3,031 (46.6%) | 3,010 (40.476) | 0.000003202 | 3,007 (33.770) | 3,082 (33.8%) | -0.002080333 |
| 2014; n (%) | 26 (0.9%) | 23 (0.8%) | 0.010893078 | 63 (1.7%) | 69 (1.9%) | -0.015043548 | 183 (2.4%) | 175 (2.3%) | 0.006601343 | 272 (1.9%) | 267 (1.9%) | 0 |
| 2015; n (%)<br>2016; n (%) | 187 (6.2%)<br>477 (15.7%) | 193 (6.4%)<br>472 (15.6%) | -0.008231777<br>0.002752331 | 450 (12.2%)<br>891 (24.1%) | 464 (12.6%)<br>861 (23.3%) | -0.012136825<br>0.018813637 | 1,518 (20.3%)<br>2.825 (37.8%) | 1,558 (20.8%)<br>2.838 (38.0%) | -0.012374437<br>-0.004122546 | 2,155 (15.2%)<br>4.193 (29.5%) | 2,215 (15.6%)<br>4,171 (29.4%) | -0.011082076<br>0.002193861 |
| 2017; n (%) | 621 (20.5%) | 630 (20.8%) | -0.007411238 | 897 (24.3%) | 881 (23.8%) | 0.011699196 | 2,950 (39.5%) | 2,905 (38.9%) | 0.012290361 | 4,468 (31.5%) | 4,416 (31.1%) | 0.00862608 |
| 2018; n (%) | 797 (26.3%) | 777 (25.6%) | 0.015969108 | 772 (20.9%) | 788 (21.3%) | -0.009803598 | 0 (0.0%) | 0 (0.0%) | 0 | 1,569 (11.0%) | 1,565 (11.0%) | 0 |
| 2019; n (%)<br>2020; n (%) | 704 (23.2%)<br>220 (7.3%) | 725 (23.9%)<br>212 (7.0%) | -0.016497898<br>0.011643529 | 621 (16.8%)<br>0 (0.0%) | 631 (17.1%)<br>0 (0.0%) | -0.00799595 | 0 (0.0%)<br>0 (0.0%) | 0 (0.0%) 0 (0.0%) | 0 | 1,325 (9.3%)<br>220 (1.5%) | 1,356 (9.5%)<br>212 (1.5%) | -0.006853375<br>0 |
| Race | 220 (7.3%) | 212 (7.0%) | 0.011043323 | 0 (0.0%) | 0 (0.0%) | 0 | 0 (0.0%) | 0 (0.0%) | 0 | 220 (1.376) | 212 (1.576) | · · |
| White; n (%) | 2,141 (70.6%) | 2,149 (70.9%) | -0.006594737 | 0 (0.0%) | 0 (0.0%) | 0 | 6,174 (82.6%) | 6,188 (82.8%) | -0.005287565 | 8,315 (58.5%) | 8,337 (58.7%) | -0.004060522 |
| Asian; n (%)<br>Black: n (%) | 50 (1.6%)<br>445 (14.7%) | 44 (1.5%)<br>457 (15.1%) | 0.008095242<br>-0.011233341 | 0 (0.0%) | 0 (0.0%) | 0 | 72 (1.0%)<br>938 (12.5%) | 66 (0.9%)<br>951 (12.7%) | 0.010309004<br>-0.006026858 | 122 (0.9%)<br>1.383 (9.7%) | 110 (0.8%)<br>1.408 (9.9%) | 0.010893078 |
| Biack, 11 (%)Hispanic; n (%) | 245 (8.1%) | 235 (7.8%) | 0.011233341 | 0 (0.0%) | 0 (0.0%) | 0 | 118 (1.6%) | 117 (1.6%) | 0 | 363 (2.6%) | 352 (2.5%) | 0.006343679 |
| North American Native; n (%) | 0 (0.0%) | 0 (0.0%) | 0 | 0 (0.0%) | 0 (0.0%) | 0 | 25 (0.3%) | 22 (0.3%) | 0 | 25 (0.2%) | 22 (0.2%) | 0 |
| Other; n (%) | 0 (0.0%) | 0 (0.0%) | 0 | 0 (0.0%) | 0 (0.0%) | 0 | 66 (0.9%) | 57 (0.8%) | 0.010893078 | 66 (0.5%) | 57 (0.4%) | 0.014941191 |
| Unknown/Missing; n (%) Gender | 151 (5.0%) | 147 (4.8%) | 0.00926502 | 0 (0.0%) | 0 (0.0%) | U | 83 (1.1%) | 75 (1.0%) | 0.009810761 | 234 (1.6%) | 222 (1.6%) | 0 |
| Males; n (%) | 1,404 (46.3%) | 1,427 (47.1%) | -0.016035478 | 1,969 (53.3%) | 1,953 (52.9%) | 0.008015485 | 2,990 (40.0%) | 2,968 (39.7%) | 0.006127613 | 6,363 (44.8%) | 6,348 (44.7%) | 0.002011118 |
| Females; n (%) | 1,628 (53.7%) | 1,605 (52.9%) | 0.016035478 | 1,725 (46.7%) | 1,741 (47.1%) | -0.008015485 | 4,486 (60.0%) | 4,508 (60.3%) | -0.006127613 | 7,839 (55.2%) | 7,854 (55.3%) | -0.002011118 |
| RegionNortheast; n (%) | 353 (11.6%) | 341 (11.2%) | 0.012586336 | 737 (20.0%) | 751 (20.3%) | -0.007479099 | 1,451 (19.4%) | 1,445 (19.3%) | 0.002531382 | 2,541 (17.9%) | 2,537 (17.9%) | 0 |
| Nortneast; n (%)South; n (%) | 1,330 (43.9%) | 1,347 (44.4%) | -0.010069283 | 1,643 (44.5%) | 1,637 (44.3%) | 0.004025335 | 3,275 (43.8%) | 3,282 (43.9%) | -0.002531382 | 6,248 (44.0%) | 6,266 (44.1%) | -0.002014314 |
| Midwest; n (%) | 676 (22.3%) | 678 (22.4%) | -0.00240044 | 848 (23.0%) | 849 (23.0%) | 0 | 1,624 (21.7%) | 1,629 (21.8%) | -0.002423977 | 3,148 (22.2%) | 3,156 (22.2%) | 0 |
| West; n (%) | 667 (22.0%) | 662 (21.8%) | 0.004835971<br>0.025841432 | 459 (12.4%)<br>7 (0.2%) | 447 (12.1%)<br>10 (0.3%) | 0.009150276<br>-0.020026051 | 1,119 (15.0%) | 1,112 (14.9%)<br>8 (0.1%) | 0.002804418 | 2,245 (15.8%) | 2,221 (15.6%) | 0.005497535 |
| Unknown+missing; n (%) Combined comorbidity score, 180 days | 6 (0.2%) | 4 (0.1%) | 0.025841432 | 7 (0.2%) | 10 (0.3%) | -0.020026051 | 7 (0.1%) | 8 (0.1%) | U | 20 (0.1%) | 22 (0.2%) | -0.025841432 |
| mean (sd) | 3.08 (2.42) | 3.13 (2.42) | -0.020661157 | 1.97 (1.78) | 1.98 (1.76) | -0.005649627 | 2.51 (2.14) | 2.52 (2.16) | -0.004651112 | 2.49 (2.12) | 2.51 (2.12) | -0.009433962 |
| median [IQR] | 3.00 [1.00, 4.00] | 3.00 [1.00, 5.00] | 0 | 2.00 [1.00, 3.00] | 2.00 [1.00, 3.00] | 0 | 2.00 [1.00, 4.00] | 2.00 [1.00, 4.00] | 0 | 2.21 (2.12) | 2.21 (2.12) | 0 |
| Lifestyle Factors Lifestyle - Smoking : n (%) | 1.128 (37.2%) | 1.123 (37.0%) | 0.004140175 | 752 (20.4%) | 742 (20.1%) | 0.007465285 | 3.003 (40.2%) | 3.057 (40.9%) | -0.014257314 | 4.883 (34.4%) | 4.922 (34.7%) | -0.006308768 |
| Lifestyle - Drug abuse or dependence; n (%) | 143 (4.7%) | 152 (5.0%) | -0.013965503 | 109 (3.0%) | 101 (2.7%) | 0.018029973 | 275 (3.7%) | 287 (3.8%) | -0.005263632 | 527 (3.7%) | 540 (3.8%) | -0.005263632 |
| Lifestyle - Alcohol abuse or dependence ; n (%) | 128 (4.2%) | 117 (3.9%) | 0.01521892 | 97 (2.6%) | 96 (2.6%) | 0 | 232 (3.1%) | 233 (3.1%) | 0 | 457 (3.2%) | 446 (3.1%) | 0.005725279 |
| Comorbidities DM - Diabetic Retinopathy; n (%) | 36 (1.2%) | 32 (1.1%) | 0.009379237 | 20 (0.5%) | 23 (0.6%) | -0.013521541 | 71 (0.9%) | 78 (1.0%) | -0.010309004 | 127 (0.9%) | 133 (0.9%) | 0 |
| DM - Diabetic Neuropathy; n (%) | 163 (5.4%) | 172 (5.7%) | -0.013103373 | 108 (2.9%) | 107 (2.9%) | 0.013321341 | 361 (4.8%) | 376 (5.0%) | -0.010309004 | 632 (4.5%) | 655 (4.6%) | -0.004798523 |
| DM - Diabetic Nephropathy; n (%) | 136 (4.5%) | 140 (4.6%) | -0.004798523 | 61 (1.7%) | 68 (1.8%) | -0.00762637 | 249 (3.3%) | 245 (3.3%) | 0 | 446 (3.1%) | 453 (3.2%) | -0.005725279 |
| DM - Diabetes with peripheral circulatory disorders; n (%) | 6 (0.2%) | 6 (0.2%) | 0 0.009379237 | 7 (0.2%) | 7 (0.2%) | 0 | 23 (0.3%) | 24 (0.3%) | 0 | 036 (0.3%) | 37 (0.3%) | 0 |
| DM - Diabetes with peripheral circulatory disorders and lower extremity amputation; n (%) DM - Diabetes with unspecified complications; n (%) | 35 (1.2%)<br>52 (1.7%) | 34 (1.1%)<br>52 (1.7%) | 0.009379237 | 16 (0.4%)<br>555 (15.0%) | 14 (0.4%)<br>573 (15.5%) | -0.013908354 | 91 (1.2%)<br>102 (1.4%) | 95 (1.3%)<br>106 (1.4%) | -0.009000794<br>0 | 142 (1.0%)<br>709 (5.0%) | 143 (1.0%)<br>731 (5.1%) | -0.004566758 |
| DM - Diabetes mellitus without mention of complications; n (%) | 600 (19.8%) | 603 (19.9%) | -0.002507081 | 46 (1.2%) | 52 (1.4%) | -0.01765699 | 1,709 (22.9%) | 1,734 (23.2%) | -0.007123349 | 2,355 (16.6%) | 2,389 (16.8%) | -0.005362296 |
| CV - Hypertension; n (%) | 1,947 (64.2%) | 1,945 (64.1%) | 0.002085246 | 1,885 (51.0%) | 1,859 (50.3%) | 0.014001526 | 5,908 (79.0%) | 5,907 (79.0%) | 0 | 9,740 (68.6%) | 9,711 (68.4%) | 0.004305568 |
| CV-Hyperlipidemia; n (%) CV-Acute MI; n (%) | 1,426 (47.0%)<br>164 (5.4%) | 1,422 (46.9%)<br>153 (5.0%) | 0.002003732<br>0.018016556 | 1,264 (34.2%)<br>140 (3.8%) | 1,249 (33.8%)<br>148 (4.0%) | 0.008444082<br>-0.010330986 | 4,068 (54.4%)<br>359 (4.8%) | 4,081 (54.6%)<br>360 (4.8%) | -0.004016307 | 6,758 (47.6%)<br>663 (4.7%) | 6,752 (47.5%)<br>661 (4.7%) | 0.002002406 |
| CV-ACS/unstable angina; n (%) | 103 (3.4%) | 103 (3.4%) | 0 | 94 (2.5%) | 95 (2.6%) | -0.010330380 | 273 (3.7%) | 268 (3.6%) | 0.00533248 | 470 (3.3%) | 466 (3.3%) | 0 |
| CV - Old MI; n (%) | 129 (4.3%) | 137 (4.5%) | -0.00975169 | 60 (1.6%) | 66 (1.8%) | -0.015471833 | 380 (5.1%) | 376 (5.0%) | 0.004566758 | 569 (4.0%) | 579 (4.1%) | -0.005072843 |
| CV - Stable angina; n (%) | 77 (2.5%) | 82 (2.7%) | -0.012568181 | 72 (1.9%) | 69 (1.9%) | 0 | 194 (2.6%)<br>1,549 (20.7%) | 189 (2.5%) | 0.006343679<br>-0.004927618 | 343 (2.4%) | 340 (2.4%) | 0<br>-0.002684358 |
| CV - Coronary atherosclerosis and other forms of chronic ischemic heart disease; n (%) CV - Other atherosclerosis: n (%) | 475 (15.7%)<br>30 (1.0%) | 471 (15.5%)<br>34 (1.1%) | 0.005511859<br>-0.009810761 | 333 (9.0%)<br>15 (0.4%) | 342 (9.3%)<br>14 (0.4%) | -0.010405288<br>0 | 1,549 (20.7%)<br>57 (0.8%) | 1,561 (20.9%)<br>66 (0.9%) | -0.004927618 | 2,357 (16.6%)<br>102 (0.7%) | 2,374 (16.7%)<br>114 (0.8%) | -0.002684358 |
| CV - Previous cardiac procedure (CABG or PTCA or Stent) + History of CABG or PTCA; n (%) | 150 (4.9%) | 140 (4.6%) | 0.01410434 | 48 (1.3%) | 50 (1.4%) | -0.008665401 | 566 (7.6%) | 564 (7.5%) | 0.003785069 | 764 (5.4%) | 754 (5.3%) | 0.004443896 |
| CV-Ischemic stroke; n (%) | 192 (6.3%) | 179 (5.9%) | 0.016713886 | 162 (4.4%) | 149 (4.0%) | 0.019942251 | 540 (7.2%) | 565 (7.6%) | -0.015280984 | 894 (6.3%) | 893 (6.3%) | 0 |
| CV-Hemorrhagic stroke; n (%) CV-TIA; n (%) | 7 (0.2%)<br>53 (1.7%) | 7 (0.2%)<br>49 (1.6%) | 0.007850082 | 2 (0.1%)<br>52 (1.4%) | 2 (0.1%)<br>50 (1.4%) | 0 | 11 (0.1%)<br>159 (2.1%) | 14 (0.2%)<br>148 (2.0%) | -0.025841432<br>0.007057056 | 020 (0.1%)<br>264 (1.9%) | 23 (0.2%)<br>247 (1.7%) | -0.025841432<br>0.015043548 |
| CV - Other cerebrovascular disease; n (%) | 99 (3.3%) | 97 (3.2%) | 0.005639422 | 74 (2.0%) | 73 (2.0%) | 0 | 246 (3.3%) | 254 (3.4%) | -0.005557486 | 419 (3.0%) | 424 (3.0%) | 0 |
| CV - Late effects of cerebrovascular disease; n (%) | 78 (2.6%) | 73 (2.4%) | 0.012810515 | 43 (1.2%) | 36 (1.0%) | 0.019175887 | 228 (3.0%) | 230 (3.1%) | -0.005815379 | 349 (2.5%) | 339 (2.4%) | 0.00646853 |
| CV - Heart failure (CHF); n (%) CV - Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) | 433 (14.3%)<br>269 (8.9%) | 439 (14.5%)<br>270 (8.9%) | -0.005696572<br>0 | 308 (8.3%)<br>165 (4.5%) | 326 (8.8%)<br>173 (4.7%) | -0.01788185<br>-0.009547328 | 1,253 (16.8%)<br>664 (8.9%) | 1,266 (16.9%)<br>681 (9.1%) | -0.002671587<br>-0.006988608 | 1,994 (14.0%)<br>1.098 (7.7%) | 2,031 (14.3%)<br>1.124 (7.9%) | -0.008607498<br>-0.007457963 |
| CV - Peripheral Vascular Disease (PVD) or PVD Surgery; n (%) CV - Other cardiac dysrhythmia; n (%) | 469 (15.5%) | 470 (8.5%) | 0 | 482 (13.0%) | 471 (12.8%) | 0.005966615 | 1,151 (15.4%) | 1,177 (15.7%) | -0.008278658 | 2,102 (14.8%) | 2,118 (14.9%) | -0.007457963 |
| CV - Cardiac conduction disorders; n (%) | 271 (8.9%) | 280 (9.2%) | -0.010456866 | 199 (5.4%) | 195 (5.3%) | 0.004443896 | 680 (9.1%) | 657 (8.8%) | 0.010509348 | 1,150 (8.1%) | 1,132 (8.0%) | 0.003675589 |
| CV-Other CVD; n (%) | 954 (31.5%) | 952 (31.4%) | 0.002153705<br>-0.00240428 | 934 (25.3%) | 917 (24.8%) | 0.011539515 | 1,999 (26.7%) | 2,016 (27.0%)<br>2,047 (27.4%) | -0.00676931<br>-0.008989059 | 3,887 (27.4%) | 3,885 (27.4%)<br>3,411 (24.0%) | 0<br>-0.007039548 |
| CV Medications - ACE inhibitors; n (%) CV Medications - ARBs; n (%) | 674 (22.2%)<br>449 (14.8%) | 675 (22.3%)<br>451 (14.9%) | -0.00240428<br>-0.002812191 | 678 (18.4%)<br>449 (12.2%) | 689 (18.7%)<br>449 (12.2%) | -0.007718039<br>0 | 2,019 (27.0%)<br>1,341 (17.9%) | 2,047 (27.4%)<br>1,351 (18.1%) | -0.008989059<br>-0.00520581 | 3,371 (23.7%)<br>2,239 (15.8%) | 3,411 (24.0%)<br>2,251 (15.8%) | 0.007039548 |
| CV Medications - Alpha blockers; n (%) | 251 (8.3%) | 265 (8.7%) | -0.014343368 | 216 (5.8%) | 222 (6.0%) | -0.008488151 | 769 (10.3%) | 756 (10.1%) | 0.006608366 | 1,236 (8.7%) | 1,243 (8.8%) | -0.003538997 |
| CV Medications - Beta blockers; n (%) | 733 (24.2%) | 714 (23.5%) | 0.016426065 | 732 (19.8%) | 720 (19.5%) | 0.007550055 | 2,528 (33.8%) | 2,539 (34.0%) | -0.004225036 | 3,993 (28.1%) | 3,973 (28.0%) | 0.002225966 |
| CV Medications - Loop Diuretics; n (%) CV Medications - Other diuretics; n (%) | 355 (11.7%)<br>74 (2.4%) | 350 (11.5%)<br>73 (2.4%) | 0.006245641 | 259 (7.0%)<br>84 (2.3%) | 267 (7.2%)<br>83 (2.2%) | -0.007787468<br>0.006742995 | 1,315 (17.6%)<br>227 (3.0%) | 1,316 (17.6%)<br>225 (3.0%) | 0 | 1,929 (13.6%)<br>385 (2.7%) | 1,933 (13.6%)<br>381 (2.7%) | 0 |
| CV Medications - Other didretics, it (%) CV Medications - Use of nitrates; n (%) | 74 (2.4%) | 68 (2.2%) | 0.006742995 | 64 (1.7%) | 63 (1.7%) | 0 | 379 (5.1%) | 365 (4.9%) | 0.009176726 | 514 (3.6%) | 496 (3.5%) | 0.005404261 |
| CV Medications - Use of statins; n (%) | 967 (31.9%) | 950 (31.3%) | 0.012905912 | 936 (25.3%) | 898 (24.3%) | 0.023157643 | 3,142 (42.0%) | 3,111 (41.6%) | 0.008109871 | 5,045 (35.5%) | 4,959 (34.9%) | 0.012563221 |
| CV Medications - Use of other lipid-lowering drugs; n (%) | 108 (3.6%)<br>608 (20.1%) | 106 (3.5%)<br>617 (20.3%) | 0.005404261<br>-0.004981432 | 151 (4.1%)<br>570 (15.4%) | 137 (3.7%)<br>553 (15.0%) | 0.0206628<br>0.011141586 | 355 (4.7%)<br>1.887 (25.2%) | 364 (4.9%)<br>1.905 (25.5%) | -0.009356117<br>-0.00689636 | 614 (4.3%)<br>3.065 (21.6%) | 607 (4.3%)<br>3.075 (21.7%) | 0 -0.002428018 |
| CV Medications - calcium channel blockers; n (%) CV Medications - Use of low weight molecular heparins; n (%) | 608 (20.1%)<br>60 (2.0%) | 61 / (20.3%)<br>58 (1.9%) | -0.004981432<br>0.007232055 | 570 (15.4%)<br>80 (2.2%) | 553 (15.0%)<br>85 (2.3%) | -0.006742995 | 1,887 (25.2%) | 1,905 (25.5%)<br>129 (1.7%) | 0.00689636 | 3,065 (21.6%)<br>277 (2.0%) | 3,075 (21.7%)<br>272 (1.9%) | 0.002428018 |
| Other Comorbidity - Osteoporosis; n (%) | 293 (9.7%) | 284 (9.4%) | 0.010207536 | 120 (3.2%) | 116 (3.1%) | 0.005725279 | 959 (12.8%) | 962 (12.9%) | -0.002988238 | 1,372 (9.7%) | 1,362 (9.6%) | 0.00338667 |
| Other Comorbidity - Dementia; n (%) | 414 (13.7%) | 419 (13.8%) | -0.002903819 | 173 (4.7%) | 161 (4.4%) | 0.014395901 | 1,321 (17.7%) | 1,317 (17.6%) | 0.002622987 | 1,908 (13.4%) | 1,897 (13.4%) | 0 |
| Other Comorbidity - Hyperthyroidism + Hypothyroidism + Other disorders of thyroid gland; n (%) Other Comorbidity - Edma: n (%) | 653 (21.5%)<br>703 (23.2%) | 626 (20.6%)<br>695 (22.9%) | 0.022078362 | 553 (15.0%)<br>596 (16.1%) | 574 (15.5%)<br>592 (16.0%) | -0.013908354<br>0.002724285 | 694 (9.3%)<br>1.352 (18.1%) | 700 (9.4%)<br>1.345 (18.0%) | -0.003434875<br>0.002600083 | 1,900 (13.4%)<br>2.651 (18.7%) | 1,900 (13.4%)<br>2.632 (18.5%) | 0.005139996 |
| Other Comorbidity - Edema; n (%) Other Comorbidity - Depression; n (%) | 703 (23.2%)<br>600 (19.8%) | 695 (22.9%)<br>590 (19.5%) | 0.007123349 | 596 (16.1%)<br>484 (13.1%) | 592 (16.0%)<br>469 (12.7%) | 0.002/24285 | 1,352 (18.1%)<br>1,562 (20.9%) | 1,345 (18.0%) | 0.002600083 | 2,651 (18.7%)<br>2,646 (18.6%) | 2,632 (18.5%) | 0.005139996 |
| Other Comorbidity - Anxiety; n (%) | 665 (21.9%) | 661 (21.8%) | 0.002419971 | 607 (16.4%) | 600 (16.2%) | 0.005414708 | 1,565 (20.9%) | 1,540 (20.6%) | 0.007398021 | 2,837 (20.0%) | 2,801 (19.7%) | 0.00752129 |
| Other Comorbidity - Pneumonia; n (%) | 551 (18.2%) | 551 (18.2%) | 0 | 502 (13.6%) | 531 (14.4%) | -0.023057149 | 1,324 (17.7%) | 1,315 (17.6%) | 0.002622987 | 2,377 (16.7%) | 2,397 (16.9%) | -0.00534952 |
| Other Comorbidity - COPD; n (%) Other Comorbidity - Asthma; n (%) | 597 (19.7%)<br>328 (10.8%) | 626 (20.6%)<br>328 (10.8%) | -0.022438553 | 344 (9.3%)<br>369 (10.0%) | 356 (9.6%)<br>368 (10.0%) | -0.010255736 | 1,780 (23.8%)<br>888 (11.9%) | 1,804 (24.1%)<br>892 (11.9%) | -0.007029454 | 2,721 (19.2%)<br>1,585 (11.2%) | 2,786 (19.6%)<br>1,588 (11.2%) | -0.010115728 |
| Other Comorbidity - Astrima; n (%) Other Comorbidity - Acute renal disease; n (%) | 406 (13.4%) | 408 (13.5%) | -0.002930932 | 369 (10.0%) | 313 (8.5%) | -0.007210169 | 1,049 (14.0%) | 1,041 (13.9%) | 0.002886276 | 1,762 (11.2%) | 1,762 (11.2%) | 0 |
| Other Comorbidity CKD Stage 1; n (%) | 10 (0.3%) | 7 (0.2%) | 0.020026051 | 5 (0.1%) | 4 (0.1%) | 0 | 21 (0.3%) | 22 (0.3%) | 0 | 36 (0.3%) | 33 (0.2%) | 0.020026051 |
| Other Comorbidity - CKD Stage 2; n (%) | 64 (2.1%) | 72 (2.4%) | -0.020229904 | 27 (0.7%) | 27 (0.7%) | 0 | 131 (1.8%) | 125 (1.7%) | 0.00762637 | 222 (1.6%) | 224 (1.6%) | 0 |
| Other Comorbidity - CKD Stage 3; n (%) | 265 (8.7%) | 270 (8.9%) | -0.007059825 | 112 (3.0%) | 119 (3.2%) | -0.011539699 | 638 (8.5%) | 658 (8.8%) | -0.010672474 | 1,015 (7.1%) | 1,047 (7.4%) | -0.01156917 |

| Other Comorbidity - Occurrence of chronic renal insufficiency w/o CKD ; n (%) Other Comorbidity - Occurrence of miscellaneous renal insufficiency; n (%) Other Comorbidity - Hypertansive nephropathy n (%) Other Comorbidity - Osteractive sleep apnex, n (%) Other Comorbidity - Osteractive sleep apnex, n (%) Other Comorbidity - Other arthritis, a rknopathies and musculoskeletal pain; n (%) Other Comorbidity - Other arthritis, a rknopathies and musculoskeletal pain; n (%) Other Comorbidity - Fractures, n (%) Other Comorbidity - Fractures, n (%) Other Comorbidity - Selpsionder, n (%) Other Comorbidity - Selpsionder, n (%) Other Comorbidity - Selpsionder, n (%) Other Comorbidity - Selpsionder, n (%) Other Comorbidity - Selpsionder, n (%) | 200 (6.6%)<br>297 (9.8%)<br>289 (9.5%)<br>269 (8.5%)<br>870 (28.7%)<br>2,025 (66.8%)<br>1,039 (34.3%)<br>331 (10.9%)<br>403 (13.3%)<br>92 (3.0%)<br>211 (7.0%) | 194 (6.4%)<br>293 (9.7%)<br>295 (9.7%)<br>273 (9.0%)<br>898 (29.6%)<br>2,049 (67.6%)<br>1,052 (34.7%)<br>342 (11.3%)<br>408 (13.5%)<br>97 (3.2%)<br>201 (6.7%)<br>117 (3.9%) | 0.008112806<br>0.003371124<br>0.006789107<br>0.014119914<br>0.019804989<br>0.017040573<br>0.008414603<br>0.012733753<br>0.005871114<br>0.011539699<br>0.011876602<br>0.02191923 | 90 (2.4%)<br>210 (5.7%)<br>133 (3.6%)<br>399 (10.8%)<br>717 (19.4%)<br>2,284 (61.8%)<br>1,079 (29.2%)<br>298 (8.1%)<br>174 (4.7%)<br>137 (3.7%)<br>105 (2.8%)<br>47 (1.3%) | 100 (2.7%)<br>220 (6.0%)<br>138 (3.7%)<br>389 (10.5%)<br>739 (20.0%)<br>2,264 (61.3%)<br>1,089 (25.5%)<br>296 (8.0%)<br>137 (3.7%)<br>94 (2.5%) | -0.019031802<br>-0.012783272<br>-0.00533248<br>0.000725329<br>-0.015085952<br>0.010278117<br>-0.005658815<br>-0.003675589<br>-0.013965503<br>0<br>0.016678813<br>0.00900794 | 518 (6.9%)<br>607 (8.1%)<br>852 (11.4%)<br>552 (7.4%)<br>2,532 (33.9%)<br>4,654 (62.3%)<br>2,509 (33.6%)<br>750 (10.0%)<br>395 (5.3%)<br>267 (3.6%)<br>520 (7.0%)<br>386 (5.2%) | 516 (6.9%)<br>607 (8.1%)<br>851 (11.4%)<br>550 (7.4%)<br>2,528 (33.8%)<br>4,631 (61.9%)<br>2,516 (33.7%)<br>746 (10.0%)<br>378 (5.1%)<br>275 (3.7%)<br>519 (6.9%)<br>370 (4.9%) | 0<br>0<br>0<br>0<br>0<br>0.002113275<br>0.008245145<br>-0.002116349<br>0<br>0.00900004<br>-0.00533248<br>0.003932333<br>0.013700558 | 808 (5.7%)<br>1,114 (7.8%)<br>1,274 (9.0%)<br>1,274 (9.0%)<br>4,119 (29.0%)<br>4,627 (32.5%)<br>1,379 (9.7%)<br>972 (6.8%)<br>496 (3.5%)<br>836 (5.9%)<br>540 (3.8%) | 810 (5.7%)<br>1,120 (7.9%)<br>1,284 (9.0%)<br>1,212 (8.5%)<br>4,165 (29.3%)<br>8,944 (63.0%)<br>4,657 (32.8%)<br>1,384 (9.7%)<br>970 (6.8%)<br>509 (3.6%)<br>816 (5.7%)<br>530 (3.7%) | 0<br>-0.003718076<br>0<br>0<br>-0.006601375<br>0.002071813<br>-0.004263336<br>0<br>-0.005404261<br>0.008556468 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure - Hip Surgery; n (%) | 33 (1.1%) | 33 (1.1%) | 0 | 27 (0.7%) | 28 (0.8%) | -0.011590746 | 86 (1.2%) | 79 (1.1%) | 0.009379237 | 146 (1.0%) | 140 (1.0%) | 0 |
| Medications DM Medications - Meditinides: n (%) | 3 (0.1%) | 3 (0.1%) | 0 | 2 (0.1%) | 4 (0.1%) | 0 | 18 (0.2%) | 17 (0.2%) | 0 | 23 (0.2%) | 24 (0.2%) | 0 |
| DM Medications - AGIs; n (%) | 0 (0.0%) | 0 (0.0%) | 0 0.00975169 | 1 (0.0%) | 1 (0.0%) | 0 | - | 308 (4.1%) | -<br>-0.005072843 | - | - | 0.04800597 |
| DM Medications - Insulin; n (%) DM Medications - Glitazones; n (%) | 137 (4.5%)<br>15 (0.5%) | 129 (4.3%)<br>11 (0.4%) | 0.00975169 | 20 (0.5%)<br>145 (3.9%) | 21 (0.6%)<br>145 (3.9%) | -0.013521541<br>0 | 299 (4.0%)<br>49 (0.7%) | 308 (4.1%)<br>43 (0.6%) | -0.005072843<br>0.012444223 | 581 (4.1%)<br>209 (1.5%) | 458 (3.2%)<br>199 (1.4%) | 0.04800597 |
| DM Medications - 1st and 2nd Generation SUs; n (%) DM Medications - DPP-4 Inhibitors: n (%) | 140 (4.6%)<br>49 (1.6%) | 142 (4.7%)<br>42 (1.4%) | -0.004749134<br>0.016454358 | 137 (3.7%)<br>75 (2.0%) | 144 (3.9%)<br>75 (2.0%) | -0.0104606 | 398 (5.3%)<br>175 (2.3%) | 399 (5.3%)<br>188 (2.5%) | 0<br>-0.013067988 | 675 (4.8%)<br>299 (2.1%) | 685 (4.8%)<br>305 (2.1%) | 0 |
| DM Medications - GLP-1 RA; n (%) | 25 (0.8%) | 20 (0.7%) | 0.011590746 | 38 (1.0%) | 38 (1.0%) | 0 | 38 (0.5%) | 40 (0.5%) | 0 | 101 (0.7%) | 98 (0.7%) | 0 |
| DM Medications - SGLT-2 Inhibitors ; n (%) DM Medications - Metformin: n (%) | 27 (0.9%)<br>285 (9.4%) | 21 (0.7%)<br>284 (9.4%) | 0.022452077 | 42 (1.1%)<br>328 (8.9%) | 44 (1.2%)<br>335 (9.1%) | -0.009379237<br>-0.006988608 | 33 (0.4%)<br>757 (10.1%) | 37 (0.5%)<br>770 (10.3%) | -0.014941191<br>-0.006608366 | 102 (0.7%)<br>1,370 (9.6%) | 102 (0.7%)<br>1,389 (9.8%) | 0<br>-0.00675776 |
| Other Medications - Use of NSAIDs; n (%) | 555 (18.3%) | 597 (19.7%) | -0.035692574 | 822 (22.3%) | 851 (23.0%) | -0.016724339 | 1,508 (20.2%) | 1,517 (20.3%) | -0.002488413 | 2,885 (20.3%) | 2,965 (20.9%) | -0.014836086 |
| Other Medications - Use of other hypertension drugs; n (%) Other Medications - Digoxin; n (%) | 143 (4.7%)<br>10 (0.3%) | 149 (4.9%)<br>9 (0.3%) | -0.009356117<br>0 | 103 (2.8%)<br>8 (0.2%) | 120 (3.2%)<br>10 (0.3%) | -0.023450027<br>-0.020026051 | 458 (6.1%)<br>51 (0.7%) | 476 (6.4%)<br>49 (0.7%) | -0.012393785<br>0 | 704 (5.0%)<br>69 (0.5%) | 745 (5.2%)<br>68 (0.5%) | -0.009091097<br>0 |
| Other Medications - Use of Anti-arrhythmics; n (%) | 12 (0.4%) | 15 (0.5%) | -0.014941191 | 13 (0.4%) | 16 (0.4%) | 0 | 36 (0.5%) | 36 (0.5%) | 0 | 61 (0.4%) | 67 (0.5%) | -0.014941191 |
| Other Medications - Use of antipsychotics; n (%) Other Medications - Use of dementia meds; n (%) | 195 (6.4%)<br>174 (5.7%) | 198 (6.5%)<br>161 (5.3%) | -0.004070982<br>0.017546054 | 154 (4.2%)<br>66 (1.8%) | 144 (3.9%)<br>66 (1.8%) | 0.01521892<br>0 | 775 (10.4%)<br>667 (8.9%) | 774 (10.4%)<br>648 (8.7%) | 0<br>0.007059825 | 1,124 (7.9%)<br>907 (6.4%) | 1,116 (7.9%)<br>875 (6.2%) | 0<br>0.008231777 |
| Other Medications - Use of antiparkinsonian meds; n (%) | 106 (3.5%) | 100 (3.3%) | 0.011035921<br>0.020657013 | 78 (2.1%) | 88 (2.4%) | -0.020229904 | 427 (5.7%) | 442 (5.9%) | -0.008556468 | 611 (4.3%) | 630 (4.4%) | -0.004902461<br>0.003785069 |
| Other Medications - Use of anxiolytics/hypnotics; n (%) Other Medications - Use of anticonvulsants; n (%) | 196 (6.5%)<br>553 (18.2%) | 182 (6.0%)<br>590 (19.5%) | -0.033243244 | 269 (7.3%)<br>525 (14.2%) | 260 (7.0%)<br>504 (13.6%) | 0.011643529<br>0.017344373 | 613 (8.2%)<br>1,679 (22.5%) | 618 (8.3%)<br>1,679 (22.5%) | -0.003634718<br>0 | 1,078 (7.6%)<br>2,757 (19.4%) | 1,060 (7.5%)<br>2,773 (19.5%) | -0.002526433 |
| Other Medications - Use of antidepressants; n (%) Other Medications - Use of lithium; n (%) | 849 (28.0%)<br>9 (0.3%) | 865 (28.5%)<br>10 (0.3%) | -0.011105971 | 901 (24.4%)<br>15 (0.4%) | 881 (23.8%)<br>12 (0.3%) | 0.014029188<br>0.01693335 | 2,600 (34.8%)<br>41 (0.5%) | 2,592 (34.7%)<br>39 (0.5%) | 0.002100064 | 4,350 (30.6%)<br>065 (0.5%) | 4,338 (30.5%)<br>61 (0.4%) | 0.002170994<br>0.014941191 |
| Other Medications - Use of Benzos; n (%) | 467 (15.4%) | 472 (15.6%) | -0.005526338 | 563 (15.2%) | 560 (15.2%) | 0 | 1,562 (20.9%) | 1,565 (20.9%) | 0 | 2,592 (18.3%) | 2,597 (18.3%) | 0 |
| Other Medication - Use of CNS stimulants; n (%) Other Medications - Use of opioids; n (%) | 25 (0.8%)<br>1,208 (39.8%) | 25 (0.8%)<br>1,228 (40.5%) | 0<br>-0.014280199 | 54 (1.5%)<br>1,666 (45.1%) | 62 (1.7%)<br>1,658 (44.9%) | -0.015939924<br>0.004020159 | 37 (0.5%)<br>3,150 (42.1%) | 47 (0.6%)<br>3,162 (42.3%) | -0.013521541<br>-0.004049587 | 116 (0.8%)<br>6,024 (42.4%) | 134 (0.9%)<br>6,048 (42.6%) | -0.010893078<br>-0.004045782 |
| Other Medications - Use of COPD/asthma meds; n (%) | 550 (18.1%) | 560 (18.5%) | -0.01034497 | 582 (15.8%) | 598 (16.2%) | -0.010911057 | 1,735 (23.2%) | 1,757 (23.5%) | -0.007091277 | 2,867 (20.2%) | 2,915 (20.5%) | -0.007451594 |
| Other Medications - Use of oral corticosteroids; n (%) Other Medications - Use of Sympatomimetic agents; n (%) | 837 (27.6%)<br>44 (1.5%) | 877 (28.9%)<br>39 (1.3%) | -0.028878088<br>0.01702328 | 953 (25.8%)<br>99 (2.7%) | 975 (26.4%)<br>109 (3.0%) | -0.013662146<br>-0.018029973 | 2,413 (32.3%)<br>73 (1.0%) | 2,401 (32.1%)<br>69 (0.9%) | 0.004280438<br>0.010309004 | 4,203 (29.6%)<br>216 (1.5%) | 4,253 (29.9%)<br>217 (1.5%) | -0.006562313<br>0 |
| Other Medications - Use of bisphosphonates; n (%) | 98 (3.2%) | 92 (3.0%) | 0.011539699 | 40 (1.1%) | 38 (1.0%) | 0.009810761 | 316 (4.2%) | 308 (4.1%) | 0.005013965 | 454 (3.2%) | 438 (3.1%) | 0.005725279 |
| Other Medications - Use of thiazide; n (%) Other Medications - Use of estrogens, progestins, androgens; n (%) | 246 (8.1%)<br>215 (7.1%) | 253 (8.3%)<br>204 (6.7%) | -0.007289615<br>0.015782439 | 233 (6.3%)<br>513 (13.9%) | 245 (6.6%)<br>504 (13.6%) | -0.012213147<br>0.008711531 | 716 (9.6%)<br>342 (4.6%) | 739 (9.9%)<br>333 (4.5%) | -0.010113486<br>0.004798523 | 1,195 (8.4%)<br>1,070 (7.5%) | 1,237 (8.7%)<br>1,041 (7.3%) | -0.010728836<br>0.007640325 |
| Healthcare Utilization HU - Bone mineral density; n (%) | 90 (3.0%) | 93 (3.1%) | -0.005815379 | 50 (1.4%) | 53 (1.4%) | 0 | 294 (3.9%) | 307 (4.1%) | -0.01020634 | 434 (3.1%) | 453 (3.2%) | -0.005725279 |
| HU - Occurrence of creatinine tests ordered ; n (%) HU - Number of D-dimer tests | 167 (5.5%) | 183 (6.0%) | -0.021479316 | 160 (4.3%) | 168 (4.5%) | -0.00975169 | 526 (7.0%) | 533 (7.1%) | -0.003906444 | 853 (6.0%) | 658 (4.6%) | 0.062521186 |
| mean (sd)median [IQR] | 0.12 (0.36)<br>0.00 [0.00, 0.00] | 0.12 (0.36)<br>0.00 [0.00, 0.00] | 0 | 0.13 (0.39)<br>0.00 [0.00, 0.00] | 0.13 (0.39)<br>0.00 [0.00, 0.00] | 0 | 0.11 (0.34)<br>0.00 [0.00, 0.00] | 0.10 (0.34)<br>0.00 [0.00, 0.00] | 0.029411765<br>0 | 0.12 (0.36)<br>0.00 (0.36) | 0.11 (0.36)<br>0.00 (0.36) | 0.027777778<br>0 |
| HU - Number of CRP, high-sensitivity CRP testsmean (sd) | 0.12 (0.52) | 0.12 (0.54) | 0 | 0.11 (0.53) | 0.11 (0.63) | 0 | 0.15 (0.61) | 0.16 (0.65) | -0.015865023 | 0.13 (0.83) | 0.14 (0.62) | -0.013650685 |
| median (IQR) HU - Colonoscopy; n (%) | 0.00 [0.00, 0.00]<br>102 (3.4%) | 0.00 [0.00, 0.00]<br>126 (4.2%) | 0<br>-0.041850988 | 0.00 [0.00, 0.00]<br>142 (3.8%) | 0.00 [0.00, 0.00]<br>130 (3.5%) | 0<br>0.015997896 | 0.00 [0.00, 0.00]<br>263 (3.5%) | 0.00 [0.00, 0.00]<br>264 (3.5%) | 0 | 0.00 (0.83)<br>507 (3.6%) | 0.00 (0.62)<br>520 (3.7%) | 0<br>-0.00533248 |
| HU - Colonoscopy; n (%)<br>HU - Flu vaccine; n (%) | 446 (14.7%) | 423 (14.0%) | 0.019967792 | 352 (9.5%) | 354 (9.6%) | -0.003402473 | 2,224 (29.7%) | 2,204 (29.5%) | 0.004381258 | 3,022 (21.3%) | 2,981 (21.0%) | 0.007346291 |
| HU - Mammogram; n (%)<br>HU - PSA test or Prostate exam for DRE; n (%) | 249 (8.2%)<br>253 (8.3%) | 241 (7.9%)<br>256 (8.4%) | 0.011026916<br>-0.003614858 | 291 (7.9%)<br>350 (9.5%) | 281 (7.6%)<br>310 (8.4%) | 0.011220031<br>0.038540897 | 665 (8.9%)<br>679 (9.1%) | 684 (9.1%)<br>668 (8.9%) | -0.006988608<br>0.006988608 | 1,205 (8.5%)<br>1,282 (9.0%) | 1,206 (8.5%)<br>1,234 (8.7%) | 0<br>0.010562758 |
| HU - Pap smear; n (%) | 106 (3.5%) | 105 (3.5%) | 0 | 225 (6.1%) | 225 (6.1%) | 0 | 187 (2.5%) | 173 (2.3%) | 0.013067988 | 518 (3.6%) | 503 (3.5%) | 0.005404261 |
| HU - Pneumonia vaccine; n (%) Frailty Score: Empirical Version 365 days (ICD-9 and ICD-10) V2 | 685 (22.6%) | 668 (22.0%) | 0.0144145 | 465 (12.6%) | 472 (12.8%) | -0.006006521 | 2,451 (32.8%) | 2,413 (32.3%) | 0.010671113 | 3,601 (25.4%) | 3,553 (25.0%) | 0.009213264 |
| mean (sd) | 0.20 (0.07) | 0.20 (0.07) | 0 | 0.16 (0.05) | 0.16 (0.05) | 0 | 0.21 (0.07) | 0.21 (0.07) | 0 | 0.19 (0.07) | 0.19 (0.07) | 0 |
| median [IQR] CHADS2 score, 180 days | 0.18 [0.14, 0.23] | 0.18 [0.14, 0.23] | 0 | 0.15 [0.12, 0.18] | 0.15 [0.13, 0.19] | 0 | 0.20 [0.16, 0.25] | 0.20 [0.16, 0.25] | 0 | 0.18 (0.07) | 0.18 (0.07) | 0 |
| mean (sd) | 0.89 (1.07)<br>1.00 [0.00, 1.00] | 0.90 (1.08)<br>1.00 (0.00, 1.00) | -0.009302225<br>0 | 0.58 (0.92) | 0.59 (0.94)<br>0.00 [0.00, 1.00] | -0.010752067<br>0 | 0.79 (0.92)<br>1.00 [0.00, 1.00] | 0.79 (0.93) | 0 | 0.76 (0.95)<br>0.74 (0.95) | 0.76 (0.97) | 0 |
| HU - Number of Hospitalizations | | | - | | | · · | | , | · · | | | |
| mean (sd)median [IQR] | 1.20 (0.57)<br>1.00 [1.00, 1.00] | 1.21 (0.61)<br>1.00 [1.00, 1.00] | -0.016939423<br>0 | 1.14 (0.43)<br>1.00 [1.00, 1.00] | 1.14 (0.43)<br>1.00 [1.00, 1.00] | 0 | 1.30 (0.71)<br>1.00 [1.00, 1.00] | 1.30 (0.65)<br>1.00 [1.00, 1.00] | 0<br>-0.440747751 | 1.24 (0.62)<br>1.00 (0.62) | 1.24 (0.59)<br>1.00 (0.59) | 0 |
| HU - Number of hospital days | 6.06 (8.57) | 6.02 (6.84) | 0.005159025 | 5.06 (6.92) | 5.11 (7.46) | -0.006949205 | 6.66 (8.13) | 6.61 (7.49) | 0.006396682 | 6.12 (7.93) | 6.09 (7.35) | 0.003923876 |
| mean (sd)median [IQR] | 4.00 [3.00, 6.00] | 4.00 [3.00, 6.00] | 0.005159025 | 3.00 [2.00, 5.00] | 3.00 [2.00, 5.00] | -0.006949205<br>0 | 4.00 [3.00, 7.00] | 4.00 [3.00, 7.00] | 0.006396682 | 6.12 (7.93)<br>3.74 (7.93) | 6.09 (7.35)<br>3.74 (7.35) | 0.003923876 |
| HU - Number of Emergency Department (ED) visitsmean (sd) | 1.78 (2.70) | 1.76 (2.25) | 0.008047622 | 3.23 (4.82) | 3.15 (5.30) | 0.015792523 | 2.10 (2.95) | 2.10 (3.36) | 0 | 2.33 (5.07) | 2.30 (3.79) | 0.006702426 |
| median [IQR] | 1.00 [1.00, 2.00] | 1.00 [1.00, 2.00] | 0 | 2.00 [0.00, 4.00] | 2.00 [0.00, 4.00] | 0 | 1.00 [1.00, 3.00] | 1.00 [1.00, 3.00] | Ö | 1.26 (5.07) | 1.26 (3.79) | 0 |
| HU - Number of internal medicine/family medicine visitsmean (sd) | 10.86 (15.64) | 11.07 (15.13) | -0.013647784 | 5.25 (7.86) | 5.28 (7.79) | -0.003833827 | 11.23 (11.34) | 11.19 (10.62) | 0.003641031 | 9.60 (16.95) | 9.63 (11.14) | -0.002091717 |
| median [IQR] | 6.00 [2.00, 14.00] | 6.00 [2.00, 14.00] | 0 | 3.00 [1.00, 7.00] | 3.00 [1.00, 7.00] | 0 | 8.00 [4.00, 14.00] | 8.00 [5.00, 14.00 | ] 0 | 6.27 (16.95) | 6.27 (11.14) | 0 |
| HU - Number of different/distinct medication prescriptionsmean (sd) | 8.43 (5.39) | 8.51 (5.40) | -0.014828539 | 7.87 (5.42) | 7.90 (5.21) | -0.005643302 | 9.82 (5.36) | 9.80 (5.24) | 0.003773343 | 9.02 (7.82) | 9.03 (5.27) | -0.001499693 |
| median [IQR]<br>HU - Number of Office visits | 7.00 [4.00, 11.00] | 8.00 [4.00, 12.00] | -0.185356732 | 7.00 [4.00, 11.00] | 7.00 [4.00, 11.00] | 0 | 9.00 [6.00, 13.00] | 9.00 [6.00, 13.00] | ] 0 | 8.05 (7.82) | 8.27 (5.27) | -0.032993243 |
| mean (sd) | 4.46 (4.12) | 4.56 (3.94) | -0.02480771 | 4.37 (4.07) | 4.38 (4.09) | -0.002450973 | 11.13 (11.80) | 11.20 (12.00) | -0.005882145 | 7.95 (13.10) | 8.01 (9.14) | -0.005312131 |
| median [IQR] HU - Number of Cardiologist visits | 3.00 [2.00, 6.00] | 4.00 [2.00, 6.00] | -0.248077102 | 3.00 [1.00, 6.00] | 3.00 [1.00, 6.00] | 0 | 8.00 [3.00, 15.00] | 8.00 [3.00, 15.00 | ] 0 | 5.63 (13.10) | 5.85 (9.14) | -0.019477815 |
| mean (sd) | 2.59 (4.05) | 2.58 (3.72) | 0.002571684 | 0.64 (1.84) | 0.65 (1.83) | -0.005449571 | 2.69 (4.21) | 2.69 (4.21) | 0 | 2.14 (5.38) | 2.14 (3.63) | 0 |
| median [IQR] HU - Number electrocardiograms | 1.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | 0 | 0.00 [0.00, 0.00] | 0.00 [0.00, 0.25] | 0 | 1.00 [0.00, 3.00] | 1.00 [0.00, 3.00] | | 0.74 (5.38) | 0.74 (3.63) | U |
| mean (sd)<br>median [IQR] | 1.91 (2.10)<br>1.00 [1.00, 3.00] | 1.90 (2.01)<br>1.00 [1.00, 3.00] | 0.004865014 | 0.78 (1.18)<br>0.00 [0.00, 1.00] | 0.77 (1.16)<br>0.00 (0.00, 1.00) | 0.008546696 | 1.96 (2.02)<br>1.00 [1.00, 3.00] | 1.95 (1.94)<br>1.00 (1.00, 3.00) | 0.005049475 | 1.64 (2.70)<br>0.74 (2.70) | 1.63 (1.79)<br>0.74 (1.79) | 0.004365584 |
| HU - Number of echocardiograms | | | - | | | · | | | | | | • |
| mean (sd)median (IQR) | 1.07 (2.92)<br>1.00 [0.00, 1.00] | 1.09 (3.00)<br>1.00 [0.00, 1.00] | -0.00675614<br>0 | 0.67 (0.74)<br>1.00 [0.00, 1.00] | 0.67 (0.79)<br>1.00 [0.00, 1.00] | 0 | 0.77 (0.94)<br>1.00 [0.00, 1.00] | 0.78 (0.95)<br>1.00 [0.00, 1.00] | -0.010581862<br>0 | 0.81 (2.26)<br>1.00 (2.26) | 0.82 (1.60)<br>1.00 (1.60) | -0.005107228<br>0 |
| HU - Number of neurologist visits | | | • | | | _ | | | _ | | | |
| mean (sd)median [IQR] | 0.59 (2.29)<br>0.00 [0.00, 0.00] | 0.60 (2.42)<br>0.00 [0.00, 0.00] | -0.004244668<br>0 | 0.35 (1.54)<br>0.00 [0.00, 0.00] | 0.35 (2.36)<br>0.00 [0.00, 0.00] | 0 | 0.55 (2.06)<br>0.00 [0.00, 0.00] | 0.55 (2.15)<br>0.00 [0.00, 0.00] | 0 | 0.51 (2.90)<br>0.00 (2.90) | 0.51 (2.27)<br>0.00 (2.27) | 0 |
| HU - Fecal occult blood (FOB) test; n (%) HU - Number of PT or aPTTt tests | 70 (2.3%) | 76 (2.5%) | -0.013067988 | 101 (2.7%) | 96 (2.6%) | 0.00622603 | 199 (2.7%) | 198 (2.6%) | 0.00622603 | 370 (2.6%) | 370 (2.6%) | 0 |
| 110 - Number of Frod de FILL Lesis | | | | | | | | | | | | |

| mean (sd)<br>median [IQR] | 0.48 (1.19)<br>0.00 [0.00, 0.00] | 0.48 (1.21)<br>0.00 [0.00, 0.00] | 0 | 0.46 (1.11)<br>0.00 [0.00, 0.00] | 0.46 (1.19)<br>0.00 [0.00, 0.00] | 0 | 0.26 (0.63)<br>0.00 [0.00, 0.00] | 0.25 (0.66)<br>0.00 [0.00, 0.00] | 0.015499685<br>0 | 0.36 (1.33)<br>0.00 (1.33) | 0.35 (0.95)<br>0.00 (0.95) | 0.008652578<br>0 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Socioeconomic Status Proxy Variables | | | | | | | | | | | | |
| SES - Mean Copay for per prescription cost (charges in U.S. \$) | | | | | | | | | | | | |
| mean (sd) | 18.05 (23.07) | 18.18 (27.14) | -0.005161322 | 11.59 (18.47) | 11.98 (20.33) | -0.020080033 | 19.52 (36.04) | 19.14 (33.98) | 0.010849347 | 17.14 (43.26) | 17.07 (29.54) | 0.001889809 |
| median [IQR] | 11.75 [4.01, 23.76] | 10.66 [3.95, 22.77] | 0.043275704 | 7.21 [1.00, 14.46] | 7.19 [0.77, 15.00] | 0.001029745 | 10.06 [2.95, 24.13] | 9.71 [2.88, 23.73] | 0.00999282 | 9.68 (43.26) | 9.26 (29.54) | 0.011338853 |
| Missing; n (%) | 272 (9.0%) | 266 (8.8%) | 0.007023903 | 719 (19.5%) | 703 (19.0%) | 0.012682127 | 452 (6.0%) | 446 (6.0%) | 0 | 1,443 (10.2%) | 1,415 (10.0%) | 0 |
| SES - Copay: pharmacy cost | | | | | | | | | | | | |
| mean (sd) | 170.24 (267.22) | 171.77 (323.09) | -0.005160655 | 92.46 (181.81) | 96.72 (189.23) | -0.022957894 | 9.92 (5.45) | 9.90 (5.33) | 0.003710345 | 65.62 (224.46) | 67.04 (177.80) | -0.007013088 |
| median [IQR] | 70.00 [10.00, 221.90] | 65.46 [10.00, 211.95] | 0.015313315 | 20.79 [0.00, 110.18 | 3] 20.00 [0.00, 112.32] | 0.00425745 | 9.00 [6.00, 13.00] | 9.00 [6.00, 13.00] | 0 | 25.09 (224.46) | 23.91 (177.80) | 0.005827778 |
| SES - Business type: Commercial vs Medicare | | | | | | | | | | | | |
| Commerical; n (%) | 1,171 (38.6%) | 1,154 (38.1%) | 0.010283158 | 2,840 (76.9%) | 2,829 (76.6%) | 0.00710188 | 0 (0.0%) | 0 (0.0%) | 0 | 4,011 (28.2%) | 3,983 (28.0%) | 0.004449523 |
| Medicare; n (%) | 1,861 (61.4%) | 1,878 (61.9%) | -0.010283158 | 854 (23.1%) | 865 (23.4%) | -0.00710188 | 0 (0.0%) | 0 (0.0%) | 0 | 2,715 (19.1%) | 2,743 (19.3%) | -0.005077794 |
| SES - Low income indicator; n (%) | 461 (15.2%) | 467 (15.4%) | -0.00555577 | 0 (0.0%) | 0 (0.0%) | 0 | 0 (0.0%) | 0 (0.0%) | 0 | 461 (3.2%) | 467 (3.3%) | -0.005639422 |
| SES - Urban vs Rural (MSA variable) | | | | | | | | | | | | |
| Urban; n (%) | 0 (0.0%) | 0 (0.0%) | 0 | 2,479 (67.1%) | 2,458 (66.5%) | 0.012740979 | 0 (0.0%) | 0 (0.0%) | 0 | 2,479 (17.5%) | 2,458 (17.3%) | 0.005275539 |
| Rural; n (%) | 0 (0.0%) | 0 (0.0%) | 0 | 365 (9.9%) | 369 (10.0%) | -0.003340775 | 0 (0.0%) | 0 (0.0%) | 0 | 365 (2.6%) | 369 (2.6%) | 0 |
| Unknown/Missing; n (%) | 0 (0.0%) | 0 (0.0%) | 0 | 850 (23.0%) | 867 (23.5%) | -0.011836599 | 0 (0.0%) | 0 (0.0%) | 0 | 850 (6.0%) | 867 (6.1%) | -0.004194449 |
| SES - Dual Status; n (%) | 0 (0.0%) | 0 (0.0%) | 0 | 0 (0.0%) | 0 (0.0%) | 0 | 2,256 (30.2%) | 2,260 (30.2%) | 0 | 2,256 (15.9%) | 2,260 (15.9%) | 0 |
| SES - Generic name prescription - unique value | | | | | | | | | | | | |
| mean (sd) | 8.43 (5.39) | 8.51 (5.40) | -0.014828539 | 7.87 (5.42) | 7.90 (5.21) | -0.005643302 | 9.82 (5.36) | 9.80 (5.24) | 0.003773343 | 9.02 (7.82) | 9.03 (5.27) | -0.001499693 |
| median [IQR] | 7.00 [4.00, 11.00] | 8.00 [4.00, 12.00] | -0.185356732 | 7.00 [4.00, 11.00] | 7.00 [4.00, 11.00] | 0 | 9.00 [6.00, 13.00] | 9.00 [6.00, 13.00] | 0 | 8.05 (7.82) | 8.27 (5.27) | -0.032993243 |
| SES - Brand name prescription - unique value | | | | | | | | | | | | |
| mean (sd) | 8.52 (5.50) | 8.60 (5.51) | -0.014532237 | 7.96 (5.53) | 8.00 (5.32) | -0.007371891 | 9.92 (5.45) | 9.90 (5.33) | 0.003710345 | 9.11 (7.97) | 9.13 (5.37) | -0.002943122 |
| median [IQR] | 8.00 [4.00, 12.00] | 8.00 [4.00, 12.00] | 0 | 7.00 [4.00, 11.00] | 7.00 [4.00, 11.00] | 0 | 9.00 [6.00, 13.00] | 9.00 [6.00, 13.00] | 0 | 8.27 (7.97) | 8.27 (5.37) | 0 |







The c-statistics for the propensity score model, pre-matching was 0.746. The post-matching c-statistic was 0.541

The c-statistics for the propensity score model, pre-matching was 0.732. The post-matching c-statistic was 0.538

The c-statistics for the propensity score model, pre-matching was 0.674. The post-matching c-statistic was 0.52